### GlaxoSmithKline group of companies

 Division
 : Worldwide Development

 Information Type
 : Reporting and Analysis Plan (RAP)

Title: Reporting and Analysis Plan for Phase IIb, Randomized (Stratified), Double-Blind (Sponsor Open), Parallel-Group, Placebo-Controlled, Dose-Finding Study of Nemiralisib (GSK2269557) Added to Standard of Care (SoC) Versus SoC Alone in Participants Diagnosed with an Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)Compound Number: GSK2269557Effective Date: 10-OCT-2018

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200879 and at the planned interim analyses.
- This RAP is intended to describe the efficacy, safety and pharmacokinetic analyses required for the study.
- This version of the RAP includes amendments to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

RAP Author(s): PPD

Statistics Leader, (Respiratory Clinical Statistics)

| Approver | Date | Approval Method |
|---|---|---|
| TA Director (Respiratory Clinical Statistics) | 10-OCT-2018 | eSignature |
| Programming Manager (Respiratory Clinical Programming) | 10-OCT-2018 | eSignature |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Principal Programmer (Respiratory Clinical Programming) | 26-SEP-2018 | Email |
| PPD | 26 SED 2019 | Email |
| Clinical Development Director (Respiratory) | 26-SEP-2018 | Email |
| PPD | 24-SEP-2018 | Email |
| Clinical Development Manager (Respiratory) | 24-3E1-2018 | Eman |
| PPD | | |
| Medical Director (Global Clinical Safety and | 25-SEP-2018 | Email |
| Pharmacovigilance) | | |
| PPD | | |
| Manager, Clinical Pharmacology (Clinical | 25-SEP-2018 | Email |
| Pharmacology Modelling and Simulation) | | |
| PPD | | |
| Director, Patient Centred Outcomes (Value Evidence & Outcomes) | 01-OCT-2018 | Email |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | ON | 8 |
| 2. | CLIMAN | | KEY PROTOCOL INFORMATION | Q |
| ۷. | 2.1. | | Dbjective(s) and Endpoint(s) | |
| | 2.1. | Study C | Design | 0<br>11 |
| | ۷.۷. | Study L | Jesign | |
| 3. | ΡΙ ΔΝ | NED AN | ALYSES | 11 |
| ٥. | 3.1. | | Analyses | |
| | 0.1. | 3.1.1. | | |
| | | J. 1. 1. | 3.1.1.1. Futility rules | |
| | 3.2. | Final A | nalyses | |
| | | | · | |
| 4. | | | PULATIONS | |
| | 4.1. | Protoco | ol Deviations | 15 |
| 5. | CONS | SIDERAT | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CON\ | | IS | |
| | 5.1. | Study T | Freatment & Sub-group Display Descriptors | 16 |
| | 5.2. | | e Definitions | |
| | 5.3. | Multice | ntre Studies | 17 |
| | 5.4. | Examin | nation of Covariates and Subgroups | 17 |
| | | 5.4.1. | Covariates | |
| | | 5.4.2. | Examination of Subgroups | 18 |
| | 5.5. | Other C | Considerations for Data Analyses and Data Handling | 00 |
| | | Conver | ntions | 20 |
| 6. | STUD | | LATION ANALYSES | |
| | 6.1. | Overvie | ew of Planned Study Population Analyses | |
| | | 6.1.1. | Concomitant medications | 20 |
| 7. | EFFIC | CACY AN | IALYSES | 21 |
| | 7.1. | | / Efficacy Analyses | |
| | | 7.1.1. | | |
| | | 7.1.2. | Primary Statistical Analyses | |
| | | | 7.1.2.1. Model Checking & Diagnostics | 23 |
| | | 7.1.3. | Sensitivity and Supportive Analyses | |
| | | 7.1.4. | Subgroup Analyses | |
| | 7.2. | Second | dary Efficacy Analyses | |
| | | 7.2.1. | Rate of exacerbations | 24 |
| | | | 7.2.1.1. Statistical analyses | 25 |
| | | | 7.2.1.2. Subgroup analyses | <mark>26</mark> |
| | | | 7.2.1.3. Exploratory analyses | <mark>26</mark> |
| | | 7.2.2. | Time to next exacerbation | <mark>26</mark> |
| | | | 7.2.2.1. Statistical analyses | <mark>27</mark> |
| | | | 7.2.2.2. Subgroup analyses | |
| | | 7.2.3. | Change from baseline in Clinic Visit trough FEV <sub>1</sub> | 27 |
| | | | 7.2.3.1. Statistical Analyses | 27 |
| | | | 7.2.3.2. Subgroup analyses | |
| | | 7.2.4. | Change from hospital discharge in clinic visit trough FEV <sub>1</sub> | 28 |

| | | 7.2.4.1. | Statistical analyses | 28 |
|---|---|---|---|---|
| | 7.2.5. | EXAcerba | ations of Chronic Pulmonary Disease Tool - | |
| | | | eported Outcome (EXACT) | 28 |
| | | 7.2.5.1. | Proportion of participants achieving EXACT- | |
| | | | defined recovery from index exacerbation | 29 |
| | | 7.2.5.2. | Time to EXACT-defined recovery from index | |
| | | 7.2.0.2. | exacerbation | 30 |
| | | 7.2.5.3. | Severity of subsequent HCRU-defined | |
| | | 1.2.5.5. | exacerbation(s) defined by EXACT | 30 |
| | | 7051 | Statistical analyses | 30 |
| | | 7.2.5.4. | Statistical analyses | 30 |
| | | 7.2.5.5. | Subgroup analyses | 31 |
| | | 7.2.5.6. | Sensitivity and supportive analyses | 31 |
| | 7.2.6. | | ssessment Test (CAT) | 31 |
| | | 7.2.6.1. | Proportion of responders using the CAT | |
| | | 7.2.6.2. | Change from baseline in CAT Total Score | 32 |
| | | 7.2.6.3. | Statistical analyses | 32 |
| | | 7.2.6.4. | Subgroup analyses | 33 |
| | 7.2.7. | St. Georg | e's Respiratory Questionnaire for COPD | |
| | | Patients ( | SGRQ-C) | 33 |
| | | 7.2.7.1. | Proportion of responders on the SGRQ Total | |
| | | | Score | 33 |
| | | 7.2.7.2. | Change from baseline in SGRQ Total Score | |
| | | 7.2.7.3. | Statistical analyses | |
| | | 7.2.7.3.<br>7.2.7.4. | | |
| | 700 | | Subgroup analyses | |
| | 7.2.8. | | nedication use | 34 |
| | | 7.2.8.1. | Rescue medication use via the clip-on | |
| | | | Propeller Sensor for MDI | |
| | | 7.2.8.2. | Statistical analyses | |
| 7.3. | | | y Analyses | |
| | 7.3.1. | Change f | rom Day 84 in Clinic Visit trough FEV₁ | 36 |
| | | 7.3.1.1. | Statistical analysis | 36 |
| | 7.3.2. | E-RS:CO | PD (Evaluating Respiratory Symptoms in COPD) | 36 |
| | 7.3.3. | | s of HCRU related to exacerbations | |
| | | 7.3.3.1. | Re-hospitalisation within 30 days of index | |
| | | | exacerbation | 37 |
| | | 7332 | Time from resolution of index exacerbation to | |
| | | 7.0.0.2. | next exacerbation | |
| | | 7.3.3.3. | Subsequent exacerbation treatment type | |
| | 7.3.4. | | Ce | |
| | 7.5. <del>4</del> . | 7.3.4.1. | Number of actuations of double-blind study | 57 |
| | | 7.3.4.1. | | |
| | | | treatment measured by the clip-on Propeller | 00 |
| | | | Sensor | |
| | | 7.3.4.2. | Missing EXACT-PRO data | 38 |
| | 7.3.5. | | tory/infective markers in blood and sputum in | |
| | | | acute exacerbation of COPD | |
| | 7.3.6. | Other spi | rometry measurements | 38 |
| | 7.3.7. | Other syr | nptoms suggestive of exacerbation | 38 |
| | 7.3.8. | | tion of exacerbating COPD participants and | |
| | | | of response to nemiralisib using machine | |
| | | | echniques | 38 |
| | | | 1 <del></del> | |
| SAFF | TY ANAI | YSES | | 39 |

8.

| | 8.1. | | | lyses | |
|---|---|---|---|---|---|
| | | 8.1.1. | | vents of Special Interest | 39 |
| | | | | Post-inhalation Cough Immediately Following Dosing | 20 |
| | | | | Paradoxical bronchospasm | |
| | 8.2. | Clinical I | | nalyses | |
| | 8.3. | | | 98 | |
| | 8.4. | | | | |
| | 0.4. | wortanty | | | 40 |
| 9. | | | | YSES | |
| | 9.1. | Population | on of Interes | t | 41 |
| | 9.2. | Drug Co | ncentration l | Measures | 41 |
| 10. | POPU | LATION F | PK ANALYS | IS | 42 |
| | 10.1. | | | netic Parameters | |
| 11. | PHARI | MACOKII | NETIC / PHA | ARMACODYNAMIC ANALYSES | 43 |
| 12. | REFE | RENCES. | | | 44 |
| 13. | | | | | 45 |
| | 13.1. | | | Deviation Management and Definitions for Per | |
| | 40.0 | | | from Per Protocol Population | |
| | 13.2. | | | nent Windows | |
| | | 13.2.1. | | of Assessment Windows for Analyses | |
| | | | | Hospital discharge | |
| | 13.3. | Annendi | | EXACT-Defined Recovery for CAT Triggerhases and Treatment Emergent Adverse | 40 |
| | 13.3. | | | | 47 |
| | | 13.3.1. | | ods | |
| | | 10.0.1. | | 12-Week Treatment Period | |
| | | | | 12-Week Follow-Up Period | |
| | | 13.3.2. | | ses | |
| | | | | Study Phases for Concomitant Medication | |
| | | 13.3.3. | | Emergent Flag for Adverse Events | |
| | 13.4. | Appendi | | splay Standards & Handling Conventions | |
| | | 13.4.1. | | Process | |
| | | 13.4.2. | | Standards | |
| | | 13.4.3. | Reporting S | Standards for Pharmacokinetic | 49 |
| | 13.5. | Appendi | x 5: Derived | and Transformed Data | 50 |
| | | 13.5.1. | | | |
| | | 13.5.2. | Study Popu | ulation | 50 |
| | | 13.5.3. | | | |
| | 13.6. | | | ng Standards for Missing Data | |
| | | 13.6.1. | | Withdrawals | |
| | | 13.6.2. | - | f Missing Data | |
| | 40 = | | | Handling of Missing and Partial Dates | |
| | 13.7. | | | of Potential Clinical Importance | |
| | | 13.7.1. | - | Values | |
| | | 13.7.2. | | | |
| | | 13.7.3. | vitai Signs | | 54 |

| 13.8. | | 8: Population Pharmacokinetic (PopPK) Analyses | |
|---|---|---|---|
| | | Population Pharmacokinetic (PopPK) Methodology | . 55 |
| | 13.8.2. | 1 \ 1 / | |
| | | Specification | |
| 13.9. | | 9: Pharmacokinetic / Pharmacodynamic Analyses | |
| | 13.9.1. | Pharmacokinetic/Pharmacodynamic Methodology | .57 |
| 13.10. | | x 10: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 13.11. | <b>Appendix</b> | ( 11: List of Data Displays | .60 |
| | 13.11.1. | Data Display Numbering | .60 |
| | 13.11.2. | Mock Example Shell Referencing | .60 |
| | 13.11.3. | Deliverables | .60 |
| | 13.11.4. | Study Population Tables | .61 |
| | 13.11.5. | Study Population Figures | .63 |
| | 13.11.6. | Efficacy Tables | .64 |
| | | 13.11.6.1. Efficacy tables for Interim Analysis 1 | .64 |
| | | 13.11.6.2. Efficacy tables for Interim Analysis 2 | .66 |
| | | 13.11.6.3. Efficacy tables for End of Treatment Interim | |
| | | Analysis and SAC | .69 |
| | 13.11.7. | Efficacy Figures | |
| | | 13.11.7.1. Efficacy Figures for Interim Analysis 1 | |
| | | 13.11.7.2. Efficacy Figures for Interim Analysis 2 | |
| | | 13.11.7.3. Efficacy Figures for End of Treatment Interim | |
| | | Analysis and SAC | .83 |
| | 13.11.8. | Safety Tables | |
| | | Safety Figures | |
| | | .Pharmacokinetic Tables | |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 13.12. | | c 12: Example Mock Shells for Data Displays | |
| | | Example shell 1 | |
| | | Example Shell 2 | |
| | | Example shell 3 | |
| | | Example Shell 4 | |
| | | Example Shell 5 | |
| | | Example Shell 6 | |
| | | Example Shell 7 | |
| | | Example Shell 8 | |
| | | Example Shell 9 | |
| | | Example Shell 101 | |
| | | Example Shell 111 | |
| | | Example Shell 12 | |
| | | Example shell 131 | |
| | | Example Shell 141 | |
| | | Example Shell 151 | |
| | | Example shell 16 | |
| | | Example Shell 17 | |
| | | Example shell 18 | |
| | | Example Shell 19 | |
| | | Example Shell 20 | |
| | | • | 117 |

# 2019N398117\_00 200879

| 40.40.00 F I. OL. II.00 | 440 |
|----------------------------|-----|
| 13.12.22. Example Shell 22 | 118 |
| 13.12.23. Example Shell 23 | 119 |
| 13.12.24. Example Shell 24 | |
| 13.12.25.Example Shell 25 | |
| 13.12.26. Example Shell 26 | |
| 13.12.27.Example Shell 27 | |
| 13.12.28. Example Shell 28 | |
| 13.12.29 Example Shell 29 | |
| 13.12.30. Example Shell 30 | |
| 13.12.31.Example Shell 31 | |
| 13.12.32. Example Shell 32 | |
| 13.12.33. Example Shell 33 | |
| 13.12.34. Example Shell 34 | |
| 13.12.35. Example shell 35 | |
| 13.12.36. Example Shell 36 | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 200879.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

This study will be undertaken in participants who present with an acute moderate or severe exacerbation of COPD requiring Standard of Care (SoC), referred to as the index exacerbation.

# 2.1. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterise the dose response of<br>nemiralisib administered in addition to<br>SoC compared with placebo and SoC<br>in participants diagnosed with an<br>acute moderate or severe<br>exacerbation of COPD Secondary Objectives | Change from baseline in Clinic Visit trough forced expiratory volume in one second (FEV <sub>1</sub> ) at Day 84 measured post-bronchodilator Secondary Endpoints |
| To characterise the dose response | Rate of moderate and severe exacerbations over the 12- |
| and efficacy of nemiralisib administered in addition to SoC compared with placebo and SoC in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>Week Treatment Period</li> <li>Time to next moderate/severe exacerbation following index exacerbation</li> <li>Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days 14, 28, 56, and 84 (Day 84: post-bronchodilator is the primary endpoint; pre-bronchodilator is a secondary endpoint) and at hospital discharge (only for participants who are hospitalized for the index exacerbation)</li> <li>Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days, 14, 28, 56, and 84 (in participants hospitalized for index exacerbation only)</li> </ul> |
| To evaluate the treatment effect of nemiralisib in addition to SoC compared with placebo and SoC on symptoms indicative of an exacerbation and on health status using Patient-Reported Outcomes (PROs) in participants diagnosed with an acute moderate or severe exacerbation of COPD | EXAcerbations of Chronic Pulmonary Disease Tool (EXACT-PRO) Proportion of participants achieving the EXACT definition of recovery from the index exacerbation by Days 14, 28, 56, and 84 Time to recovery from index exacerbation Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT COPD Assessment Test (CAT) Proportion of responders using the CAT at Treatment Days 28, 56, and 84, and following EXACT defined |

| Objectives | Endpoints |
|---|---|
| To evaluate the usage of rescue medication in patients diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>recovery from the index exacerbation</li> <li>Change from baseline (Day 1) in CAT total score at Days 28, 56, and 84 and following EXACT defined recovery from the index exacerbation</li> <li>St. George's Respiratory Questionnaire (SGRQ) Total Score</li> <li>Proportion of responders on the SGRQ total score as measured by the SGRQ for COPD Patients (SGRQ-C) at Days 28, 56, and 84</li> <li>Change from baseline (Day 1) in SGRQ total score at Days 28, 56, and 84</li> <li>Rescue medication use (occasions/day), averaged over each week of treatment and over the 84-day treatment period</li> <li>The percentage of rescue-free days (24-hour periods) during each week of treatment and over the 84-day</li> </ul> |
| To evaluate the population pharmacokinetics of nemiralisib in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>Plasma nemiralisib concentrations and derived PK parameters (e.g., area under the curve [AUC (0-24) and AUC(0-t)], maximum concentration [Cmax], time at maximum concentration [Tmax], Ctrough) as appropriate will be collected in a subset of randomized participants (approximately 300) at selected sites as follows: trough (pre-dose) for the study treatment and post-dose for the study treatment from 0-1 hour and &gt;1 to 6 hours on Days 14 and 28 of the 12-Week Treatment Period</li> </ul> |
| To assess the safety and tolerability of<br>nemiralisib and placebo in participants<br>diagnosed with an acute moderate or<br>severe exacerbation of COPD | <ul> <li>Incidence of adverse events (AEs; including serious AEs and AE of Special Interest [AESI])</li> <li>Vital signs (pulse rate, systolic and diastolic blood pressure) (measured at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>12-lead electrocardiogram (ECG) assessments (performed at clinic Visits 1 [Screening], 3 [Day 14], 6 [Day 84], and 7 [Day 112] or Early Withdrawal Visit)</li> <li>Clinical laboratory tests (hematology and chemistry; performed at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>Incidence of COPD exacerbations</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To further characterize the dose<br>response, and efficacy, of nemiralisib<br>administered in addition to SoC<br>compared with placebo and SoC in<br>participants diagnosed with an acute<br>moderate or severe exacerbation of<br>COPD | <ul> <li>Rate of mild exacerbations over the 12-Week Treatment Period</li> <li>Rate of all exacerbations (mild, moderate and severe combined) over the 12-Week Treatment Period</li> <li>Time to next exacerbation (mild, moderate and severe combined)</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To evaluate the treatment effect of<br>nemiralisib in addition to SoC<br>compared with placebo and SoC on<br>symptom stability following an<br>exacerbation using Patient-Reported<br>Outcomes in participants diagnosed<br>with an acute moderate or severe<br>exacerbation of COPD | Stability of symptoms post recovery measured using E-RS:COPD (Evaluating Respiratory Symptoms in COPD) and subscales from Randomization (Visit 2) to Day 84 (Visit 6) |
| To explore the PK/PD relationship for<br>nemiralisib | <ul> <li>Relationship between drug exposure and<br/>Pharmacodynamic responses (e.g. efficacy, heart rate,<br/>clinical laboratory analytes and blood biomarkers) in the<br/>PK subset of participants (approximately 300) at selected<br/>sites</li> </ul> |
| To evaluate the treatment effect of<br>nemiralisib in addition to SoC<br>compared with placebo and SoC on<br>HCRU in participants who experience<br>a severe exacerbation of COPD | <ul> <li>Measures of HCRU related to severe exacerbations (e.g.,<br/>hospitalizations, length of hospital stay, re-hospitalization<br/>within 30 days, number of Emergency Room [ER] visits,<br/>etc.)</li> </ul> |
| To evaluate compliance with study treatment | Number of actuations of the double-blind study treatment<br>as measured by the clip-on Propeller Sensor (for<br>countries where the Propeller Sensor for ELLIPTA is<br>available) |
| To evaluate inflammatory markers in<br>blood in relation to acute exacerbation<br>of COPD | <ul> <li>Blood samples collected at Screening through Visit 7 (as part of the clinical laboratory blood samples) for analysis of blood eosinophil counts and inflammatory mediators</li> <li>Blood samples for analysis of inflammatory biomarkers (including but not limited to: high sensitivity C-reactive protein [hs-CRP], chemokine interferon-γ inducible protein 10 kDa (CXCL10)], and procalcitonin) collected at Visit 1 (Screening)</li> </ul> |
| To evaluate inflammatory and infective markers in sputum in relation to acute exacerbation of COPD | <ul> <li>Spontaneous sputum sample for analysis of inflammatory<br/>and infective markers collected at Screening/Day 1 (pre-<br/>dose) and Day 56 in participants who are willing and able<br/>to provide a sample</li> </ul> |
| To evaluate the potential post-<br>treatment impact of double-blind study<br>treatment during the 12-Week Post-<br>Treatment Follow-Up Period | <ul> <li>Change from baseline (Day 84) in Clinic Visit trough FEV1 measured pre- and postbronchodilator at Day 112, 140 and 168</li> <li>Rate of moderate and severe COPD exacerbation(s) during the 12-Week Follow-Up Period</li> <li>Rate of moderate and severe COPD exacerbation(s) over the 24 week study duration</li> <li>Time to next exacerbation following cessation of double blind study treatment</li> <li>Proportion of responders using the CAT at Days 112 and 168</li> <li>Change from baseline (Day 1) in CAT Total score at Days 112 and 168</li> <li>Proportion of responders on the SGRQ Total Score as measured by the SGRQ-C at Days 112 and 168</li> <li>Change from baseline (Day 1) in SGRQ total score at</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | Days 112 and 168 |
| | Severity of subsequent HCRU exacerbation defined by<br>EXACT |
| | E-RS: COPD and subscales from last dose of double-<br>blind study treatment |
| | Rescue medication use up to Day 112 |

# 2.2. Study Design

This is a Phase IIb, multicenter, randomized, stratified (by index COPD exacerbation severity [moderate or severe] and by whether or not the participant is in the PK Subgroup), double-blind (Sponsor Open), placebo-controlled, parallel-group study in participants who present with an acute moderate or severe exacerbation of COPD requiring Standard of Care (SoC).

This study consists of a Screening Period, a 12-Week Treatment Period and a 12-Week Post-Treatment Follow-Up Period. Randomization and the first dose of the double-blind study treatment administration (Visit 2/Day 1) should take place in the morning, as soon as possible following determination of eligibility and completion of the baseline measures, including the EXACT-PRO questionnaire for the day of randomization, and FEV<sub>1</sub> measurement and no later than 48 hours after the start of SoC.

PK Subgroup: Sparse PK sampling will be conducted in a subgroup of participants at selected sites. The PK Subgroup will be identical to the main study in terms of the study population, design, and conduct, with the exception of blood draws (3 per visit on Days 14 and 28) for PK analysis.

### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

Ongoing data reviews of unblinded safety data, conducted by an Internal Safety Review Committee (iSRC), will be performed throughout the trial. Details will be documented in the iSRC charter.

Interim analyses of the primary endpoint and key secondary endpoints to inform internal decision making will be conducted periodically throughout the trial. The first analysis (Interim Analysis 1) is planned to occur when approximately 170 participants complete 28 days of treatment, where approximately 50 of the 170 participants have an index exacerbation defined as severe. A change that could arise from this interim analysis is a specification of the stratification proportions by index exacerbation severity status (moderate or severe). This decision will be based on inspection of all available endpoints at the interim analysis.

Further interim analyses will be performed, depending on the observed recruitment rate. At least one interim analysis of the primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator will be performed to

determine whether or not any adjustments to the randomization ratio across doses would help optimize the characterization of the dose response profile for nemiralisib. This analysis (Interim Analysis 2) is planned to occur when approximately 300 participants complete 84 days of treatment or when approximately 400 participants remain to be randomized, whichever occurs first. Adjustments could include ceasing randomization to an existing dose(s) of nemiralisib and/or modification of the allocation ratios for the existing nemiralisib doses and/or addition of a 25mcg dose. Other changes may include specification of the stratification proportions by index exacerbation severity status.

An interim analysis of efficacy and safety data collected during the Double-Blind Treatment Period will be conducted when the last participant in the study has completed the 12-week Double-Blind Treatment Period (End of Treatment Interim Analysis). The aim of this analysis is to provide GSK with timely data to inform internal decision making, prior to the end of study.

The following table describes the endpoints that will be analysed/summarised at each interim:

| Interim | Purpose of interim | Endpoints |
|---|---|---|
| Interim Analysis 1 | To inform internal decision making | <ul> <li>Change from baseline in FEV<sub>1</sub> at Days 14, 28, and 56 measured pre- and post-bronchodilator</li> <li>Other spirometry measures (percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio</li> <li>On-treatment exacerbations</li> <li>Proportion of participants achieving EXACT-defined recovery by Days 14, 28, 56 and 84</li> </ul> |

| Interim | Purpose of interim | Endpoints |
|---|---|---|
| Interim Analysis 2 | To determine if any adjustments to the randomization ratio would help characterize the dose response profile for nemiralisib | <ul> <li>Endpoints listed for Interim Analysis 1 and also: <ul> <li>Change from baseline in FEV<sub>1</sub> at Day 84 measured pre- and post-bronchodilator</li> <li>Rate of (on-treatment) exacerbations over the 12-Week Treatment Period</li> <li>Time to next (on-treatment) exacerbation during the 12-Week Treatment Period</li> <li>Proportion of responders using the CAT</li> <li>Change from baseline in CAT Total Score</li> <li>Proportion of responders using the SGRQ</li> <li>Change from baseline in SGRQ Total Score</li> <li>Rescue medication use, as measured in eDiary</li> </ul> </li> </ul> |
| End of Treatment<br>Interim Analysis | To inform internal decision making | Selected Efficacy and Safety endpoints as defined in Appendix 11: List of Data Displays |

The statistical methods of analyses are described in Section 7.

The Respiratory Data Sciences Group will apply machine learning techniques to the interim data to determine if identifiable phenotypic sub-population(s) of COPD participants are present at baseline, and if they result in different responses to Nemiralisib, to predict which participants will respond to Nemiralisib therapy, and to identify/quantify relationship(s) between different endpoints and response measures. Details of these analyses will be described in a separate RAP and results will be reported separately to the Clinical Study Report (CSR).

The following functions will be unblinded to interim analysis data: Clinical Statistics, Clinical Programming and Respiratory Data Sciences Group. Other member of GSK will be unblinded to group level summary data following the interim analyses (as documented internally).

# 3.1.1. Futility analyses

At least one interim analysis for futility will be performed. The first analysis will occur at Interim Analysis 2, i.e. when 300 participants complete 84 days of treatment, or when approximately 400 participants remain to be randomized, whichever occurs first.

Futility will be assessed in a sequential manner.

- 1)Futility will first be assessed for the primary endpoint of change from baseline in FEV<sub>1</sub> at Day 84 by fitting a suitable dose response model, as described in Section 7.1.2.
- 2)If the posterior predictive probability of declaring success for this endpoint is low across all doses, then futility will be assessed for the rate of (on-treatment) exacerbations endpoint.
- 3)If the posterior predictive probability of declaring success for this endpoint is low, then the study may be stopped.

Any decision to stop will be made after a review of all the data summarised/analysed at the time of the interim, including the proportion of participants achieving the EXACT-defined recovery.

### 3.1.1.1. Futility rules

The decision rules for futility are defined as follows.

## Change from baseline in FEV1 at Day 84

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, across all doses, where success at the end of the trial for change from baseline in FEV<sub>1</sub> is defined as demonstrating >90% posterior probability that the true difference from placebo for any dose of nemiralisib is greater than 0.

### Rate of on-treatment (moderate/severe) exacerbations

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, where success at the end of the trial for rate of exacerbations is defined as demonstrating >80% posterior probability that the true rate reduction on 750 mcg dose versus placebo >0%.

If a different dose arm appears to be more efficacious than the 750 mcg arm, then futility may be assessed using the rate reduction for this arm versus placebo.

The pre-determined rules will act as guidelines for stopping the study for futility. All of the data summarised/analysed at the time of the interim will be reviewed prior to any decision to stop the study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE)<br>Population | All participants who are screened for eligibility. | Study Population |
| Modified Intent<br>To treat (MITT)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment.</li> <li>Participants will be analyzed according to the treatment that they were randomized to.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Per Protocol (PP)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment, excluding any participants with an important protocol deviation.</li> <li>Participants will be analyzed according to the treatment that they were randomized to.</li> </ul> | Sensitivity analyses of efficacy |
| Safety Population | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>Participants will be summarised according to the treatment that they actually received. <ul> <li>If participants receive &gt;1 treatment, then they will be summarised according to the most frequently dosed treatment. In cases where the frequency is equal, the participant will be assigned the lowest dose strength of nemiralisib</li> </ul> </li> </ul> | Safety |
| Pharmacokinetic<br>(PK) Population | <ul> <li>All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values).</li> <li>Participants will be summarised according to the treatment that they actually received</li> </ul> | • PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Randomization System D | | Data Displays fo | Data Displays for Reporting |
| Code | Description | Description | Order in TLF |
| Α | Placebo | Placebo | 1 |
| В | GSK2269557 12.5 mcg | NEMI 12.5 mcg | 2 |
| С | GSK2269557 25 mcg* | NEMI 25 mcg | 3 |
| D | GSK2269557 50 mcg | NEMI 50 mcg | 4 |
| Е | GSK2269557 100 mcg | NEMI 100 mcg | 5 |
| F | GSK2269557 250 mcg | NEMI 250 mcg | 6 |
| G | GSK2269557 500 mcg | NEMI 500 mcg | 7 |
| Н | GSK2269557 750 mcg | NEMI 750 mcg | 8 |

<sup>\*</sup> The nemiralisib dose of 25 mcg may be added following the results of an un-blinded interim analysis if further characterization of the lower end of the dose response curve is required.

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. NEMI 12.5 mcg vs Placebo
- 2. NEMI 25 mcg vs Placebo
- 3. NEMI 50 mcg vs Placebo
- 4. NEMI 100 mcg vs Placebo
- 5. NEMI 250 mcg vs Placebo
- 6. NEMI 500 mcg vs Placebo
- 7. NEMI 750 mcg vs Placebo

### 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Post-bronchodilator Baseline  $FEV_1$  is defined as the latest  $FEV_1$  measured prior to the first dose of study treatment and post-bronchodilator.

Pre-bronchodilator Baseline  $FEV_1$  is defined as the latest  $FEV_1$  measured prior to the first dose of study treatment and pre-bronchodilator.

Baseline CAT Total Score is defined as CAT Total Score measured prior to the first dose of study treatment on Day 1.

Baseline SGRQ Total Score is defined as SGRQ Total Score measured prior to the first dose of study treatment on Day 1.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

A centred baseline will be derived for each participant by subtracting the mean baseline across all participants from each participant's baseline value. The 'centred' baseline may be used instead of Baseline in the statistical analyses to aid convergence.

### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site and country.

# 5.4. Examination of Covariates and Subgroups

#### 5.4.1. Covariates

The list of covariates may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. The key covariates of interest are Index exacerbation severity, Smoking history and Region. Additional covariates of clinical interest may also be considered. The decision to include covariates in the model will be based on their impact on the model fit and/or convergence and will be detailed in the CSR.

A centred covariate will be derived for each participant by subtracting the mean covariate across all participants from each participant's covariate value. The 'centred' covariate may be used in place of the covariate in the statistical analyses to aid convergence.

| Covariate | Details |
|---|---|
| Index exacerbation severity | Categorical variable (Moderate or Severe) derived using the stratification variable from the randomisation system. |
| Age (at screening) | Continuous variable derived as described in Section 13.6.2.1 |
| ВМІ | Continuous variable derived using Height and Weight variables collected in eCRF: BMI = Weight (kg) / (Height (m)) <sup>2</sup> |
| Gender | Categorical variable (Male or Female), collected in eCRF |
| Country | Categorical variable |
| Region | <ul> <li>Categorical variable derived using Country as:</li> <li>Americas: Canada, Mexico, United States</li> <li>Asia: Australia, Korea</li> <li>Eastern Europe: Poland, Romania, Russia</li> <li>Western Europe: France, Germany, Italy, Netherlands, Spain, Sweden, U.K.</li> </ul> |
| Smoking history | Categorical variable (Current or Former), collected in eCRF |
| Baseline COPD maintenance therapy type | Categorical variable derived depending on data observed. Possible categories of interest are: Monotherapy vs. Dual therapy vs. Triple therapy |
| Index exacerbation type | Categorical variable: New or Relapse, derived using the question: "Other than the current prescription, for the index exacerbation, has the subject received oral/systemic corticosteroids and/or antibiotics for a COPD exacerbation within the last 7 days?" in the eCRF: New = No Relapse = Yes |
| Number of exacerbations in the previous 12 months Categorical variable derived from "Total number of COPD exacerbations in the last 12 months" in the eCRF. Possible categories of interest are: 0 vs. 1 vs. ≥2 | |
| Baseline COPD ICS therapy use | Categorical variable (ICS Use or Non-ICS Use) derived from review of concomitant medications |
| Baseline Blood Biomarker Status | Categorical variable derived from Screening time-point for the following: High sensitivity CRP • Bacterial: >10 mg/L • Non-Bacterial: ≤10 mg/L Procalcitonin • Bacterial: >0.1 µg/L • Non-Bacterial: ≤ 0.1 µg/L Eosinophils • High: ≥0.15 GI/L • Low: <0.15 GI/L |

# 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Index exacerbation severity | Moderate vs. Severe |
| Baseline COPD maintenance therapy type | Possible categories of interest are: Monotherapy vs. Dual therapy vs. Triple therapy |
| Index exacerbation type | New vs. Relapse |
| Number of exacerbations in the previous 12 months | Possible categories of interest are: 0 vs. 1 vs. ≥2 |
| Gender | Male vs. Female |
| Smoking status | Current vs. Former |
| Baseline COPD ICS therapy use | ICS Use vs. Non-ICS Use |
| Baseline Blood Biomarker Status | For High sensitivity CRP: Bacterial vs. Non-Bacterial |
| | For Procalcitonin: Bacterial vs. Non-Bacterial |
| | For Eosinophils: High vs. Low |

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 13.2 | Appendix 2: Assessment Windows |
| Section 13.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| Section 13.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 13.5 | Appendix 5: Derived and Transformed Data |
| Section 13.6 | Appendix 6: Reporting Standards for Missing Data |
| Section 13.7 | Appendix 7: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "APE" and/or "MITT" populations, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

### 6.1.1. Concomitant medications

Concomitant medications will be summarised by treatment group. Separate summaries of Baseline and On-treatment (Step-up) COPD Maintenance Therapy, and duration of OCS use will also be presented.

Additional summaries or sensitivity analyses of on-treatment COPD maintenance therapy (step-up therapy) may be performed if the data indicate that further investigation is warranted.

### 7. EFFICACY ANALYSES

Details of the outputs are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Further details for use in the endpoint derivations below can be found in Appendix 5: Derived and Transformed Data.

# 7.1. Primary Efficacy Analyses

### 7.1.1. Primary Endpoint

The primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day 84 – Post-bronchodilator Baseline  $FEV_1$ 

### 7.1.2. Primary Statistical Analyses

The primary endpoint will be analysed by fitting a suitable dose response model. The following models will be fitted, and the one that gives the best fit to the data will be selected: Bayesian 4-parameter  $E_{max}$  dose response model, 3-parameter  $E_{max}$  model and a Log-linear model.

The 4-parameter  $E_{max}$  dose response model will take the form:

Change from baseline FEV<sub>1</sub> = 
$$(E0 + a_1 * baseline) + \frac{(E_{max} + b_1 * baseline) * Dose^{\gamma}}{ED50^{\gamma} + Dose^{\gamma}}$$

The 3-parameter  $E_{max}$  dose response model will take the form:

Change from baseline 
$$FEV_1 = (E0 + a_1 *baseline) + \frac{(E_{max} + b_1 *baseline) *Dose}{ED50 + Dose}$$

Where: E0 = the response at dose = 0 (placebo)

 $E_{max}$  = the maximal response

ED50 =the dose that yields 50% of the maximal response

 $\gamma$  = the slope parameter

a<sub>1</sub>, b<sub>1</sub>, are covariates for explanatory parameters

Initially, normal non-informative priors will be used for the E0,  $a_1$ ,  $a_2$ , and  $E_{max}$  parameters with mean 0 and standard deviation 1E6 L. A functional uniform prior will be used for the ED50 and slope parameters (Bornkamp, 2014), where the prior density for the functional uniform prior is based on all the parameters in the model. An inverse -

gamma prior with shape of 0.001 and scale of 0.001 will be used for the residual variance. However, if a prior distribution appears not to be truly non-informative then alternative prior distributions may be used.

Parameters will be blocked such that the MCMC procedure samples from E0,  $a_1$ ,  $b_1$ , and  $E_{max}$ , first, then the ED50 and slope parameters and then finally the residual variance parameter. For the functional uniform priors, the density will be calculated for values of dose from 0.0001 to 750 in steps of 50 (i.e. 0.0001, 50.0001, 100.0001,..., 750.0001). For the continuous covariates, the density will be calculated from the minimum to the maximum in 10 equal steps. For binary covariates the density will be calculated for values 0 and 1. If the model does not converge including covariates, the model may be fitted with covariates removed.

If the log-linear model is fitted an offset of 1 will be used.

The posterior median change from baseline with 95% Highest Posterior Density (HPD) Credible Intervals, will be presented for each dose along with the adjusted median difference from placebo with 95% HPD, calculated at the mean baseline value across the treatment arms. Posterior probabilities that the true improvement is greater than 0 mL and 75 mL will also be presented. Graphical representation of the dose response across the full dose range will also be produced to allow inference to be made for the non-studied doses based upon the model fit.

### For the futility analysis:

The predictive probability of success at the end of the study will be calculated (assuming the randomisation ratios remain the same after the interim) for each dose using the formula suggested by Spiegelhalter, 2004 as follows:

Predictive probability = 
$$1 - \Phi \left[ \frac{\sqrt{n_1}}{\sqrt{m_1}} z_{09} - \sqrt{\frac{n_1 + m_1}{m_1}} \frac{y_n}{\sigma} \right]$$

Where  $n_1$  is the number of subjects with Day 84 data in the active arm of interest,  $m_1$  is the number of subjects yet to be observed in the active arm of interest,  $y_n$  is the posterior mean difference from placebo from the fitted model, and  $\sigma$  is the standard deviation of the posterior mean difference from placebo.

### For the possible adaptations at Interim Analysis 2:

If the study is not deemed futile, and either the 4 parameter or 3 parameter  $E_{\text{max}}$  dose response curves has successfully been fitted to the data then adaptation of the randomisation schedule will be considered, to drop, add or amend doses from the randomisation scheme.

The adaptation will be done by comparing the relative information from alternative randomisation schemes with the original randomisation schemes, such to find the design

that provides the most information about the dose response relationship. The efficiency ratio (ER) for an alternative scheme comparted to the original, will be calculated as:

$$ER(\theta_i) = \left(\frac{|M(\xi_1, \theta_i)|}{|M(\xi_F, \theta_i)|}\right)^{\frac{1}{p}}, i=1,...,1000$$

Where  $M(\xi, \theta)$  is the information matrix for the design  $\xi$  and model parameters  $\theta = (e0, emax, ed50, \gamma, a_1, b_1)^T$ ,  $\xi_1$  is the alternative design one and  $\xi_F$  is the fixed original design, and p is the number of parameters (Dette, 2008). In order to ensure any adaptation is robust to the variability in the parameter estimates at the interim analysis, 1000 samples will be generated from the posterior distribution of the parameters  $\theta_1, \dots, \theta_{1000}$  and the ER calculated for each set of parameter. Adaptation will then only take place if the median ER is >1.05 and the 10<sup>th</sup> percentile of the ER is >1. The efficiency ratio will be estimated using the mean baseline value across the population.

The alternative designs that will be considered will depend on the dose response model fitted but could include:

- 1. Add 25mcg dose
- 2. Add 25mcg dose, drop 500mcg dose
- 3. Add 25mcg dose, drop 250 mcg and 500 mcg doses
- 4. Drop 12.5mcg dose
- 5. Drop 12.5 mcg and 50mcg doses

The potential adaption may also be verified in the moderate and severe subgroups to ensure the adaption is beneficial across both groups.

### 7.1.2.1. Model Checking & Diagnostics

The following list of convergence diagnostics will be applied for each parameter:

- The Monte Carlo Standard Errors (MCSE) should be compared with the standard deviation (SD) of the posterior distribution to ensure that only a fraction of the posterior variability is due to the simulation. The number of samples generated and/or the thinning may be increased to reduce the ratio of the MCSE/SD as deemed necessary.
- The Geweke diagnostic test will be used to assess whether the mean estimates have converged by comparing means from the early and latter part of the Markov chain using a z-score t-test. Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.
- Trace plots of samples versus the simulation index will be visually inspected to assess some aspects of convergence. The centre of the chain should appear stable with very small fluctuations, i.e., the distribution of points should not change as the chain progresses and the posterior mean and variance are relatively constant.
- Autocorrelation plots will be visually inspected to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).

## 7.1.3. Sensitivity and Supportive Analyses

If there are greater than 20% of participants with an important protocol deviation that results in exclusion from the Per Protocol Population, the primary analysis may be repeated using the Per Protocol Population.

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 will also be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant. All post-baseline scheduled visits will be included in the analysis using Day. Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

A further sensitivity analysis may be performed where Baseline  $FEV_1$  is replaced with the  $FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge for participants who were hospitalised for their index exacerbation, i.e. who were randomized with a Severe index exacerbation but kept as Baseline  $FEV_1$  for participants who were randomized with a Moderate index exacerbation.

### 7.1.4. Subgroup Analyses

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will be performed by fitting separate models to each level of the severity subgroup.

A subgroup analysis of change from baseline in clinic visit trough  $FEV_1$  by index exacerbation severity will also be performed by including a treatment-by-severity-by-Day interaction term in the Bayesian Repeated Measures model.

# 7.2. Secondary Efficacy Analyses

### 7.2.1. Rate of exacerbations

Rate of exacerbation is defined as the frequency of exacerbations (subsequent to the index exacerbation) within the specified time period, for example, the 12-Week Treatment Period or the 24-Week Study Period.

The length of time on treatment or in study, depending on the specified time-period, for each participant will be calculated for each endpoint as follows:

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| Rate of (on-treatment) exacerbations, summarised by: | 12-Week Treatment Period | Time from date of randomisation to date of last dose of study |
| Moderate/severe exacerbations | | treatment |
| Moderate exacerbations | | |
| Severe exacerbations | | |
| All (mild, moderate and | | |

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| severe) exacerbations | | |
| Rate of (on-or off-treatment) exacerbations, summarised by: | 12-Week Treatment Period | Time from date of randomisation to Day 84 (Visit 6) Visit Date. |
| <ul><li>Moderate/severe exacerbations</li><li>All exacerbations</li></ul> | | For participants who withdraw early from the study: Time from date of randomisation to date of study withdrawal |
| Rate of (off-treatment) exacerbations, summarised by: • Moderate/severe exacerbations • Moderate exacerbations • Severe exacerbations | 12-Week Follow Up Period | Time from date of last dose of study treatment to date of study withdrawal/completion |
| Rate of (on- and off- treatment) exacerbations, summarised by: • Moderate/severe exacerbations • Moderate exacerbations • Severe exacerbations | Full 24-Week Study Period | Time from date of randomisation to date of study withdrawal/completion |

Refer to Section 13.5 for further details regarding the length of time derivation

### 7.2.1.1. Statistical analyses

The rate of exacerbations will be analysed using a Bayesian generalized linear model assuming a negative binomial distribution for the underlying exacerbation rate with a log link function. An offset to account for the length of time on treatment or in study, depending on the specified time-period, for each participant (as described above) will be included in the model as  $\log_e$  (length of time).

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The median exacerbation rates for each dose arm per 12 weeks, along with the median ratio in exacerbation rates (nemiralisib/placebo) per 12 weeks for each dose, will be estimated and corresponding 95% HPD credible intervals presented. The probability that the true exacerbation rate ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore estimates of the exacerbation rates for pooled data from 500 mcg plus 750 mcg will also be presented.

### 7.2.1.2. Subgroup analyses

A subgroup analysis of exacerbation rate by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

### 7.2.1.3. Exploratory analyses

A summary of exacerbation rate by the following groups will be presented and, if feasible, a subgroup analyses may be performed:

- Index exacerbation type (New or Relapse)
- Number of exacerbations in previous 12 months  $(0, 1 \text{ or } \ge 2)$ .

### 7.2.2. Time to next exacerbation

Time to next (on-treatment) exacerbation following index exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation whilst on study treatment. Participants who did not have an exacerbation whilst on study treatment will be censored at the date of their last dose of study treatment.

Time to next (on-or off-treatment) exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation occurring up to Day 84. Participants who have not had an exacerbation during the 12-Week Treatment Period will be censored at Day 84 or the date of study withdrawal, for participants who withdrew from the study prior to Day 84.

Time to next exacerbation following cessation of study treatment is defined as time from the date of last dose of study treatment until the date of onset of the next exacerbation whilst off study treatment during the 12-Week Follow Up Period. Participants who have not had an exacerbation off-treatment will be censored at the date of their last follow up assessment.

Time to next exacerbation will be analysed by severity, as follows:

| Endpoint | Time period |
|---|---|
| Time to next (on-treatment) exacerbation, summarised by: | 12-Week Treatment Period |
| Moderate/severe exacerbations | |
| All (mild, moderate and severe) exacerbations | |
| Time to next (on-or off-treatment) exacerbation, summarised by: • Moderate/severe exacerbations • All exacerbations | 12-Week Treatment Period |
| Time to next exacerbation following cessation of treatment, summarised by: Moderate/severe exacerbations | 12-Week Follow Up Period |

Refer to Section 13.5 for further details regarding the length of time derivation

### 7.2.2.1. Statistical analyses

Time to next exacerbation will be analysed using a Bayesian Cox proportional hazards model with the "Efron" method for handling ties.

Kaplan-Meier (KM) estimates of the probability of exacerbation will also be presented.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The hazard ratio and corresponding 95% HPD credible intervals for each nemiralisib dose versus placebo will be presented. The probability that the true hazard ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore an estimate of hazard ratio for pooled data from 500 mcg plus 750 mcg nemiralisib doses versus placebo will also be presented.

### 7.2.2.2. Subgroup analyses

A subgroup analysis of time to exacerbation by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

## 7.2.3. Change from baseline in Clinic Visit trough FEV<sub>1</sub>

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56 measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day X – Post-bronchodilator Baseline  $FEV_1$ 

Where Day X is Day 14, 28, and 56.

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56, 84 measured prebronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day X – Pre-bronchodilator Baseline  $FEV_1$ 

Where Day X is Day 14, 28, 56, and 84.

### 7.2.3.1. Statistical Analyses

Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured post-bronchodilator will be analysed using a dose response model and repeated measures analysis as described for the primary endpoint in Section 7.1.2.

Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured pre-bronchodilator will be analysed using a repeated measures analysis as described in Section 7.1.2

### 7.2.3.2. Subgroup analyses

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will be performed.

## 7.2.4. Change from hospital discharge in clinic visit trough FEV<sub>1</sub>

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> will be derived only for participants who were hospitalised for their index exacerbation and who have been subsequently discharged.

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day  $X - FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day  $X - FEV_1$  measured prior to dosing and post-bronchodilator on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Note, as per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the FEV<sub>1</sub> assessment will be assigned the hospital discharge assessment and the Day 14 assessment will be missing. Refer to Section 13.2.1.1 for further details.

In addition, if discharge takes place after Day 14, the Day 14 assessment will be missing for this analysis.

### 7.2.4.1. Statistical analyses

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> will be analysed using a repeated measures analysis as described in Section 7.1.2 if there are a sufficient number of participants to provide a meaningful analysis, otherwise the data will be summarised.

# 7.2.5. EXAcerbations of Chronic Pulmonary Disease Tool - Patient Reported Outcome (EXACT)

The EXACT is a 14-item daily diary designed to provide a measure of patient-reported symptoms of COPD exacerbation. An EXACT Total Score, ranging from 0 to 100, where

higher scores indicate a more severe condition, will be derived for each day of diary collection according to the instructions in the EXACT User Manual (Version 8.0, Evidera, 2016).

The electronic EXACT diary does not allow a study patient to skip individual items, therefore no missing data are expected for individual items. However, if missing values occur for individual items, the Total Score that contains the item will be set to missing for that day. Moderate-to-severe COPD patients are expected to experience symptom(s) each day, and a score of zero on all 14 EXACT items is likely to represent a situation where in order to complete the diary quickly, the respondent did not accurately report their daily symptom(s), therefore if the EXACT Total Score is 0, it will be set to missing.

A 3-day Rolling Average EXACT Total Score will be calculated for each day, X, as:

(EXACT Total Score on Day X-1 + EXACT Total Score on Day X + EXACT Total Score on Day X+1) / (Number of days with non-missing values)

Note, for Day 1, the Rolling Average EXACT Total Score will be calculated as the average of EXACT Total Score on Days 1 (Randomisation) and 2 only, since no EXACT data is collected prior to randomisation. Similarly, the Rolling Average EXACT Total Score for the last study day will be calculated as the average of EXACT Total Score on the last day and on the day before the last day.

The Rolling Average EXACT Total Score will be calculated for each day as long as at least 1 EXACT total score in the sequence is present. Therefore, only in the case where EXACT total scores are missing for 3 consecutive days in a row (or 2 consecutive days in the case of the first and last day rolling average calculation), will the rolling average score be missing.

The Maximum Observed Value (MOV) is defined as the highest Rolling Average EXACT Total Score observed within the first 14 days of randomisation. Note: this definition differs from the definition in the EXACT User Manual of "the highest rolling average EXACT score observed in the context of an EXACT exacerbation within the first 14 days of the exacerbation", since the date of the index exacerbation is likely to be prior to randomisation.

# 7.2.5.1. Proportion of participants achieving EXACT-defined recovery from index exacerbation

EXACT-defined recovery from the index exacerbation is defined as a decrease in the Rolling Average EXACT Total Score  $\geq 9$  points from the Maximum Observed Value, sustained for  $\geq 7$  days, with the first of the 7 days defined as the recovery day.

The proportion of participants achieving EXACT-defined recovery from the index exacerbation by Days 14, 28, 56, and 84 will be calculated as:

(Number of participants who experience an EXACT-defined recovery on or before Day X) / (Total number of participants in the MITT population)

Where Day X is 14, 28, 56, and 84.

### 7.2.5.2. Time to EXACT-defined recovery from index exacerbation

Time to EXACT-defined recovery from index exacerbation is defined as time from the date of randomisation until date of the first EXACT-defined recovery day during the 12-Week Treatment Period, where EXACT-defined recovery is described in Section 7.2.5.1. Participants who did not experience EXACT-defined recovery during the 12-Week Treatment Period will be censored at the date of their last dose of study treatment.

# 7.2.5.3. Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT is defined as the highest EXACT Total Score (not using the 3-day Rolling Average) during the period from date of onset of the subsequent HCRU-exacerbation until date of EXACT-defined recovery of subsequent exacerbation.

Note, in this case, the Maximum Observed Value and EXACT-defined recovery are derived using the date of onset of the subsequent HCRU-exacerbation.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will only be derived for participants who have had a subsequent exacerbation. If a participant has more than one subsequent exacerbation, severity will be calculated for each subsequent exacerbation.

### 7.2.5.4. Statistical analyses

The proportion of participants achieving EXACT-defined recovery from the index exacerbation will be analysed using a Bayesian logistic regression model. Separate models will be fitted for each time-point.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The results of the analysis will be presented in terms of odds ratios together with its associated 95% HPD credible interval. The probability that the true odds ratio is greater than 1, in addition to other values appropriately selected based on the data, will be presented.

Time to EXACT-defined recovery from index exacerbation will be analysed using the same techniques as described in Section 7.2.2.1.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will be summarised for each treatment group and reported by study period. The severity of subsequent HCRU-defined exacerbation(s) occurring whilst a participant is on treatment will be reported as during the 12-Week Treatment Period and the severity of subsequent HCRU-defined exacerbation(s) occurring after the last dose of study treatment will be reported as during the 12-Week Follow-up Period.

## 7.2.5.5. Subgroup analyses

A subgroup analysis of the proportion of participants achieving EXACT-defined recovery from the index exacerbation by Index Exacerbation Severity will be performed by including a treatment-by-severity term in the model.

### 7.2.5.6. Sensitivity and supportive analyses

Sensitivity analyses exploring the impact of any missing data, and changes to the definition of EXACT-defined recovery may be conducted and may be performed post-SAC.

# 7.2.6. COPD Assessment Test (CAT)

The COPD Assessment Test (CAT) is a patient completed questionnaire developed to measure the health status of patients with COPD. The CAT consists of eight items, each on a six-point scale: 0 (no impact) to 5 (high impact). The CAT Score will be calculated for each study day of collection by summing the scores for all questions. The CAT Score ranges from 0 to 40, where higher scores indicate a more severe condition.

### 7.2.6.1. Proportion of responders using the CAT

The proportion of responders using the CAT will only be derived for participants with a baseline CAT Total Score  $\geq 2$ .

The Proportion of responders using the CAT is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq 2$  on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84 and the study day following EXACT-defined recovery from the index exacerbation. See Section 13.2.1.2 for details for cases where the study day following EXACT-defined recovery occurs within a scheduled assessment window.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

### Exploratory – Follow-Up Period

The Proportion of responders using the CAT at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq 2$  on or before Day X)/(Total number of participants in the MITT population)

Where Day X is Day 112 and Day 168 and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

### 7.2.6.2. Change from baseline in CAT Total Score

Change from baseline in CAT Total Score is defined as:

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is 28, 56, 84 and the study day following EXACT defined recovery from the index exacerbation. See Section 13.2.1.2 for details for cases where the study day following EXACT-defined recovery occurs within a scheduled assessment window.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

### Exploratory – Follow-Up Period

The Change from baseline in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is Day 112 and Day 168.

The Change from end of treatment in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – CAT Total Score on Day 84

Where Day X is Day 112 and Day 168.

### 7.2.6.3. Statistical analyses

The proportion of responders using CAT will be analysed using the same techniques as described in Section 7.2.5.4.

Change from baseline/end of treatment in CAT Total Score will be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant.

All post-baseline scheduled visits will be included in the analysis using Day.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

Adjusted posterior median change from baseline and corresponding 95% HPD credible intervals will be summarised for each treatment by time-point, together with estimated treatment differences (GSK – Placebo) and corresponding 95% HPD credible intervals. The posterior probability that the true treatment difference is less than 0, in addition to other values appropriately selected based on the data, will also be presented.

## 7.2.6.4. Subgroup analyses

A subgroup analysis of the proportion of responders using CAT and the change from baseline in CAT Total Score by Index exacerbation severity will be performed by including a treatment-by-severity term and a treatment-by-severity-by-Day term in the Bayesian logistic regression and Bayesian Repeated Measures models, respectively.

# 7.2.7. St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)

St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) is a 40-item questionnaire designed specifically to focus on COPD patients. SGRQ-C will be scored to be equivalent to the SGRQ Total Score, ranging from 0 to 100, where higher scores reflect worse health-related quality of life. SGRQ Total Scores will be calculated for each day of collection according to the instructions in SGRQ-C Manual (Version 1.3, March 2016).

### 7.2.7.1. Proportion of responders on the SGRQ Total Score

The proportion of responders on the SGRQ Total Score will only be derived for participants with a baseline SGRQ Total Score ≥4.

Proportion of responders on the SGRQ Total Score is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84.

### Exploratory – Follow-Up Period

The Proportion of responders on the SGRQ Total Score at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is Day 112 and Day 168 and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

### 7.2.7.2. Change from baseline in SGRQ Total Score

Change from baseline in SGRQ Total Score is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is Day 28, 56, and 84.

### Exploratory – Follow-Up Period

The Change from baseline in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is Day 112 and Day 168.

The Change from end of treatment in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – SGRQ Total Score on Day 84

Where Day X is Day 112 and Day 168.

### 7.2.7.3. Statistical analyses

Change from baseline/end of treatment in SGRQ Total Score and the proportion of responders on the SGRQ Total Score will be analysed using the same techniques as described in Section 7.2.6.3.

### 7.2.7.4. Subgroup analyses

Subgroup analyses of change from baseline in SGRQ Total Score and the proportion of responders on the SGRQ Total Score by Index exacerbation severity will be conducted as described in Section 7.2.6.4.

### 7.2.8. Rescue medication use

All participants will record rescue medication use in the eDiary. Rescue medication use will be recorded as the number of occasions of rescue medication use each day.

The Mean Number of Occasions of Rescue Medication Use Per Day is defined as:

(Sum of the number of occasions of rescue medication use each day within the time-period) / (Total number of days with non-missing values within the time-period)

The Percentage of Rescue-Free Days is defined as:

(Sum of the number of days where the number of occasions of rescue medication use is zero within the time-period) / (Total number of days with non-missing values within the time-period)\*100

Where the time-period is defined as follows:

Week 1 of the 12-Week Treatment Period: Day 1 to Day 7

Week 2 of the 12-Week Treatment Period: Day 8 to Day 14

Week 3 of the 12-Week Treatment Period: Day 15 to Day 21

Week 4 of the 12-Week Treatment Period: Day 22 to Day 28

Week 5 of the 12-Week Treatment Period: Day 29 to Day 35

Week 6 of the 12-Week Treatment Period: Day 36 to Day 42

Week 7 of the 12-Week Treatment Period: Day 43 to Day 49

Week 8 of the 12-Week Treatment Period: Day 50 to Day 56

Week 9 of the 12-Week Treatment Period: Day 57 to Day 63

Week 10 of the 12-Week Treatment Period: Day 64 to Day 70

Week 11 of the 12-Week Treatment Period: Day 71 to Day 77

Week 12 of the 12-Week Treatment Period: Day 78 to Day of last dose

Over the 12-Week Treatment Period: Day 1 to Day of last dose.

### Exploratory – Follow-Up Period

Rescue medication use up to Day 112 will also be summarised by including the timeperiods:

Week 13 (Follow-up Period): (Day of last dose + 1) to (Day of last dose + 1) + 6 days

Week 14 (Follow-up Period): (Day of last dose + 7) to (Day of last dose + 1) + 13 days

Week 15 (Follow-up Period): (Day of last dose + 14) to (Day of last dose + 1) + 20 days

Week 16 (Follow-up Period): (Day of last dose +21) to (Day of last dose +1) +27 days

For a subject to be counted in the time periods for rescue medication use, they must have at least one eDiary entry recorded during that time period.

### 7.2.8.1. Rescue medication use via the clip-on Propeller Sensor for MDI

A subset of participants from countries where the Propeller Sensor for MDI is available will also record rescue medication use via the clip-on Propeller Sensor for MDI. A supportive summary of rescue medication use via the clip-on Propeller Sensor for MDI for these participants will be presented.

Rescue medication use via the clip-on Propeller Sensor for MDI is defined in the same way as rescue medication use via the eDiary, except that the number of actuations will be used instead of the number of occasions in accordance with the way the data is captured.

### 7.2.8.2. Statistical analyses

The Mean Number of (on-treatment) Occasions of Rescue Medication Use Per Day will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

The Percentage of (on-treatment) Rescue-Free Days will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

Rescue medication use via the clip-on Propeller Sensor for MDI will be summarised in the same way as rescue medication use via the eDiary.

# 7.3. Exploratory Efficacy Analyses

## 7.3.1. Change from Day 84 in Clinic Visit trough FEV<sub>1</sub>

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day X – Day 84 post-bronchodilator  $FEV_1$ 

Where Day X is Day112, Day 140 and Day 168.

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day X – Day 84 pre-bronchodilator  $FEV_1$ 

Where Day X is Day 112, Day 140 and Day 168.

Participants who discontinue study treatment prior to Day 84 will be excluded from this analysis.

### 7.3.1.1. Statistical analysis

Change from Day 84 in Clinic Visit trough FEV<sub>1</sub> will be analysed using the same techniques as described for Change from baseline in CAT Total Score in Section 7.2.6.3.

A subgroup analysis of change from Day 84 in FEV<sub>1</sub> will be performed by including a treatment-by-severity-by-Day term in the Bayesian Repeated Measures model.

### 7.3.2. E-RS:COPD (Evaluating Respiratory Symptoms in COPD)

Change from baseline in E-RS: COPD and subscales will be summarised by treatment group. Exploratory analyses related to E-RS: COPD and subscales may be performed post SAC.

# 7.3.3. Measures of HCRU related to exacerbations

Unscheduled Healthcare Utilisation will be summarised separately for exacerbation-related, COPD-related or non-COPD related; each summary will be presented by all patients (i.e. moderate and severe index exacerbation combined), and separately by index exacerbation severity.

The number of days of hospital admission for the index and subsequent exacerbations will also be summarised by treatment group.
#### 7.3.3.1. Re-hospitalisation within 30 days of index exacerbation

Re-hospitalisation within 30 days of index exacerbation is defined as 30 days from the date of hospital discharge until the date of next hospital admission (+ 1 day, to account for study day derivation), for participants who were hospitalised for their index exacerbation.

Exacerbation-related, COPD-related and Non-COPD-related hospital admissions are collected in separate eCRFs. The date of hospital admission is not collected in the COPD-related eCRF, therefore the date of next hospital admission will be estimated using the earliest of:

- Date of hospital admission for exacerbation-related hospitalisations
- Date of contact for COPD-related hospitalisations, where the number of inpatient hospitalisation days >0
- Date of hospital admission for non-COPD-related hospitalisations.

The proportion of participants who were re-hospitalised within 30 days of the index exacerbation will be summarised by each treatment arm.

#### 7.3.3.2. Time from resolution of index exacerbation to next exacerbation

Time from resolution of index exacerbation to next exacerbation is defined as time from the date of (Investigator-defined) resolution of index exacerbation until the date of onset of the subsequent exacerbation.

A summary of time from resolution of index exacerbation to next exacerbation will be presented. Participants who did not have a subsequent exacerbation or for whom the index exacerbation was not resolved will be excluded from the summary.

Time from resolution of index exacerbation to next exacerbation will only be derived for the first subsequent exacerbation following the index exacerbation.

#### 7.3.3.3. Subsequent exacerbation treatment type

A summary of the type of treatment for subsequent exacerbations (OCS, antibiotics, or both) may also be presented.

#### 7.3.4. Compliance

Compliance with study treatment for all participants is captured from the dose counter on the ELLIPTA and the overall percentage compliance will be summarised by each treatment group.

Reported compliance with study treatment is also captured daily in the eDiary from the question "Did you take this morning's dose of study medication"?

The percentage of reported compliance for each participant is calculated as:

(Sum of the number of days where the question was answered with 'Y') / (Number of days from first dose of study treatment to last dose of study treatment) x 100

Overall percentage of reported compliance will also be summarised by each treatment group.

# 7.3.4.1. Number of actuations of double-blind study treatment measured by the clip-on Propeller Sensor

Percentage compliance via the clip-on Propeller Sensor for ELLIPTA in the subset of participants from countries where the Propeller Sensor for ELLIPTA is available is calculated as:

(Sum of the number of days with actuation > 0) / (Number of days from first dose of study treatment to last dose of study treatment) x 100

Overall percentage compliance will be summarised by each treatment group.

#### 7.3.4.2. Missing EXACT-PRO data

Missing EXACT-PRO data will be summarised by treatment group.

# 7.3.5. Inflammatory/infective markers in blood and sputum in relation to acute exacerbation of COPD

Results of the analysis of blood/spontaneous sputum samples of eosinophil counts and inflammatory/infective mediators/markers will be summarised by treatment group.

Further analyses of inflammatory/infective markers may be performed, for example split by CRP high, CRP low, Procalcitonin high, etc. categories.

#### 7.3.6. Other spirometry measurements

Percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio will be summarised by treatment group.

#### 7.3.7. Other symptoms suggestive of exacerbation

Responses to questions in the eDiary related to symptoms of sputum purulence (colour), fever, sore throat, wheezing and colds collected in the eDiary will be listed by treatment group.

# 7.3.8. Classification of exacerbating COPD participants and prediction of response to nemiralisib using machine learning techniques

Exploratory analysis of endpoints using machine learning techniques will be performed which will include classification of COPD participants, identification of parameters which describe a responder, and prediction of response to nemiralisib using baseline data. Details of these analyses will be described in a separate RAP and results may be reported separately to the CSR.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. The details of the planned displays will be provided in Appendix 11: List of Data Displays.

#### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards.

### 8.1.1. Adverse Events of Special Interest

Adverse events of special interest (AESI) are significant identified or potential risks identified in the nemiralisib clinical development programme.

#### 8.1.1.1. Post-inhalation Cough Immediately Following Dosing

Post-inhalation cough immediately following dosing is an AESI and will be evaluated during study Visits 2-6 in the 12-Week Double-Blind Treatment Period. Investigators (or medically qualified designees) will monitor participants for potential study treatment tolerability issues, including post-inhalation cough, within 5 minutes immediately following dosing.

The percentage of patients experiencing post-inhalation cough following dosing, regardless of whether it was also reported as an AE, overall and by each visit will be summarised for each treatment group. The type of cough, time to onset and duration of cough, and severity will also be summarised.

In addition, any post-inhalation cough immediately following dosing reported as an adverse event during the clinic visit observation or during the course of the study will be summarised by treatment group.

#### 8.1.1.2. Paradoxical bronchospasm

Paradoxical bronchospasm is an AESI, defined using the Preferred Terms Bronchospasm and Bronchospasm paradoxical and will be summarised by treatment group.

## 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and liver function tests will be based on GSK Core Data Standards.

# 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

# 8.4. Mortality

A summary of all-cause mortality by treatment will be presented.

## 9. PHARMACOKINETIC ANALYSES

### 9.1. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 9.2. Drug Concentration Measures

Plasma nemiralisib concentrations of GSK2269557 will be listed and summarised by dose, day and time. Drug levels will be summarised by day (14, 28), dose and time intervals (trough, 0-<1h, 1-6h).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 13.4.3 Reporting Standards for Pharmacokinetic).

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

#### 10. POPULATION PK ANALYSIS

A dataset for population PK analysis will be provided by Statistics and Programming based on the NONMEM data specifications in Section 13.8.2.

Conduct of the population PK analyses will be based on the current guidance which contains specific recommendations for working practices, processes and standards for population PK and PK/PD analysis conducted by Clinical Pharmacology Modelling and Simulation (CPMS) [Analysis & Reporting, 2017].

The sparse PK samples will be subjected to a validated population PK model for nemiralisib currently under development.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR. Analyses and reporting of the population PK model will be in accordance with the FDA and EMEA guidance on population PK, PK-PD analyses.

#### 10.1. Derived Pharmacokinetic Parameters

The exposure parameters (e.g. AUC,  $C_{max}$ ) will be derived from the individual post-hoc estimates from the POP PK model. These will be summarized across dose treatments, subgroups (e.g., gender, race) or as a function of a continuous variable (e.g., age).

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

If statistical analyses suggest an effect of nemiralisib on primary and other key clinical endpoints, an integrated longitudinal population dose/exposure versus clinical response on analysis key parameters including FEV<sub>1</sub> and exacerbation rate will be undertaken. Participant characteristics influencing the relationship will be evaluated.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

## 12. REFERENCES

Bornkamp, B. (2014). Practical considerations for using functional uniform prior distributions for dose-response estimation in clinical trials. Biometrical Journal, 56(6), 947-962. doi: 10.1002/bimj.201300138.

Dette, H., Bretz, F., Pepelyshev, A. & Pinheiro, J., (2008). Optimal Designs for Dose-Finding Studies. Journal of the American Statistical Association, 103:483, 1255-1237. doi: 10.1198/016214508000000427.

Evidera. (2016). The Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Patient-Reported Outcome (PRO) USER MANUAL (Version 8.0).

Spiegelhalter, D.J., Abrams, K.R. & Myles, J.P., (2004). Bayesian Approaches to Clinical Trials and Health-Care Evaluation. John Wiley & Sons, Ltd.

#### 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 13.1.1. Exclusions from Per Protocol Population

Protocol deviations will be reviewed regularly throughout the course of the study, as described in Protocol Deviation Management Plan (PDMP). Deviations which will result in exclusion from the Per Protocol population will be assigned on a case-by-case basis prior to database freeze (DBF).

Decisions on whether or not the subject should be excluded from the PP population because the incorrect treatment was taken, due to the incorrect container being dispensed, will be identified after unblinding (i.e. post DBF). A PD of "incorrect treatment" will be added to the reporting dataset.

#### 13.2. Appendix 2: Assessment Windows

#### 13.2.1. Definitions of Assessment Windows for Analyses

#### 13.2.1.1. Hospital discharge

As per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the FEV<sub>1</sub> assessment will be assigned the hospital discharge FEV<sub>1</sub> assessment and the Day 14 assessment will be missing.

For all other analyses and summaries that include participants who were hospitalised for their index exacerbation, an additional Analysis Timepoint of "HOSPTIAL DISCHARGE" will be derived. However, in the cases where discharge takes place between Day 11 and Day 17 (inclusive), participants will be summarised under DAY 14 and a footnote to say that participants who were discharged at Day 14 are summarised under DAY 14 will be included.

#### 13.2.1.2. EXACT-Defined Recovery for CAT Trigger

If the study day following EXACT-defined recovery for a participant occurs within a scheduled assessment window, an additional analysis time-point will be programmatically created for that scheduled visit. For example, if EXACT-defined recovery occurred on Day 56, then a Day 56 Visit will be programmatically created with the data from the Recovery visit so that it can be summarised/analysed in both the Visit and Recovery categories.

Due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery from the index exacerbation is not derived according to the EXACT User Manual. Instead, it has been derived using a 3-day Rolling Average that is calculated as the mean EXACT score [Day X-2, Day X-1, Day X].

# 13.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

#### 13.3.1. Study Periods

#### 13.3.1.1. 12-Week Treatment Period

The 12-Week Treatment Period is assigned from Study Day 1 to Study Day 84.

#### 13.3.1.2. 12-Week Follow-Up Period

The 12-Week Follow-up Period is assigned from Study Day 85 to Study Day 168.

#### 13.3.2. Study Phases

Exacerbation events during the 12-Week Treatment Period will be classified according to their occurrence from randomisation until treatment discontinuation/study withdrawal days, as detailed below.

| Study Phase | Occurring from randomisation until |
|---|---|
| On-Treatment during the 12-Week Treatment Period | Treatment Stop Day |
| On- or Off-Treatment during the 12-Week Treatment | Day 84 or Study Withdrawal Day if Treatment Stop |
| Period | Day is < Day 84 |

#### 13.3.2.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before Randomisation Date |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 13.3.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop |
| Emergent | date plus 10 days. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 13.4. Appendix 4: Data Display Standards & Handling Conventions

#### 13.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | HARP Compound : \arprod\gsk2269557\mid200879 |
| Analysis Datasets | |
| For all interim analyses, except for the End of Treatment Interim Analysis, datasets will be created according to Legacy GSK A&R dataset standards. | |

For the End of Treatment Interim Analysis and the final reporting effort, datasets will be created

# Generation of RTF Files

RTF files will be generated for the final reporting effort.

#### 13.4.2. Reporting Standards

according to current CDISC standards

#### General

0 - 64----

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Figures will be produced using PROC SGPLOT in SAS

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places.
- For lab parameters results that contain a character value of '<', or '>', e.g. '<X' or '>X', the parameter value will be imputed with X.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits will be included in summary tables of the worst-case results by potential clinical<br/>importance criteria only.</li> </ul> | |
| All unscheduled vi | sits will be included in listings. |
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

# 13.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 13.8.2 Population Pharmacokinetic (PopPK) Dataset Specification. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in the CPMS RAP. |

#### 13.5. Appendix 5: Derived and Transformed Data

#### 13.5.1. **General**

#### **Multiple Measurements at One Analysis Time Point**

 Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Randomisation Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### Time from date of randomisation and time from date of last dose of study treatment

- For endpoints that use the time from the date of randomisation to a reference date, time will be calculated as
  - (Ref Date Randomisation Date) + 1
- For endpoints that use the time from the date of last dose of study treatment to a reference date, time will be calculated as
  - (Ref Date (Last Dose Date + 1)) +1

### 13.5.2. Study Population

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:
 Duration of Exposure in Days = Treatment Stop Date – (Treatment Start Date) + 1

#### 13.5.3. Safety

#### **Adverse Events**

#### **AE'S of Special Interest**

- Post-inhalation cough: Lower level term (LLT) to be included is "coughing after drug inhalation"
- Paradoxical bronchospasm: Preferred Terms to be included are "Bronchospasm paradoxical" and "Bronchospasm"

# 13.6. Appendix 6: Reporting Standards for Missing Data

## 13.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) is defined as completing all phases of the study including the last scheduled study visit |
| | A participant is considered to have completed the Treatment Period, if he/she has completed the last on-treatment study visit (Visit 6) |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will not be summarised (and will be listed only). |

# 13.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 13.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Age | <ul> <li>The eCRF collects year of birth only. Day and Month will be imputed by Data Management using a PPD for the day and PPD for the month</li> <li>Age will then be derived referenced to the Screening Date</li> <li>A footnote to say that age has been imputed will be included in any outputs containing age.</li> </ul> |

# 13.7. Appendix 7: Values of Potential Clinical Importance

# 13.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male 18-64 years | 7.1 | 19.9 |
| Hoomoglobin | G/DL | Male 65+ years | 7.1 | 19.9 |
| Haemoglobin | | Female 18-64 years | 7.1 | 19.9 |
| | | Female 65+ years | 7.1 | 19.9 |
| Lymphocytes | GI/L | | 0.85 | 4.1 |
| Total Absolute Neutrophil Count | GI/L | | 1.5 | 8 |
| Platelet Count | GI/L | | 31 | 1499 |
| White Blood Cell count | GI/L | 18-64 years | 1.1 | 10.8 |
| Write blood Cell Courit | | 65+ years | 1.1 | 10.8 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 32 | 50 |
| Calcium | mmol/L | | 1.5 | 3.24 |
| | | Male 40-49 years | 69 | 160 |
| | | Male 50-59 years | 67.2 | 160 |
| | | Male 60-69 years | 67.2 | 160 |
| Creatinine | | Male 70+ years | 59.2 | 160 |
| Creatifile | | Female 40-49 years | 52.2 | 160 |
| | | Female 50-59 years | 53 | 160 |
| | | Female 60-69 years | 53 | 160 |
| | | Female 70+ years | 55.7 | 160 |
| | mmol/L | 13-49 years | 2.2 | 27.8 |
| Glucose | IIIIIIOI/L | 50+ years | 2.2 | 27.8 |
| Potassium | mmol/L | | 2.8 | 6.5 |
| Sodium | mmol/L | | 120 | 160 |
| | mmol/L | 13-64 years | 2.5 | 15 |
| Urea/BUN | IIIIIOI/L | 65+ years | 2.5 | 15 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 2x ULN |
| | µmol/L | | 2xULN T.Bilirubin + ≥ 3x ULN ALT |
| T. Bilirubin + ALT | | High | |
| | U/L | _ | |
| Direct Bilirubin | µmol/L | | 0 – 6 |

# 13.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 530 |
| Absolute PR Interval | msec | < 110 | > 240 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc mse | | | > 60 |

# 13.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 95 | > 160 |
| Diastolic Blood Pressure | mmHg | < 55 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

### 13.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

#### 13.8.1. Population Pharmacokinetic (PopPK) Methodology

All analysis will be performed in the validated Modelling and Analysis Platform (MAP). MAP consists of a Linux desktop containing various modelling applications, including NONMEM, PsN, Pirana, R and RStudio. All software versions used will be documented.

The population PK analysis will be performed in the following sequence of steps:

- 1. Exploratory data analysis/data check out.
- 2. Base structural model development.
- 3. Covariate analysis.
- 4. Model refinement.
- 5. Model evaluation.
- 6. Model application using simulation

The above analysis and reporting steps follow EMEA

(http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC500003067.pdf) and FDA population PK guidances (https://www.fda.gov/downloads/drugs/guidances/UCM072137.pdf)

Key components of these regulatory guidelines on population PK are also included in the Global CPMS guidance for pop pk RAP (https://connect.gsk.com/sites/cpms/TandD/Guidances).

#### 13.8.2. Population Pharmacokinetic (PopPK) Dataset Specification

Statistics & Programming, in discussion with CPMS, will provide a NONMEM dataset.

Column headings in NONMEM-ready datasets and specifications should be consistent to minimise the programming process, and facilitate a smooth transfer of projects between users as needed. IDSL standards will be followed where possible.

A list of most common standardised variable names for NONMEM datasets can be found in Table below.

## List of Variable Names for NONMEM-Ready Datasets for PopPK Analysis

| DNMEM line exclusion identifier DNMEM subject identifier udy ID |
|------------------------------------------------------------------|
| ıdy ID |
| bject identifier for study |
| ique identifier for a study site |
| NMEM Amount of drug administered then EVID =1- dose event record |
| it of AMT (mg) |
| NMEM Additional dose |
| ug Concentration |
| it of CONC (ng/mL) |
| tural log of CONC column |
| ug label e.g 557 |
| wer Limit of quantification |
| tural log of LLQ column |
| ldy day number of record or of dosing |
| sma sample time after last dose |
| it of TIME (h) |
| se amount |
| NMEM Event ID If row has dose then EVID=1 else EVID =0 |
| EVID=1 then this is a dose event record |
| EVID = 0 then this is an observation record |
| NMEM Inter-dose interval II=24 – dose every day |
| eady state item SS= 1 refers to steady state |
| NMEM Missing data value then MDV=1 else MDV=0 |
| bject Age (yrs) |
| bject gender 0 = Male 1 =Female |
| bject gender text Male or Female |
| seline Body Mass Index |
| seline Subject weight |
| entifier for inhibitor CYP3A4 1 =Yes, 0 = No |
| ibitor Name |
| entifier for inducer CYP3A4 1 =Yes, 0 = No |
| lucer Name |
| i O i O Littly that i so le lo k k s s le le |

If observation record e.g CONC has "NA" or "NS" then assign CONC cell as "."

If observation record e.g CONC has "NQ" or "BQL" then assign CONC cell as "." and MDV = 1 -this means value can be estimated by model

Missing covariate data should be imputed as "-99.

### 13.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

#### 13.9.1. Pharmacokinetic/Pharmacodynamic Methodology

PK-PD analysis of Nemiralisib will be guided by the results of the formal statistical analyses on the key clinical endpoints. The aims of the PK-PD analyses will contribute towards the dose selection in future studies using an integrated longitudinal analysis framework.

The objective is to explore an integrated modelling framework to characterise the longitudinal FEV1 response versus dose (average systemic exposure) during on- & off-treatment phases

$$FEV1_i(t_{ij}) = FEV1_{i,base} \cdot (1 + f(t_{ij}, dose_i, x_i) + \varepsilon_{ij} \text{ with } \varepsilon_{ij} \sim N(0, \sigma 2)$$

A longitudinal nonlinear mixed-effects model will be used to describe the FEV1 response over time measured for each patient (i) at each visit (tij) with  $\varepsilon$  denoting the normal distributed residual variability with mean 0 and variance  $\sigma$ 2. The function f() describes the relative change from observed FEV1 at baseline (FEV1, base) and any influence of patient characteristics on FEV1 response will be assessed.

Joint relationship between time to first exacerbation and FEV1 change as function of dose/exposure and patient covariates will be assessed.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

# 13.10. Appendix 10: Abbreviations & Trade Marks

# 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| APE | All Participants Enrolled |
| AUC | Area Under the Curve |
| BMI | Body Mass Index |
| CAT | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| COPD | Chronic Obstructive Pulmonary Disease |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CSV | Comma Separated Values |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| ERS | Evaluating Respiratory Symptoms |
| EXACT | Exacerbations of Chronic Pulmonary Disease Tool |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FEV1 | Forced Expiratory Volume in one second |
| FVC | Forced Vital Capacity |
| GSK | GlaxoSmithKline |
| HCRU | Health Care Resource Use |
| HPD | Highest Posterior Density |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| iSRC | Independent Safety Review Committee |
| KM | Kaplan-Meier |

| LLT | Lower Level Term |
|--------|----------------------------------------------------------|
| MCMC | Markov Chain Monte Carlo |
| MCSE | Monte Carlo Standard Errors |
| MDI | Metered Dose Inhaler |
| MITT | Modified Intent To Treat |
| OCS | Oral Corticosteroids |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| PRO | Patient Reported Outcomes |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SGRQ | St. George's Respiratory Questionnaire |
| SGRQ-C | St. George's Respiratory Questionnaire for COPD Patients |
| SoC | Standard of Care |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |

# 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| COPD Assessment Test (CAT) |
| ELLIPTA |
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| E-RS: COPD |
| EXACT-PRO |
| NONMEM |
| Propeller Sensor |
| SAS |
| SGRQ |

## 13.11. Appendix 11: List of Data Displays

## 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays for SAC:

| Section | Tables | Figures |
|------------------|--------------------------|----------------|
| Study Population | 1.1 to 1.31 | 1.3 |
| Efficacy | 2.1 to 2.107 2.1 to 2.20 | |
| Safety | 3.1 to 3.33 | 3.1 to 3.4 |
| Pharmacokinetic | 4.1 to 4.2 | Not applicable |
| Section | Listings | |
| ICH Listings | 1 to 27 | |
| Other Listings | 28 to 30 | |

## 13.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

#### 13.11.3. Deliverables

| Delivery | Description |
|---|---|
| IA | Interim Analysis (except the End of treatment Phase Interim Analysis) |
| EOT | End of Treatment Phase Interim Analysis |
| SAC Statistical Analysis Complete | |

# 13.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | MITT | ES8 | Summary of Subject Status and Reason for Study Withdrawal | | EOT, SAC |
| 1.2. | MITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | EOT, SAC |
| 1.3. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| 1.4. | APE | NS1 | Summary of Number of Participants by Country and Site ID | For EOT, use MITT population and summarise country only: Summary of Number of Participants by Country | EOT, SAC |
| Protoc | ol Deviation | | | | • |
| 1.5. | MITT | DV1 | Summary of Important Protocol Deviations | | SAC |
| 1.6. | MITT | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | ation Analysed | | | | |
| 1.7. | MITT | SP1 | Summary of Study Populations | | SAC |
| 1.8. | MITT | SP2 | Summary of Exclusions from the Per Protocol/Safety Population | | SAC |
| Demog | graphic and Bas | seline Characteris | tics | | 1 |
| 1.9. | MITT | DM1 | Summary of Demographic Characteristics | Use the following ranges for the Age<br>Group row: ≤64; 65-74; ≥75 | EOT, SAC |
| 1.10. | APE | DM11 | Summary of Age Ranges | | SAC |
| 1.11. | MITT | DM5 | Summary of Race and Racial Combinations | | SAC |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.12. | MITT | MH4 | Summary of Past Medical Conditions | | SAC |
| 1.13. | MITT | MH4 | Summary of Current Medical Conditions | | SAC |
| 1.14. | MITT | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 1.15. | MITT | SU1 | Summary of Smoking History at Screening | | EOT, SAC |
| 1.16. | MITT | SU1 | Summary of Smoking Status Over the 12-Week Treatment Period | | SAC |
| 1.17. | MITT | SU1 | Summary of Smoking Status Over the 12-Week Follow-Up Period | | SAC |
| 1.18. | MITT | Example 7 | Summary of COPD Duration at Screening | | SAC |
| 1.19. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening | Use categories 0;1;2;3;≥3. Summarise moderate/severe, moderate; severe Include 7-Day History of COPD Exacerbations | EOT, SAC |
| 1.20. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening by Country | | SAC |
| Conco | mitant Medicati | ons | | · | |
| 1.21. | MITT | Example 14 | Summary of Baseline COPD Maintenance Therapy | For EOT use categories: Triple,<br>Non-triple | EOT, SAC |
| 1.22. | MITT | Example 14 | Summary of Baseline ICS Therapy | For EOT use categories: Yes, No | EOT, SAC |
| 1.23. | MITT | Example 15 | Summary of On-Treatment COPD Maintenance (Step-up) Therapy | | SAC |
| 1.24. | MITT | CM1 | Summary of Concomitant Medications During 12-Week<br>Treatment Period | | SAC |
| 1.25. | MITT | Example 16 | Summary of Duration of On-Treatment OCS | | EOT, SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.26. | MITT | Example 16 | Summary of Duration of On-Treatment OCS Excluding Non-COPD medications | | EOT, SAC |
| 1.27. | MITT | CM1 | Summary of Concomitant Medications During 12-Week Follow-<br>Up Period | | SAC |
| Exposu | re and Treatmen | t Compliance | | | |
| 1.28. | MITT | Example 36 | Summary of Exposure to Study Treatment | | EOT, SAC |
| 1.29. | MITT | Example 2 | Summary of Overall Treatment Compliance Measured by the Dose Counter on the ELLIPTA | | EOT, SAC |
| 1.30. | MITT | Example 2 | Summary of Reported Treatment Compliance from the Daily eDiary | | SAC |
| 1.31. | MITT | Example 2 | Summary of Overall Treatment Compliance Measured by the Clip-on Propeller Sensor for ELLIPTA | | SAC |

# 13.11.5. Study Population Figures

| Study F | Study Population Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | MITT | Example 4 | Plot of COPD Exacerbation History at Screening (Moderate) | | EOT |
| 1.2. | MITT | Example 4 | Plot of COPD Exacerbation History at Screening (Severe) | | EOT |
| 1.3. | MITT | Example 4 | Plot of COPD Exacerbation History at Screening (Moderate/Severe) | | EOT |

# 13.11.6. Efficacy Tables

## 13.11.6.1. Efficacy tables for Interim Analysis 1

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | IA1 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | IA1 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator (Dose Response Model) | | IA1 |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator (Dose Response Model) | | IA1 |
| 2.7. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.8. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.9. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | IA1 |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Pre-bronchodilator (Repeated Measures Model) | | IA1 |
| 2.11. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| 2.12. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| Rate of | Exacerbations | | | | |
| 2.13. | MITT | Example 5 | Summary of On-treatment Exacerbations | | IA1 |
| 2.14. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Severity | | IA1 |
| EXAce | rbations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.15. | MITT | Example 9 | Summary of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | Exclude statistical analysis information (summary only) | IA1 |
| 2.16. | MITT | Example 9 | Summary of Proportion of Participants Achieving the EXACT-<br>definition of Recovery by Index Exacerbation Severity | Exclude statistical analysis information (summary only) | IA1 |
| Other S | Spirometry Mea | sures | | | |
| 2.17. | MITT | Example 3 | Summary of Spirometry Measurements | | IA1 |
| 2.18. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA1 |

# 13.11.6.2. Efficacy tables for Interim Analysis 2

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | e from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator Include additional row for hospital discharge visit for Severe group | IA2 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | IA2 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.9. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.10. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.12. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.13. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.14. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.15. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.16. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.17. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.18. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Pre-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.19. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.20. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| 2.21. | MITT | Example 32 | Summary of Efficiency Ratio for Possible Adaptions to Randomization Ratio | | IA2 |
| Rate of | Exacerbations | 1 | | | |
| 2.22. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations | | IA2 |
| 2.23. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | IA2 |
| 2.24. | MITT | Example 6 | Statistical Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations | | IA2 |
| 2.25. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | IA2 |
| EXAce | rbations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | , | |
| 2.26. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | IA2 |
| 2.27. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | IA2 |
| COPD | Assessment Te | st (CAT) | | · | |
| 2.28. ) | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score | | IA2 |
| 2.29. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the CAT Total Score by Visit | | IA2 |
| 2.30. | MITT | Example 11 | Statistical Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) | | IA2 |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) | | |
| 2.31. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score | | IA2 |
| 2.32. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the SGRQ Total Score by Visit | | IA2 |
| 2.33. | MITT | Example 11 | Statistical Analysis of Change from Baseline in SGRQ Total Score (Repeated Measures Model) | | IA2 |
| Rescue | Medication Us | se | | | |
| 2.34. | MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | IA2 |
| 2.35. | MITT | RM1 | Summary of Percentage of Rescue-Free Days | | IA2 |
| Other S | Spirometry Mea | sures | | · | |
| 2.36. | MITT | Example 3 | Summary of Spirometry Measurements | | IA2 |
| 2.37. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA2 |

## 13.11.6.3. Efficacy tables for End of Treatment Interim Analysis and SAC

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | EOT, SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | EOT, SAC |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator (Dose Response Model) | | SAC |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator (Dose Response Model) | | SAC |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator (Dose Response Model) | | SAC |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator (Dose Response Model) | | SAC |
| 2.9. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | SAC |
| 2.10. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | SAC |
| 2.11. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | SAC |
| 2.12. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | SAC |
| 2.14. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | SAC |
| 2.15. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | SAC |
| 2.16. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | SAC |
| 2.17. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.18. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV₁ | | |
| 2.19. | MITT | Example 3 | Summary of Change from Hospital Discharge in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | SAC |
| 2.20. | MITT | Example 11 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | SAC |
| 2.21. | MITT | Example 11 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) Measured Pre-bronchodilator (Repeated Measures Model) | | SAC |
| Change | from Day 84 in | n Clinic Visit trouç | gh FEV <sub>1</sub> | | |
| 2.22. | MITT | Example 3 | Summary of Change from Day 84 in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | SAC |
| 2.24. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Pre-bronchodilator (Repeated Measures Model) | | SAC |
| 2.25. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | SAC |
| 2.26. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | SAC |
| Rate of | f Exacerbations | ; | | • | |
| 2.27. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.28. | MITT | Example 5 | Summary of On-treatment (Mild/Moderate/Severe) Subsequent Exacerbations | | SAC |
| 2.29. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent<br>Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.30. | MITT | Example 6 | Statistical Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.31. | MITT | Example 6 | Statistical Analysis of On-treatment (Mild/Moderate/Severe) Subsequent Exacerbations | | SAC |
| 2.32. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.33. | MITT | Example 5 | Summary of On-treatment Subsequent Exacerbations by Index Exacerbation Type | | SAC |
| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | MITT | Example 5 | Summary of On-treatment Subsequent Exacerbations by Number of Exacerbations in Previous 12 Months | | SAC |
| 2.35. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent<br>Exacerbations by Baseline Maintenance Therapy | | EOT, SAC |
| 2.36. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Baseline Maintenance Therapy | | EOT, SAC |
| 2.37. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations by Baseline ICS Therapy | | EOT, SAC |
| 2.38. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Baseline ICS Therapy | | EOT, SAC |
| 2.39. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by EXACT Recovery Status at Day 14 | | EOT, SAC |
| 2.40. | MITT | Example 12 | Summary of Number of On-treatment Subsequent (Moderate/Severe) Exacerbations Treated with Steroids/Antibiotics | | EOT, SAC |
| 2.41. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Baseline Blood Biomarker Status | | EOT, SAC |
| 2.42. | MITT | Example 5 | Summary of On-or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | SAC |
| 2.43. | MITT | Example 5 | Summary of On-or Off-treatment (Mild/Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | SAC |
| 2.44. | MITT | Example 5 | Summary of On-or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period by Index Exacerbation Severity | | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.45. | MITT | Example 6 | Statistical Analysis of On- or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | EOT, SAC |
| 2.46. | MITT | Example 6 | Statistical Analysis of On- or Off-treatment (Mild/Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | SAC |
| 2.47. | MITT | Example 6 | Subgroup Analysis of On- or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period by Index Exacerbation Severity | | SAC |
| 2.48. | MITT | Example 5 | Summary of Off-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.49. | MITT | Example 5 | Summary of Off-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | SAC |
| 2.50. | MITT | Example 6 | Statistical Analysis of Off-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.51. | MITT | Example 6 | Subgroup Analysis of Off-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | SAC |
| 2.52. | MITT | Example 5 | Summary of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period | | SAC |
| 2.53. | MITT | Example 5 | Summary of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period by Index Exacerbation Severity | | SAC |
| 2.54. | MITT | Example 6 | Statistical Analysis of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period | | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.55. | MITT | Example 6 | Subgroup Analysis of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period by Index Exacerbation Severity | | SAC |
| Time to | Next Exacerba | ation | | | |
| 2.56. | MITT | Example 8 | Statistical Analysis of Time to next On-treatment Exacerbation | | EOT, SAC |
| 2.57. | MITT | Example 8 | Subgroup Analysis of Time to next On-treatment Exacerbation by Index Exacerbation Severity | | EOT, SAC |
| 2.58. | MITT | Example 8 | Statistical Analysis of Time to next On- or Off-treatment Exacerbation During the 12-Week Treatment Period | | SAC |
| 2.59. | MITT | Example 8 | Statistical Analysis of Time to next On- or Off-treatment Exacerbation During the 12-Week Treatment Period by Index Exacerbation Severity | | SAC |
| 2.60. | MITT | Example 8 | Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment | | SAC |
| 2.61. | MITT | Example 8 | Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment by Index Exacerbation Severity | | SAC |
| EXAce | rbations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.62. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | EOT, SAC |
| 2.63. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | EOT, SAC |
| 2.64. | MITT | Example 8 | Summary and Statistical Analysis of Time to EXACT-defined Recovery | | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.65. | MITT | Example 10 | Summary of Severity of Subsequent HCRU-defined<br>Exacerbation During 12-Week Treatment Period | Also split by moderate and severe | SAC |
| 2.66. | MITT | Example 10 | Summary of Severity of Subsequent HCRU-Defined Exacerbation During 12-Week Follow-up Period | Also split by moderate and severe | SAC |
| 2.67. | MITT | Example 35 | Summary of Missing On-treatment EXACT-PRO data | | EOT, SAC |
| 2.68. | MITT | Example 35 | Summary of Missing Off-treatment EXACT-PRO data | | SAC |
| COPD | Assessment Te | est (CAT) | | | |
| 2.69. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score | | EOT, SAC |
| 2.70. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score by Index Exacerbation Severity | | SAC |
| 2.71. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the CAT Total Score by Visit | | EOT, SAC |
| 2.72. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders Using the CAT Total Score by Visit by Index Exacerbation Severity | | SAC |
| 2.73. | MITT | Example 11 | Statistical Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.74. | MITT | Example 11 | Subgroup Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | SAC |
| 2.75. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score | | SAC |
| 2.76. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score by Index Exacerbation Severity | | SAC |
| 2.77. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) | | SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.78. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | SAC |
| St. Geo | rge's Respirat | ory Questionnaire | (SGRQ) | | |
| 2.79. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score | | EOT, SAC |
| 2.80. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score by Index Exacerbation Severity | | SAC |
| 2.81. | MITT | Example 9 | Statistical Analysis of Proportion of Responders on the SGRQ<br>Total Score by Visit | | EOT, SAC |
| 2.82. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders on the SGRQ<br>Total Score by Index Exacerbation Severity | | SAC |
| 2.83. | MITT | Example 11 | Statistical Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.84. | MITT | Example 11 | Subgroup Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) by Index Exacerbation Severity | | SAC |
| 2.85. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score | | SAC |
| 2.86. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score by Index Exacerbation Severity | | SAC |
| 2.87. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in SGRQ Total Score (Repeated Measures Model) | | SAC |
| 2.88. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in SGRQ<br>Total Score (Repeated Measures Model) by Index Exacerbation<br>Severity | | SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| E-RS: ( | COPD | 1 | | | |
| 2.89. | MITT | Example 3 | Summary of Change from Baseline in E-RS: COPD and Subscales | | SAC |
| Rescue | Medication Us | se | | | |
| 2.90. | MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | EOT, SAC |
| 2.91. | MITT | RM1 | Summary of Percentage of Rescue-Free Days | | EOT, SAC |
| 2.92. | MITT | RM1 | Summary of Mean Number of Actuations of Rescue Medication Use Per Day Via the Clip-on Propeller Sensor for MDI | | SAC |
| 2.93. | MITT | RM1 | Summary of Percentage of Rescue-Free Days Via the Clip-on Propeller Sensor for MDI | | SAC |
| Health | care Resource | Utilisation | | | |
| 2.94. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilisation | | SAC |
| 2.95. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilization by Index Exacerbation Severity | | SAC |
| 2.96. | MITT | Example 21 | Summary of Exacerbation Related Hospitalizations | | SAC |
| 2.97. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation | | SAC |
| 2.98. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | SAC |
| 2.99. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation | | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.100. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | SAC |
| 2.101. | MITT | Example 22 | Summary of Re-hospitalization Within 30 days of Index Exacerbation | | SAC |
| 2.102. | MITT | Example 24 | Summary of Time from Resolution of Index Exacerbation to Next Exacerbation | | SAC |
| 2.103. | MITT | Example 23 | Summary of Subsequent Exacerbation Treatment | | SAC |
| Other S | pirometry Mea | sures | | | |
| 2.104. | MITT | Example 3 | Summary of Spirometry Measurements | | EOT, SAC |
| 2.105. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | EOT, SAC |
| Inflamn | natory/infective | Markers in Blood | d and Sputum | | |
| 2.106. | MITT | Example 3 | Summary of Inflammatory Markers in Blood | For EOT only include Screening timepoint | EOT, SAC |
| 2.107. | MITT | Example 3 | Summary of Inflammatory Markers in Sputum | | SAC |

# 13.11.7. Efficacy Figures

## 13.11.7.1. Efficacy Figures for Interim Analysis 1

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | e from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | IA1 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | IA1 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 measured post-bronchodilator | | IA1 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |

## 13.11.7.2. Efficacy Figures for Interim Analysis 2

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | IA2 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | IA2 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator | | IA2 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator | | IA2 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.13. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator | | IA2 |
| 2.14. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.15. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| Time to | Next Exacerba | ation | | | |
| 2.16. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Moderate/Severe) Exacerbation | | IA2 |
| 2.17. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Mild/Moderate/Severe) Exacerbation | | IA2 |

## 13.11.7.3. Efficacy Figures for End of Treatment Interim Analysis and SAC

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | SAC |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | SAC |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator | | SAC |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator | | SAC |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | SAC |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | SAC |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | SAC |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | SAC |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | SAC |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | SAC |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | SAC |
| 2.13. | MITT | Example 31 | Plot of Adjusted Posterior Medians (95% HPD Crl) of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator | | EOT, SAC |
| 2.14. | MITT | Example 31 | Plot of Adjusted Posterior Medians (95% HPD Crl) of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC |
| 2.15. | MITT | Example 31 | Plot of Adjusted Posterior Medians (95% HPD Crl) of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC |
| Time to | Next Exacerba | ation | | | |
| 2.16. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Moderate/Severe) Exacerbation | | EOT, SAC |
| 2.17. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Mild/Moderate/Severe) Exacerbation | | SAC |
| 2.18. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-or Off-treatment (Moderate/Severe) Exacerbation During the 12-Week Treatment Period | | SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-or Off-treatment (Mild/Moderate/Severe) Exacerbation During the 12-Week Treatment Period | | SAC |
| 2.20. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next (Moderate/Severe) Exacerbation Following Cessation of Study Treatment | | SAC |

# 13.11.8. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | | EOT, SAC |
| 3.2. | Safety | AE1 | Summary of Post-Treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Treatment Emergent Adverse Events by Overall Frequency | | EOT, SAC |
| 3.4. | Safety | AE1 | Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term | | EOT, SAC |
| 3.5. | Safety | AE15 | Summary of Common (>=5%) Non-serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | | SAC |
| 3.6. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.7. | Safety | AE1 | Summary of Treatment Emergent Adverse Events for<br>Participants with Absolute Neutrophil Count Below Lower Value of PCI | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | , | |
| 3.8. | Safety | AE16 | Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | | EOT, SAC |
| 3.9. | Safety | AE16 | Summary of Fatal Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | Only with subcategory: Number of Fatal SAEs | EOT, SAC |
| 3.10. | Safety | AE1 | Summary of Serious Treatment Emergent Drug-related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.11. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | EOT, SAC |
| 3.12. | Safety | AE1 | Summary of Post-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.13. | Safety | AE1 | Summary of Treatment Emergent Adverse Events of Special Interest by Lower Level Term | | EOT, SAC |
| 3.14. | Safety | AE1 | Summary of Treatment Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term | | EOT, SAC |
| 3.15. | Safety | Example 17 | Summary of Post-Inhalation Cough by Visit | | EOT, SAC |
| 3.16. | Safety | Example 28 | Summary of Post-Inhalation Cough by Visit and Cough Type | | EOT, SAC |
| 3.17. | Safety | Example 33 | Summary of Post-Inhalation (PI) Cough at Any Visit | | EOT, SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Chemistry | / | | | |
| 3.18. | Safety | LB1 | Summary of Chemistry Data | For EOT summarise Alkaline<br>Phosphates at Screening only | EOT, SAC |
| 3.19. | Safety | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.20. | Safety | LB1 | Summary of Hematology Data | For EOT summarise Eosinophils,<br>Monocytes, Lymphocytes at Screening<br>only | EOT, SAC |
| 3.21. | Safety | LB1 | Summary of Change from Baseline in Hematology | Only for WBC, lymphocytes, neutrophils | SAC |
| 3.22. | Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.23. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC |
| 3.24. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC |
| ECG | | | | | |
| 3.25. | Safety | EG1 | Summary of ECG Findings | Include Worst Case<br>Post-Baseline row | EOT, SAC |
| 3.26. | Safety | EG2 | Summary of ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | EOT, SAC |
| 3.27. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | SAC |
| 3.28. | Safety | Example 27 | Summary of QTcF Categories | | SAC |
| 3.29. | Safety | Example 27 | Summary of QTcB Categories | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.30. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.31. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.32. | Safety | Example 25 | Summary of ECG Abnormalities for Participants with Any Abnormal ECG Interpretation | | EOT, SAC |
| Vital Si | gns | | | | |
| 3.33. | Safety | VS1 | Summary of Vital Signs | | SAC |
| 3.34. | Safety | VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |

# 13.11.9. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | Laboratory | | | | |
| 3.1. | Safety | LB7 | LFT Shift from Baseline to Maximum | | EOT, SAC |
| 3.2. | Safety | Example 34 | Plot of Laboratory Data at Screening | | EOT, SAC |
| 3.3. | Safety | Example 13 | Median (range) Absolute Neutrophil Count by Time and Treatment | | SAC |
| ECG | | | | | |
| 3.4. | Safety | EG8 | Distribution of QTcF Change by Time and Treatment | | SAC |

### 13.11.10. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | Pharmacokinetic Concentration-Time Data | | | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK2269557 Pharmacokinetic Concentration-Time Data | | SAC |
| 4.2. | PK | PK05 | Summary of Log-Transformed Plasma GSK2269557 Pharmacokinetic Concentration-Time Data | | SAC |

# 13.11.11. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | MITT | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | MITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 4. | MITT | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | | SAC |
| 5. | MITT | TA1 | Listing of Planned and Actual Treatments | | SAC |
| Protoc | ol Deviations | | | | |
| 6. | MITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 7. | MITT | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | , | |
| 8. | MITT | SP3 | Listing of Participants Excluded from Per Protocol Population | For participants excluded from MITT population (i.e. participants in the MITT but not in PP) | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | MITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 10. | MITT | DM9 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | MITT | CP_CM3 | Listing of Concomitant Medications | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | re and Treatmo | ent Compliance | | | |
| 12. | Safety | EX3 | Listing of Exposure Data | | SAC |
| Advers | e Events | | | | |
| 13. | Safety | AE8 | Listing of All Adverse Events | | SAC |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Seriou | s and Other Sig | nificant Adverse | -<br>Events | | |
| 16. | Safety | AE8 | Listing of Fatal Serious Adverse Events | | SAC |
| 17. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 18. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | | SAC |
| All Lab | oratory | | | | |
| 22. | Safety | LB5 | Listing of All Chemistry Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 23. | Safety | LB14 | Listing of Chemistry Data with Character Results | | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Safety | LB5 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 25. | Safety | LB14 | Listing of all Hematology Data with Character Results | | SAC |
| ECG | | | | | |
| 26. | Safety | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | | SAC |
| 27. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal Finding | | SAC |

## 13.11.12. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 28. | MITT | Example 29 | Listing of Subjects who Received Incorrect Medication | | SAC |
| 29. | PK | PK07 | Listing of Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 30. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC |

## 13.12. Appendix 12: Example Mock Shells for Data Displays

### 13.12.1. Example shell 1

Example Shell X

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Exacerbation History at Screening

| | Treatment A (N=100) | Treatment B (N=100) | Total<br>(N=200) |
|---|---|---|---|
| Moderate COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Severe COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Total number of moderate/severe COPD exacerbations | | | |
| n | 911 | 899 | 1810 |
| 0 | 313 (34%) | 317 (35%) | 630 (35%) |
| 1 | 252 (28%) | 253 (28%) | 505 (28%) |
| >=2 | 346 (38%) | 329 (37%) | 675 (37%) |

Note: Number of COPD exacerbations reported in the 12 months prior to the Screening Visit.

xx (x%)

xx (x%)


## **13.12.2. Example Shell 2**

100% - < 120%

>=120%

Protocol: XYZ100001 

| | Treatm<br>(N=100 | | | tal<br>200) |
|------------------------|------------------|-------|--------|-------------|
| Overall compliance (%) | | | | |
| n | XX | XX | XX | |
| Mean | XX | XX | XX | |
| SD | XX | XX | XX | |
| Median | XX | XX | XX | |
| Min. | XX | XX | XX | |
| Max. | xx | XX | XX | |
| Compliance interval | | | | |
| < 80% | xx (x | %) xx | (x%) x | x (x%) |
| 80% - < 100% | xx (x | %) xx | (x%) x | x (x%) |

xx (x%)

xx (x%)

xx (x%)

xx (x%)


## 13.12.3. Example shell 3

Example Shell X
Protocol: ABC123456

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Change from Baseline in FEV1 (L)  $\qquad \qquad \text{Measured post-bronchodilator}$ 

| Visit | | N | Treatment 2 | Arm | | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Day 1 | 200 | <br>P | lacebo | | 200 | 0 | .111 0.1 | 111 0. | .100 -0. | 11 1.1 | <br>.1 |
| - | | 200 | GSK2269557 | 12.5 | mcg | 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | | 200 | GSK2269557 | 50 | mcg | 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | | 200 | GSK2269557 | 100 | mcg | 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | | 200 | GSK2269557 | 250 | mcg | 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | | 200 | GSK2269557 | 500 | mcg | 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | | 200 | GSK2269557 | 750 | mcg | 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| Day 14 | 200 | Р | lacebo | | 200 | 0 | .111 0.1 | .111 0. | .100 -0. | 11 1.1 | 11 |
| | | 200 | GSK2269557 | 12.5 | mcg | 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | | 200 | GSK2269557 | 50 | mcg | 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | | 200 | GSK2269557 | 250 | mcg | 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | | 200 | GSK2269557 | 500 | mcg | 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | | 200 | GSK2269557 | 750 | mcq | 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |


## 13.12.4. Example Shell 4

Protocol: ABC123456

Population: Intent-to-Treat/Safety/Other study specific

Figure X

Plot of Number of Exacerbations in Previous 12 Months (Moderate/Severe)



Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Statistical Analysis of Change from Baseline in FEV1 (ml)
Measured post-bronchodilator

| Visit | Treatment Comparison | Adjusted<br>Median<br>Difference | Std Dev | 95% Credible<br>Interval | Prob Treat. Diff >0 (%) |
|---|---|---|---|---|---|
| Day 14 | GSK2269557 12.5 mg vs<br>Placebo | x.xx | х.хх | (x.xx, x.xx) | X.XX |
| | GSK2269557 50 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 100 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 250 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | X.XX |
| | GSK2269557 500 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 750 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| Day 28 | GSK2269557 12.5 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 50 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | X.XX |
| | GSK2269557 100 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |

## **13.12.5. Example Shell 5**

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific
Table X
Summary of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Number of moderate/severe exacerbations per subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |
| 4 | 0 | 2 (2%) |
| 5 | 0 | 1 (1%) |
| >5 | 0 | 1 (1%) |
| Subjects with >=1 moderate/severe exacerbation | 13 (13%) | 28 (28%) |
| Total Number of moderate/severe exacerbations | 21 | 49 |
| Number of moderate exacerbations per Subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |

## **13.12.6. Example Shell 6**

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific
Table X
Statistical Analysis of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Moderate/severe exacerbations Annual exacerbation rate (95% CrI) Active vs. Placebo | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx) |
| Ratio Pr Diff <1 Percent reduction in rate (95% CrI) | | 0.85 (x.xx, x.xx)<br>x.xx<br>15% (x.xx, x.xx) |
| Predictive probability (%) [1] [only when required] | xx% | , , , , , , , |
| Moderate exacerbations Annual exacerbation rate (95% CrI) Active vs. Placebo | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx) |
| Ratio Pr Diff <1 Percent reduction in rate (95% CrI) | | 0.85 (x.xx, x.xx)<br>x.xx<br>15% (x.xx, x.xx) |

<sup>[1]</sup> Predictive posterior probability of success at end of study, where success is Pr(Reduction>0%)>80% PPD

## 13.12.7. **Example Shell 7**

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific
Table X

Summary of COPD Duration at Screening

| | Treatme (N=100) | | Treatme (N=100) | | Total<br>(N=200) | |
|---|---|---|---|---|---|---|
| Duration of COPD: | | | | | | |
| n | 100 | | 99 | | 199 | |
| <1 year | XX | (x%) | XX | (x%) | XX | (x%) |
| >=1 to <5 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=5 to <10 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=10 to <15 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=15 to <20 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=20 to <25 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=25 years | XX | (x%) | XX | (x%) | XX | (x%) |

### 13.12.8. **Example Shell 8**

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary and Analysis of Time to Next On-treatment Moderate/Severe Exacerbation (days) up to Day 84

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Number of Subjects with Event Number of Subjects Censored | 10 (10%)<br>90 (90%) | 14 (14%)<br>86 (86%) |

Treatment A vs. Placebo
Hazard Ratio
95% Credible Interval

X.XX
(x.xx, x.xx)

Note: Hazard ratio and 95% Credible Interval are from a Bayesian Cox proportional hazards model

## 13.12.9. **Example Shell 9**

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Statistical Analysis of Proportion of Participants Achieving EXACT-definition of Response

| | Treatment A $(N=100)$ | Treatment B $(N=100)$ |
|---|---|---|
| Day 14 | | |
| n | X.XX | X.XX |
| Responder | | x.xx (x%) |
| Non-responder | x.xx (x%) | |
| Active vs. Placebo | , , | , |
| Odds Ratio (OR) (95% CrI) | x.xx (x.xx | x, x.xx) x.xx (x.xx, x.xx |
| Pr OR >1 | x.xx x.x | xx |
| Day 28 | | |
| n | X.XX | x.xx |
| Responder | x.xx (x%) | x.xx (x%) |
| Non-responder | x.xx (x%) | x.xx (x%) |
| Active vs. Placebo | | |
| Odds Ratio (95% CrI) | x.xx (x.xx, x | x.xx) x.xx (x.xx, x.xx) |
| Pr Diff >1 | X . XX | X . XX |

## 13.12.10. Example Shell 10


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of severity of subsequent HCRU-defined exacerbation during 12-Week Treatment Period

| Treatment | N | n | Mean | SD | Median | Min. | Max. |
|-----------|----|----|-------|-------|--------|-------|-------|
| Placebo | 30 | 30 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Trt A | 30 | 30 | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx |
| Trt B | 30 | 30 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

## 13.12.11. Example Shell 11

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Mixed Model Repeated Measures Analysis of CAT Total Score

| | | atment A Trea (N=100) (N= | tment B<br>100) |
|---|---|---|---|
| Day 28 | | | |
| n | X.XX | x.xx | |
| Adjusted mean score change (SE)<br>Active - Placebo | ) x.xx | (x) x.xx | (x) |
| Difference (SE) | X.XX | (x.xx) $x.xx$ | (x.xx) |
| 95% (CrI) | X.XX | X.XX | |
| Pr Diff >0 | x.xx | X.XX | |
| Day 56 | | | |
| n | X.XX | x.x | X |
| Adjusted mean score change (SE)<br>Active - Placebo | ) x.xx | (x) x.xx | (x) |
| Difference (SE) | X.XX | (x.xx) $x.xx$ | (x.xx) |
| 95% (CrI) | X.XX | X.XX | |
| Pr Diff >0 | X.XX | X.XX | |

## 13.12.12. Example Shell 12

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of the Number of Subsequent (On-treatment) Exacerbations Treated with Steroids/Antibiotics

| | Treatment A (N=100) | Treatment B (N=100) |
|---------------------|---------------------|---------------------|
| Total exacerbations | 50 | 51 |
| Treatment | | |
| Antibiotics | 30 | 40 |
| Steroids | 50 | 40 |
| Both | 30 | 30 |

## 13.12.13. Example shell 13

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific

Figure X Median (range) Absolute Neutrophil Count by Time and Treatment



## 13.12.14. Example Shell 14


Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of Baseline COPD Maintenance Therapy

| Therapy category | Treatm<br>(N=8 | | Treatment B (N=79) | |
|---|---|---|---|---|
| Any medication at baseline | 70 (8 | 36%) | 50 | (63%) |
| Monotherapy<br>LAMA only | X (2 | , | | (x%)<br>(x%) |
| Dual therapy<br>ICS/LABA<br>Dual bronchodilator | x (2<br>x | (x%) | Х | (x%)<br>(x%)<br>(xx%) |
| Triple therapy LAMA/ICS/LABA | • | <%)<br>(x%) | X<br>0 | (x%) |

## 13.12.15. Example Shell 15


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of On-Treatment COPD Maintenance (Step-up) Therapy

| | Treatment A | Treatment B |
|---------------------|-------------|-------------|
| Therapy category | (N=81) | (N=79) |
| Any Step-up Therapy | 70 (86%) | 50 (63%) |
# 13.12.16. Example shell 16


Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of OCS use

| | Treatment A (N=81) | Treatment B (N=79) |
|---|---|---|
| OCS use for index exacerbation Total number of Days of OCS use | 81 (100%) | 79 (100%) |
| Mean | Xx | XX |
| SD | Xx | XX |
| Median | Xx | XX |
| Min. | Xx | XX |
| Max. | Xx | XX |
| On-treatment OCS use | xx (xx%) | xx (xx%) |
| Total number of Days of OCS use | | |
| Mean | Xx | XX |
| SD | Xx | XX |
| Median | Xx | XX |
| Min. | Xx | XX |
| Max. | Xx | XX |

# 13.12.17. Example Shell 17


Population: Safety

Visit: VISIT 2 (RANDOMISATION)

| | | acebo<br>=43) | 50 | K2269557<br>mcg<br>=14) | 100 | X2269557<br>D mcg<br>=15) | 25 | K2269557<br>0 mcg<br>=16) | 50 | SK2269557<br>)0 mcg<br>J=14) | 750 | (2269557<br>mcg<br>(42) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Did subject experience PI cough? [1] | | | | | | | | | | | | |
| n | 20 | | 10 | | 12 | | 15 | | 1 | _2 | 35 | |
| Yes | 7 | (35%) | 4 | (40%) | 6 | (50%) | 3 | (20%) | | 6 (50%) | 12 | (34%) |
| No | 13 | (65%) | 6 | (60%) | 6 | (50%) | 12 | (80%) | | 6 (50%) | 23 | (66%) |
| Type of cough | | | | | | | | | | | | |
| Single cough | 4 | (57%) | 2 | (50%) | 1 | (17%) | 1 | (33%) | 1 | (17%) | 2 | (17%) |
| Intermittent cough | 2 | (29%) | 2 | (50%) | 5 | (83%) | 1 | (33%) | 4 | (67%) | 5 | (42%) |
| Continuous cough | 1 | (14%) | 0 | | 0 | | 1 | (33%) | 1 | (17%) | 5 | (42%) |
| Severity of cough | | | | | | | | | | | | |
| Mild | 5 | (71%) | 3 | (75%) | 3 | (50%) | 2 | (67%) | 1 | (17%) | 6 | (50%) |
| Moderate | 2 | (29%) | 1 | (25%) | 2 | (33%) | 1 | (33%) | 5 | (83%) | 4 | (33%) |
| Severe | 0 | | 0 | | 1 | (17%) | 0 | | 0 | | 2 | (17%) |
| Time to onset of PI cough (minutes) | | | | | | | | | | | | |
| 0-1 | 6 | (86%) | 3 | (75%) | 6 | (100%) | 3 | (100%) | 6 | (100%) | 12 | (100응) |
| >1-2 | 1 | (14%) | 1 | (25%) | 0 | | 0 | | 0 | | 0 | |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| Duration of PI cough (minutes) | | | | | | | | | | | | |
| <=1 | 6 | (86%) | 3 | (75%) | 5 | (83%) | 3 | (100%) | 5 | (83%) | 11 | (92%) |
| >1-2 | 1 | (14%) | 1 | (25%) | 1 | (17%) | 0 | | 1 | (17%) | 1 | (8%) |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |

| | | CC | ONFII | DENTIAL | | | | | 201 | 9N39 | 98117_00<br>200 | )<br>1879 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| >5-10<br>>10-30<br>>30 | X<br>X<br>X | | X<br>X<br>X | | | | | | | | | |
| Number of subjects reporting cough as AE/SAE Mild Moderate Severe | 2<br>x<br>x<br>x | (29%)<br>(x%)<br>(x%)<br>(x%) | 1<br>x<br>x<br>x | (25%) | 4 | (67%) | 0 | 2 | (33%) | 3 | (25%) | |

<sup>[1]</sup> Percentages are calculated using the number of subjects evaluated at visit as the denominator.

All other percentages are calculated using the number of subjects with a PI cough at visit as the denominator.

### 13.12.18. Example shell 18


Population: Intent-to-Treat/Safety/Other study specific Figure X

Plot of Dose Response Model of Change from Baseline in FEV1



[Footnote to describe the fitted model]

### 13.12.19. Example Shell 19

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | | Treatment (N=100) | |
|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | 97<br>3 | (97%)<br>( 3%) | 19<br>81 | (19%)<br>(81%) |
| Number of Home Visits (day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>90<br>4<br>0<br>0<br>0 | (90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2<br>4 | (92%)<br>(4%)<br>(<1%) |
| Number of Home Visits (night) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>100 (<br>0<br>0<br>0<br>0 | (100%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | | atment A<br>LOO) | Trea<br>(N=1 | atment B<br>LOO) |
|---|---|---|---|---|---|
| Number of Office/Practice Visits | n | 911 | | 899 | |
| | 0 | 846 | (93%) | 808 | (90%) |
| | 1 | | (5%) | | |
| | 2 | | (1%) | | |
| | 3 | | (<1%) | | |
| | >3 | 3 | (<1%) | 2 | (<1%) |
| | Total [1] | 103 | | 140 | |
| Number of Urgent Care/Outpatient Visits | n | 911 | | 899 | |
| . J | 0 | | (97%) | | (98%) |
| | 1 | | (2%) | | (1%) |
| | 2 | | (<1%) | | |
| | 2<br>3 | | (<1%) | | (<1%) |
| | >3 | 4 | (<1%) | 2 | (<1%) |
| | Total [1] | 54 | | 37 | |
| Number of Emergency Room Visits | n | 911 | | 899 | |
| | 0 | 906 | (>99%) | | (>99%) |
| | 1 | 5 | (<1%) | | (<1%) |
| | 2 | 0 | | | (<1%) |
| | 2<br>3 | 0 | | 0 | |
| | >3 | 0 | | 0 | |
| | Total [1] | 5 | | 7 | |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Days in Intensive Care | n | 911 | 899 |
| - | 0 | 910 (>99%) | 894 (>99%) |
| | 1 | 0 | 0 |
| | 2 | 0 | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 1 (<1%) | 4 (<1%) |
| | Total [2] | 12 | 40 |
| Number of Days in General Ward | n | 911 | 899 |
| | 0 | 896 (98%) | 878 (98%) |
| | 1 | 0 | 2 (<1%) |
| | 2 | 1 (<1%) | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 14 (2%) | 18 (2%) |
| | Total [2] | 119 | 258 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

### 13.12.20. Example Shell 20


Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of Non-COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | | Treatment (N=100) | |
|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | 97<br>3 | (97%)<br>( 3%) | 19<br>81 | (19%)<br>(81%) |
| Number of Days in Accident and emergency | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>90<br>4<br>0<br>0<br>0 | (90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2<br>4 | (92%)<br>(4%)<br>(<1%) |
| Number of Days in General Ward | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>100 (<br>0<br>0<br>0<br>0 | (100%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) |

# 13.12.21. Example Shell 21

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of Exacerbation Related Hospitalizations

| | | Treatment B (N=100) |
|-----------------------------------|------|---------------------|
| Index exacerbation | | |
| Participants with hospitalization | x.xx | x.xx |
| Number of hospitalizations | X.XX | x.xx |
| Mean duration (days) | X.XX | X.XX |
| SD | X.XX | X.XX |
| Median duration (days) | x.xx | x.xx |
| Minimum duration (days) | X.XX | X.XX |
| Maximum duration (days) | X.XX | x.xx |
| Subsequent exacerbations | | |
| Participants with hospitalization | x.xx | x.xx |
| Number of hospitalizations | X.XX | X.XX |
| Mean duration (days) | X.XX | X.XX |
| SD | x.xx | X.XX |
| Median duration (days) | X.XX | X.XX |
| Minimum duration (days) | x.xx | X.XX |
| Maximum duration (days) | X.XX | X.XX |

### 13.12.22. Example Shell 22

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of Re-hospitalization Within 30 days of Index Exacerbation

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Re-hospitalization Within 30 days | Yes | 97 (97%) | 19 (19%) |
| | No | 3 (3%) | 81 (81%) |

# 13.12.23. Example Shell 23


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Subsequent Exacerbation Treatment

| | Treatment A (N=81) | Treatment B (N=79) |
|-------------------------|--------------------|--------------------|
| Subsequent exacerbation | 70 (86%) | 50 (63%) |
| ocs | X (x%) | X (x%) |
| Antibiotics | x (x%) | x (x%) |
| OCS and antibiotics | X (x%) | X (x%) |

### 13.12.24. Example Shell 24

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of Time from Resolution of Index Exacerbation to Next Exacerbation

| | Treatment A (N=100) | Treatment B (N=100) |
|-------------------------|---------------------|---------------------|
| Subsequent exacerbation | x.xx | X.XX |
| Mean duration (days) | x.xx | X.XX |
| SD | X.XX | X.XX |
| Median duration (days) | X.XX | x.xx |
| Minimum duration (days) | X.XX | x.xx |
| Maximum duration (days) | X.XX | x.xx |

### 13.12.25. Example Shell 25


Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of ECG Abnormalities for Participants with Any Abnormal Clinically Significant ECG Interpretation

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Visit 2 (Day 1) | | |
| Abnormal - Clinically significant | 10 (10%) | 15 (15%) |
| Any finding | 5 (50%) | 5 (33%) |
| ST depression | 5 (50%) | 5 (33%) |
| Short PR Interval | 0 | 5 (33%) |
| T wave inversion | 0 | 5 (33%) |

Includes Scheduled, unscheduled and Early Withdrawal visits. Participants may have more than one abnormality at each visit.

### 13.12.26. Example Shell 26


Population: Intent-to-Treat/Safety/Other study specific

Table X

Statistical Analysis of Change from Baseline in FEV1 (mL) (Dose Response Model)
Measured post-bronchodilator

| | Placebo<br>(N=xx) | DNX 5mg<br>(N=xx) | DNX 10mg<br>(N=xx) | DNX 25mg<br>(N=xx) | DNX 35mg<br>(N=xx) | DNX 50mg (N=xx) |
|---|---|---|---|---|---|---|
| n [1] | XX | XX | xx | xx | xx | xx |
| Posterior Adj. Median Change<br>95% HPD Credible Interval | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) |
| Active - Placebo<br>Posterior Adj. Median<br>Difference | | x.xx | x.xx | x.xx | x.xx | x.xx |
| 95% HPD Credible Interval | | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) |
| Prob(Difference>0) Predictive probability (%) [2] [only if required] | | xx% | xx% | xx% | xx% | xx% |

<sup>[1]</sup> Number of subjects with data contributing to the analysis.

<sup>[2]</sup> Predictive posterior probability of success at end of study, where success is Pr(Difference>0)>90%. Note: Model fitted was a....[insert as appropriate].

### 13.12.27. Example Shell 27

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of QTc(F) (msec) Categories

| | Trea<br>(N=1 | tment A<br>00) | Trea<br>(N=1 | tment B<br>00) |
|---|---|---|---|---|
| Screening | | | | |
| n | XX | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |
| Day 1 (Baseline) | | | | |
| n | XX | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |
| Day 14 | | | | |
| n | XX | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |

### 13.12.28. Example Shell 28

>30

Protocol: ABC123456
Population: Safety

Visit 2 (Day 1) Type of cough: Single cough Treatment A (N=100)Did subject experience event [1]? 12 (24%) Cough severity Mild 6 (50%) Moderate 5 (42%) Severe 1 (8%) Time to onset of PI cough (minutes) 0 - 12 (17%) >1-2 3 (25%) >2-3 4 (33%) >3-4 3 (25%) >4-5>5 Duration of PI cough (minutes) 7 (58%) >1 - 2 2 (17%) >2 - 3 3 (25%) >3 - 4 >4 - 5 >5 - 10 >10 - 30

[1] Percentages are calculated using the number of subjects evaluated at visit as the denominator.

2019N398117\_00 200879

All other percentages are calculated using the number of subjects with particular cough type at visit as the denominator.


Population: Safety

| Visit 2 (Day 1) Type of cough: Single cough | Treatment A (N=100) |
|----------------------------------------------|---------------------|
| Number of subjects reporting cough as AE/SAE | 4 (33%) |
| Mild | 2 (17%) |
| Moderate | 2 (17%) |
| Severe | 0 |

### 2019N398117\_00 200879


Population: Safety

#### 

| Visit 2 (Day 1) Type of cough: Intermittent cough | Treatment A<br>(N=100) |
|---|---|
| Did subject experience event [1]? | 11 (22%) |
| Cough severity | |
| Mild | 2 (18%) |
| Moderate | 6 (55%) |
| Severe | 3 (27%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 1 (9%) |
| >1-2 | 4 (36%) |
| >2-3 | 6 (55%) |
| >3-4 | 0 |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 0 |
| >1 - 2 | 3 (27%) |
| >2 - 3 | 6 (55%) |
| >3 - 4 | 1 (9%) |
| >4 - 5 | 0 |
| >5 - 10 | 0 |
| >10 - 30 | 1 (9%) |
| >30 | 0 |

### 2019N398117\_00 200879


Population: Safety

| Visit 2 (Day 1) Type of cough: Intermittent cough | Treatment A (N=100) |
|---------------------------------------------------|---------------------|
| Number of subjects reporting cough as AE/SAE | 5 (45%) |
| Mild | 1 (9%) |
| Moderate | 2 (18%) |
| Severe | 2 (18%) |


Population: Safety

### 

| Did subject experience event [1]? $4$ (8%) |
|--------------------------------------------|
| Cough severity |
| Mild 1 (25%) |
| Moderate 2 (50%) |
| Severe 1 (25%) |
| 1 (200) |
| Time to onset of PI cough (minutes) |
| 0-1 3 (75%) |
| >1-2 |
| >2-3 |
| >3-4 |
| >4-5 |
| >5 |
| Duration of PI cough (minutes) |
| <=1 0 |
| >1 - 2 0 |
| >2 - 3 0 |
| >3 - 4 1 (25%) |
| >4 - 5 1 (25%) |
| >5 - 10 0 |
| >10 - 30 1 (25%) |
| >30 1 (25%) |

2019N398117\_00 200879


Population: Safety

Visit 2 (Day 1)

| Type of cough: Continuous cough | Treatment A (N=100) |
|---|---|
| Number of subjects reporting cough as AE/SAE<br>Mild | 2 (50%)<br>1 (25%) |
| Moderate<br>Severe | 1 (25%)<br>0 |

REPEAT FOR EACH VISIT

# 13.12.29. Example Shell 29

Protocol: MID200879 

Population: Intent-to-Treat

Listing X

Listing of Subjects who Received Incorrect Medication

| Randomized<br>Treatment | Centre/<br>Subj | Start<br>Date of<br>Dosing | End<br>Date of<br>Dosing | Duration<br>(Days) | Dispense Visit | Dispense<br>Date | Actual<br>Treatment<br>Dispensed |
|---|---|---|---|---|---|---|---|
| GSK2269557 500 mcg | PPD | xxxxxxxx | XXXXXXXX | XX | Visit 3 (Week 0) | XXFEB2013 | GSK2269557 500 mcg |
| | | XXXXXXXXX<br>XXXXXXXXX | XXXXXXXXX<br>XXXXXXXXX | XX<br>XX | Visit 5 (Week 4) Visit 6 (Week 8) | | GSK2269557 100 mcg<br>GSK2269557 500 mcg |

### 13.12.30. Example Shell 30


Population: Intent-to-Treat/Safety/Other study specific

 $Figure \ X \\ Kaplan-Meier \ Plot \ of \ Time \ to \ Next \ On-treatment \ Exacerbation \ During \ the \ 12-Week \ Treatment \ Period$ 



## 13.12.31. Example Shell 31


Population: Intent-to-Treat/Safety/Other study specific

Figure X
Plot of Repeated Measures Model of Change from Baseline in FEV1 Measured Post-bronchodilator



### 13.12.32. Example Shell 32

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Efficiency Ratio for Possible Adaptions to Randomization Ratio

| | Median | 10 <sup>th</sup> Percentile |
|---|---|---|
| Design 1: Add 25mcg dose | XX | XX |
| Design 2: Add 25mcg dose, drop 500mcg dose | XX | XX |
| Design 3: Add 25mcg dose, drop 250 mcg and 500 mcg doses | XX | XX |
| Design 4: Drop 12.5mcg dose | XX | XX |
| Design 5: Drop 12.5mcg and 50mcg doses | XX | XX |

### 13.12.33. Example Shell 33


Population: Safety

Table X
Summary of Post-Inhalation (PI) Cough at Any Visit

| | | acebo<br>=43) | 50 | mcg | 100 | | 250 | K2269557<br>) mcg<br>=16) | 500 | (2269557<br>) mcg<br>=14) | 750 | 2269557<br>mcg<br>:42) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Did subject experience PI cough at any vi | sit | ? | | | | | | | | | | |
| Yes | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) |
| No | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) |
| Maximum Severity of cough | | | | | | | | | | | | |
| Mild | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | X | (xx%) |
| Moderate | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx) | Χ | (xx%) | Χ | (xx%) |
| Severe | 0 | | 0 | | Χ | (xx%) | 0 | | 0 | | Χ | (xx%) |
| Maximum Duration of PI cough (minutes)[1 | ] | | | | | | | | | | | |
| Mean | Х | | Х | | Х | | Х | | Х | | Х | |
| SD | X | | X | | Х | | Х | | X | | X | |
| Median | X | | X | | Х | | Х | | X | | X | |
| Minimum | X | | X | | Х | | Х | | X | | X | |
| Maximum | Х | | X | | Х | | X | | Х | | Х | |
| Number of occurrences of PI cough | | | | | | | | | | | | |
| 0 | Х | | Х | | Х | | Х | | Х | | Х | |
| 1 | Х | | Х | | Х | | Х | | Х | | Х | |
| 2 | Х | | X | | Х | | X | | Х | | X | |
| 3 | Х | | X | | Х | | X | | Х | | X | |
| 4 | X | | Х | | Х | | Х | | Х | | X | |

<sup>[1]</sup> Duration from the maximum severity cough

### 13.12.34. Example Shell 34

Protocol: ABC123456 Population: Safety


Figure X Plot of Laboratory Data at Screening



# 13.12.35. Example shell 35

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Missing On-treatment EXACT-PRO data

| | Placebo<br>(N=300) | GSK2269557<br>50 mcg<br>(N=100) | GSK2269557<br>100 mcg<br>(N=100) | GSK2269557<br>250 mcg<br>(N=100) | GSK2269557<br>500 mcg<br>(N=100) | GSK2269557<br>750 mcg<br>(N=300) |
|---|---|---|---|---|---|---|
| No. subjects missing >4 consecutive days | X (xx%) | X (xx%) | X (xx%) | X (xx%) | X (xx%) | X (xx%) |
| Number of missing days | | | | | | |
| Mean | X.xx | X.xx | X.xx | X.xx | X.xx | X.xx |
| Median | X.xx | X.xx | X.xx | X.xx | X.xx | X.xx |
| Minimum | X.xx | X.xx | X.xx | X.xx | X.xx | X.xx |
| Maximum | X.xx | X.xx | X.xx | X.xx | X.xx | X.xx |

### 13.12.36. Example Shell 36

Example EX1

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of Exposure to Study Treatment

| | | Treatment A (N=100) | <pre>Treatment B (N=100)</pre> |
|---|---|---|---|
| Time on Study Treatment(days) | n | 97 | 100 |
| | Mean | 15.6 | 11.2 |
| | SD | 13.23 | 9.46 |
| | Median | 11.5 | 8.0 |
| | Min. | 1 | 1 |
| | Max. | 64 | 50 |
| | < 28 days | 20 (21%) | 20 (20%) |
| | 28 days to 42 days | 50 (52%) | 50 (50%) |
| | 43 days to 56 days | 10 (10%) | 10 (10%) |
| | 57 days to 70 days | xx (xx%) | xx (xx%) |
| | >70 days | Xx (xx%) | Xx (xx%) |

#### The GlaxoSmithKline group of companies

200879

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title

: Reporting and Analysis Plan for Phase IIb, Randomized (Stratified), Double-Blind (Sponsor Open), Parallel-Group, Placebo-Controlled, Dose-Finding Study of Nemiralisib (GSK2269557) Added to Standard of Care (SoC) Versus SoC Alone in Participants Diagnosed with an Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)

Compound Number : GSK2269557

Effective Date : 08-MAY-2018

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200879 and at the planned interim analyses.
- This RAP is intended to describe the efficacy, safety and pharmacokinetic analyses required for the study.
- This version of the RAP includes amendments to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

RAP Author(s): PPD

Statistics Leader, (Respiratory Clinical Statistics)

| Approver | Date | Approval Method |
|---|---|---|
| TA Director (Respiratory Clinical Statistics) | 08-MAY-2018 | Email |
| PPD | | |
| Programming Manager (Respiratory Clinical Programming) | 03-MAY-2018 | Email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### The GlaxoSmithKline group of companies

200879

### **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Programmer (Respiratory Clinical Programming) | 02-MAY-2018 | Email |
| Clinical Development Director (Respiratory) | 03-MAY-2018 | Email |
| Clinical Development Manager (Respiratory) | 01-MAY-2018 | Email |
| Medical Director (Global Clinical Safety and Pharmacovigilance) | 01-MAY-2018 | Email |
| PPD Manager, Clinical Pharmacology (Clinical Pharmacology Modelling and Simulation) | 01-MAY-2018 | Email |
| Director, Patient Centred Outcomes (Value Evidence & Outcomes) | 03-MAY-2018 | Email |

200879

### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | N | 8 |
| 2. | CLIMA | | KEY PROTOCOL INFORMATION | Q |
| ۷. | 2.1. | | Objective(s) and Endpoint(s) | |
| | 2.1. | Study C | Design | 11 |
| | ۷.۷. | Study L | /esigit | |
| 3. | PLAN | NED ANA | ALYSES | 11 |
| - | 3.1. | | Analyses | |
| | | 3.1.1. | Futility analyses | |
| | | | 3.1.1.1. Futility rules | |
| | 3.2. | Final Ar | nalyses | |
| 4. | A N I A I | Veie DO | PULATIONS | 15 |
| 4. | 4.1. | | Deviations | |
| | 4.1. | Protoco | Deviations | 15 |
| 5. | CONS | SIDERAT | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CON\ | | IS | |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | |
| | 5.3. | | ntre Studies | |
| | 5.4. | | ation of Covariates and Subgroups | |
| | | 5.4.1. | Covariates | |
| | | 5.4.2. | Examination of Subgroups | 18 |
| | 5.5. | | Considerations for Data Analyses and Data Handling | 10 |
| | | Conven | 10015 | 19 |
| 6. | STUD | | LATION ANALYSES | |
| | 6.1. | Overvie | ew of Planned Study Population Analyses | |
| | | 6.1.1. | Concomitant medications | 19 |
| 7 | | \ | ALVOEO | 00 |
| 7. | | | ALYSES | |
| | 7.1. | 7.1.1. | / Efficacy Analyses | |
| | | 7.1.1.<br>7.1.2. | Primary Endpoint Primary Statistical Analyses | |
| | | 1.1.2. | 7.1.2.1. Model Checking & Diagnostics | |
| | | 7.1.3. | Sensitivity and Supportive Analyses | |
| | | 7.1.4. | Subgroup Analyses | |
| | 7.2. | | lary Efficacy Analyses | |
| | , . <u>-</u> . | | Rate of exacerbations | |
| | | | 7.2.1.1. Statistical analyses | |
| | | | 7.2.1.2. Subgroup analyses | |
| | | | 7.2.1.3. Exploratory analyses | |
| | | 7.2.2. | Time to next exacerbation | |
| | | | 7.2.2.1. Statistical analyses | |
| | | | 7.2.2.2. Subgroup analyses | |
| | | 7.2.3. | Change from baseline in Clinic Visit trough FEV <sub>1</sub> | |
| | | | 7.2.3.1. Statistical Analyses | |
| | | | 7.2.3.2. Subgroup analyses | |
| | | 7.2.4. | Change from hospital discharge in clinic visit trough FEV <sub>1</sub> . | 27 |

200879

| | | | 7.2.4.1. Statistical analyses | 27 |
|---|---|---|---|---|
| | | 7.2.5. | EXAcerbations of Chronic Pulmonary Disease Tool - | |
| | | | Patient Reported Outcome (EXACT) | 27 |
| | | | 7.2.5.1. Proportion of participants achieving EXACT- | |
| | | | defined recovery from index exacerbation | 28 |
| | | | 7.2.5.2. Time to EXACT-defined recovery from index | |
| | | | exacerbation | 29 |
| | | | 7.2.5.3. Severity of subsequent HCRU-defined | |
| | | | exacerbation(s) defined by EXACT | 29 |
| | | | 7.2.5.4. Statistical analyses | 29 |
| | | | 7.2.5.5. Subgroup analyses | 30 |
| | | | 7.2.5.6. Sensitivity and supportive analyses | |
| | | 7.2.6. | COPD Assessment Test (CAT) | |
| | | 7.2.0. | 7.2.6.1. Proportion of responders using the CAT | 30 |
| | | | 7.2.6.2. Change from baseline in CAT Total Score | |
| | | | 7.2.6.3. Statistical analyses | |
| | | | 7.2.6.4. Subgroup analyses | |
| | | 7.2.7. | St. George's Respiratory Questionnaire for COPD | |
| | | 1.2.1. | Patients (SGRQ-C) | 22 |
| | | | 7.2.7.1. Proportion of responders on the SGRQ Total | 32 |
| | | | Score | 22 |
| | | 700 | 7.2.7.4. Subgroup analyses | |
| | | 7.2.8. | Rescue medication use | 33 |
| | | | 7.2.8.1. Rescue medication use via the clip-on | 0.4 |
| | | | Propeller Sensor for MDI | 34 |
| | 7.0 | | 7.2.8.2. Statistical analyses | |
| | 7.3. | | tory Efficacy Analyses | |
| | | 7.3.1. | Change from Day 84 in Clinic Visit trough FEV <sub>1</sub> | |
| | | | 7.3.1.1. Statistical analysis | |
| | | 7.3.2. | | |
| | | 7.3.3. | Measures of HCRU related to exacerbations | 35 |
| | | | 7.3.3.1. Re-hospitalisation within 30 days of index | |
| | | | exacerbation | 36 |
| | | | 7.3.3.2. Time from resolution of index exacerbation to | |
| | | | next exacerbation | |
| | | | 7.3.3.3. Subsequent exacerbation treatment type | |
| | | 7.3.4. | Compliance | 36 |
| | | | 7.3.4.1. Number of actuations of double-blind study | |
| | | | treatment measured by the clip-on Propeller | |
| | | | Sensor | 37 |
| | | 7.3.5. | Inflammatory/infective markers in blood and sputum in | |
| | | | relation to acute exacerbation of COPD | 37 |
| | | 7.3.6. | Other spirometry measurements | 37 |
| | | 7.3.7. | Other symptoms suggestive of exacerbation | |
| | | 7.3.8. | Classification of exacerbating COPD participants and | |
| | | - | prediction of response to nemiralisib using machine | |
| | | | learning techniques | 37 |
| 8. | SAFE | TY ANAL | YSES | 37 |
| | 8.1. | | e Events Analyses | |
| | | | • | |

| | | | | 2 | 00879 |
|---|---|---|---|---|---|
| | | 8.1.1. | 8.1.1.1. Po | nts of Special Interest<br>ost-inhalation Cough Immediately Following | |
| | 8.2. | | aboratory Ana | osinglyses | 38 |
| | 8.3.<br>8.4. | | | | |
| 9. | PHARI<br>9.1. | | | SES | |
| | 9.2. | | | easures | |
| 10. | | | | tic Parameters | |
| 11 | | | | MACODYNAMIC ANALYSES | |
| | | | | WAGOD HANNIO ANALTOLO | |
| 13. | 13.1. | Appendix<br>Protocol | 1: Protocol D | eviation Management and Definitions for Per | 41 |
| | 13.2. | 13.1.1. | Exclusions fro | om Per Protocol Populationnt Windows | 41 |
| | | 13.2.1. | Definitions of 13.2.1.1. Ho | Assessment Windows for Analysesospital discharge | 42<br>42 |
| | 13.3. | | 3: Study Pha | KACT-Defined Recovery for CAT Triggerses and Treatment Emergent Adverse | |
| | | 13.3.1. | | S | |
| | | | 13.3.1.1. 12 | 2-Week Treatment Period | 43 |
| | | | | 2-Week Follow-Up Period | |
| | | 13.3.2. | | 3 | |
| | | 13.3.3. | | udy Phases for Concomitant Medicationnergent Flag for Adverse Events | |
| | 13.4. | | | ay Standards & Handling Conventions | |
| | | 13.4.1. | | ocess | |
| | | 13.4.2. | Reporting Sta | andards | 44 |
| | | 13.4.3. | | andards for Pharmacokinetic | |
| | 13.5. | | | nd Transformed Data | |
| | | 13.5.1.<br>13.5.2. | | tion | |
| | | 13.5.2. | | | |
| | 13.6. | | | Standards for Missing Data | |
| | | 13.6.1. | | ithdrawals | |
| | | 13.6.2. | | lissing Data | |
| | | | | andling of Missing and Partial Dates | |
| | 13.7. | | | Potential Clinical Importance | |
| | | 13.7.1.<br>13.7.2. | • | alues | |
| | | 13.7.2. | | | |
| | 13.8. | | | Pharmacokinetic (PopPK) Analyses | |
| | | | | narmacokinetic (PopPK) Methodology | |

200879

| | 13.8.2. | Population Pharmacokinetic (PopPK) Dataset | |
|---|---|---|---|
| | | Specification | .51 |
| 13.9. | Appendix | (9: Pharmacokinetic / Pharmacodynamic Analyses | .53 |
| | | Pharmacokinetic/Pharmacodynamic Methodology | |
| 13.10. | | c 10: Abbreviations & Trade Marks | |
| | 13.10.1. | Abbreviations | 54 |
| | | Trademarks | |
| 13.11. | | c 11: List of Data Displays | |
| | | Data Display Numbering | |
| | 13.11.2. | Mock Example Shell Referencing | 56 |
| | 13.11.3. | Deliverables | 56 |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | 10.11.0. | 13.11.5.1. Efficacy tables for Interim Analysis 1 | |
| | | 13.11.5.2. Efficacy tables for Interim Analysis 2 | |
| | | 13.11.5.3. Efficacy tables for End of Treatment Interim | |
| | | Analysis and SAC | 65 |
| | 13 11 6 | Efficacy Figures | 76 |
| | 10.11.0. | 13.11.6.1. Efficacy Figures for Interim Analysis 1 | |
| | | 13.11.6.2. Efficacy Figures for Interim Analysis 2 | |
| | | 13.11.6.3. Efficacy Figures for End of Treatment Interim | |
| | | Analysis and SAC | 79 |
| | 13 11 7 | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 13 12 | Annendiy | (12: Example Mock Shells for Data Displays | 20 |
| 15.12. | 13 12 1 | Example shell 1 | 80 |
| | | Example Shell 2 | |
| | | Example shell 3 | |
| | | Example Shell 4 | |
| | | Example Shell 5. | |
| | | Example Shell 6 | |
| | | Example Shell 7 | |
| | | Example Shell 8 | |
| | | Example Shell 9 | |
| | | Example Shell 10 | |
| | | Example Shell 111 | |
| | | Example Shell 121 | |
| | | Example shell 13 | |
| | | Example Shell 14 | |
| | | Example Shell 151 | |
| | | Example shell 16 | |
| | | Example Shell 171 | |
| | | Example shell 18 | |
| | | Example Shell 19 | |
| | | Example Shell 201 | |
| | | Example Shell 21 | |
| | | Example Shell 221 Example Shell 23 | |
| | | Example Shell 24 | |
| | 10.14.44 | . LAGITIVIE OTICII 44 | 110 |

200879

| 13.12.25.Example Shell 25 | 119 |
|----------------------------|-----|
| 13.12.26.Example Shell 26 | |
| 13.12.27.Example Shell 27 | |
| 13.12.28.Example Shell 28 | 122 |
| 13.12.29 Example Shell 29 | 128 |
| 13.12.30. Example Shell 30 | 129 |
| 13.12.31.Example Shell 31 | 130 |
| 13.12.32.Example Shell 32 | 131 |
| 13.12.33.Example Shell 33 | 132 |
200879

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 200879.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterise the dose response of<br>nemiralisib administered in addition to<br>SoC compared with placebo and SoC<br>in participants diagnosed with an<br>acute moderate or severe<br>exacerbation of COPD | <ul> <li>Change from baseline in Clinic Visit trough forced<br/>expiratory volume in one second (FEV<sub>1</sub>) at Day 84<br/>measured post-bronchodilator</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To characterise the dose response and efficacy of nemiralisib administered in addition to SoC compared with placebo and SoC in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>Rate of moderate and severe exacerbations over the 12-Week Treatment Period</li> <li>Time to next moderate/severe exacerbation following index exacerbation</li> <li>Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days 14, 28, 56, and 84 (Day 84: post-bronchodilator is the primary endpoint; pre-bronchodilator is a secondary endpoint) and at hospital discharge (only for participants who are hospitalized for the index exacerbation)</li> <li>Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days, 14, 28, 56, and 84 (in participants hospitalized for index exacerbation only)</li> </ul> |
| To evaluate the treatment effect of nemiralisib in addition to SoC compared with placebo and SoC on symptoms indicative of an exacerbation and on health status using Patient-Reported Outcomes (PROs) in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>EXAcerbations of Chronic Pulmonary Disease Tool (EXACT-PRO)</li> <li>Proportion of participants achieving the EXACT definition of recovery from the index exacerbation by Days 14, 28, 56, and 84</li> <li>Time to recovery from index exacerbation</li> <li>Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT</li> <li>COPD Assessment Test (CAT)</li> <li>Proportion of responders using the CAT at Treatment Days 28, 56, and 84, and following EXACT defined recovery from the index exacerbation</li> <li>Change from baseline (Day 1) in CAT total score at Days 28, 56, and 84 and following EXACT defined recovery from the index exacerbation</li> </ul> |

200879

| Objectives | Endpoints |
|---|---|
| To evaluate the usage of rescue<br>medication in patients diagnosed with<br>an acute moderate or severe<br>exacerbation of COPD | St. George's Respiratory Questionnaire (SGRQ) Total Score Proportion of responders on the SGRQ total score as measured by the SGRQ for COPD Patients (SGRQ-C) at Days 28, 56, and 84 Change from baseline (Day 1) in SGRQ total score at Days 28, 56, and 84 Rescue medication use (occasions/day), averaged over each week of treatment and over the 84-day treatment period The percentage of rescue-free days (24-hour periods) during each week of treatment and over the 84-day |
| To evaluate the population pharmacokinetics of nemiralisib in participants diagnosed with an acute moderate or severe exacerbation of COPD | treatment period Plasma nemiralisib concentrations and derived PK parameters (e.g., area under the curve [AUC (0-24) and AUC(0-t)], maximum concentration [Cmax], time at maximum concentration [Tmax], Ctrough) as appropriate will be collected in a subset of randomized participants (approximately 300) at selected sites as follows: trough (pre-dose) for the study treatment and post-dose for the study treatment from 0-1 hour and >1 to 6 hours on Days 14 and 28 of the 12-Week Treatment Period |
| To assess the safety and tolerability of<br>nemiralisib and placebo in participants<br>diagnosed with an acute moderate or<br>severe exacerbation of COPD | <ul> <li>Incidence of adverse events (AEs; including serious AEs and AE of Special Interest [AESI])</li> <li>Vital signs (pulse rate, systolic and diastolic blood pressure) (measured at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>12-lead electrocardiogram (ECG) assessments (performed at clinic Visits 1 [Screening], 3 [Day 14], 6 [Day 84], and 7 [Day 112] or Early Withdrawal Visit)</li> <li>Clinical laboratory tests (hematology and chemistry; performed at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>Incidence of COPD exacerbations</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To further characterize the dose<br>response, and efficacy, of nemiralisib<br>administered in addition to SoC<br>compared with placebo and SoC in<br>participants diagnosed with an acute<br>moderate or severe exacerbation of<br>COPD | <ul> <li>Rate of mild exacerbations over the 12-Week Treatment Period</li> <li>Rate of all exacerbations (mild, moderate and severe combined) over the 12-Week Treatment Period</li> <li>Time to next exacerbation (mild, moderate and severe combined)</li> </ul> |

200879

| Objectives | Endpoints |
|---|---|
| To evaluate the treatment effect of<br>nemiralisib in addition to SoC<br>compared with placebo and SoC on<br>symptom stability following an<br>exacerbation using Patient-Reported<br>Outcomes in participants diagnosed<br>with an acute moderate or severe<br>exacerbation of COPD | Stability of symptoms post recovery measured using E-RS:COPD (Evaluating Respiratory Symptoms in COPD) and subscales from Randomization (Visit 2) to Day 84 (Visit 6) |
| To explore the PK/PD relationship for<br>nemiralisib | Relationship between drug exposure and<br>Pharmacodynamic responses (e.g. efficacy, heart rate,<br>clinical laboratory analytes and blood biomarkers) in the<br>PK subset of participants (approximately 300) at selected<br>sites |
| To evaluate the treatment effect of<br>nemiralisib in addition to SoC<br>compared with placebo and SoC on<br>HCRU in participants who experience<br>a severe exacerbation of COPD | <ul> <li>Measures of HCRU related to severe exacerbations (e.g.,<br/>hospitalizations, length of hospital stay, re-hospitalization<br/>within 30 days, number of Emergency Room [ER] visits,<br/>etc.)</li> </ul> |
| To evaluate compliance with study treatment | Number of actuations of the double-blind study treatment<br>as measured by the clip-on Propeller Sensor (for<br>countries where the Propeller Sensor for ELLIPTA is<br>available) |
| To evaluate inflammatory markers in<br>blood in relation to acute exacerbation<br>of COPD | <ul> <li>Blood samples collected at Screening through Visit 7 (as part of the clinical laboratory blood samples) for analysis of blood eosinophil counts and inflammatory mediators</li> <li>Blood samples for analysis of inflammatory biomarkers (including but not limited to: high sensitivity C-reactive protein [hs-CRP], chemokine interferon-γ inducible protein 10 kDa (CXCL10)], and procalcitonin) collected at Visit 1 (Screening)</li> </ul> |
| To evaluate inflammatory and infective markers in sputum in relation to acute exacerbation of COPD | Spontaneous sputum sample for analysis of inflammatory<br>and infective markers collected at Screening/Day 1 (pre-<br>dose) and Day 56 in participants who are willing and able<br>to provide a sample |
| To evaluate the potential post-<br>treatment impact of double-blind study<br>treatment during the 12-Week Post-<br>Treatment Follow-Up Period | <ul> <li>Change from baseline (Day 84) in Clinic Visit trough FEV1 measured pre- and postbronchodilator at Day 112, 140 and 168</li> <li>Rate of moderate and severe COPD exacerbation(s) during the 12-Week Follow-Up Period</li> <li>Rate of moderate and severe COPD exacerbation(s) over the 24 week study duration</li> <li>Time to next exacerbation following cessation of double blind study treatment</li> <li>Proportion of responders using the CAT at Days 112 and 168</li> <li>Change from baseline (Day 1) in CAT Total score at Days 112 and 168</li> <li>Proportion of responders on the SGRQ Total Score as measured by the SGRQ-C at Days 112 and 168</li> <li>Change from baseline (Day 1) in SGRQ total score at</li> </ul> |

200879

| Objectives | En | dpoints |
|------------|----|-----------------------------------------------------|
| | | Days 112 and 168 |
| | • | Severity of subsequent HCRU exacerbation defined by |
| | | EXACT |
| | • | E-RS: COPD and subscales from last dose of double- |
| | | blind study treatment |
| | • | Rescue medication use up to Day 112 |

# 2.2. Study Design

This is a Phase IIb, multicenter, randomized, stratified (by index COPD exacerbation severity [moderate or severe] and by whether or not the participant is in the PK Subgroup), double-blind (Sponsor Open), placebo-controlled, parallel-group study in participants who present with an acute moderate or severe exacerbation of COPD requiring Standard of Care (SoC).

This study consists of a Screening Period, a 12-Week Treatment Period and a 12-Week

Post-Treatment Follow-Up Period. Randomization and the first dose of the double-blind study treatment administration (Visit 2/Day 1) should take place in the morning, as soon as possible following determination of eligibility and completion of the baseline measures, including the EXACT-PRO questionnaire for the day of randomization, and FEV<sub>1</sub> measurement and no later than 48 hours after the start of SoC.

PK Subgroup: Sparse PK sampling will be conducted in a subgroup of participants at selected sites. The PK Subgroup will be identical to the main study in terms of the study population, design, and conduct, with the exception of blood draws (3 per visit on Days 14 and 28) for PK analysis.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

Ongoing data reviews of unblinded safety data, conducted by an Internal Safety Review Committee (iSRC), will be performed throughout the trial. Details will be documented in the iSRC charter.

Interim analyses of the primary endpoint and key secondary endpoints to inform internal decision making will be conducted periodically throughout the trial. The first analysis (Interim Analysis 1) is planned to occur when approximately 170 participants complete 28 days of treatment, where approximately 50 of the 170 participants have an index exacerbation defined as severe. A change that could arise from this interim analysis is a specification of the stratification proportions by index exacerbation severity status (moderate or severe). This decision will be based on inspection of all available endpoints at the interim analysis.

Further interim analyses will be performed, depending on the observed recruitment rate. At least one interim analysis of the primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator will be performed to determine whether or not any adjustments to the randomization ratio across doses would help optimize the characterization of the dose response profile for nemiralisib. This analysis (Interim Analysis 2) is planned to occur when approximately 300 participants

200879

complete 84 days of treatment or when approximately 400 participants remain to be randomized, whichever occurs first. Adjustments could include ceasing randomization to an existing dose(s) of nemiralisib and/or modification of the allocation ratios for the existing nemiralisib doses and/or addition of a 25mcg dose. Other changes may include specification of the stratification proportions by index exacerbation severity status.

An interim analysis of efficacy data collected during the Double-Blind Treatment Period will be conducted when the last participant in the study has completed the 12-week Double-Blind Treatment Period (End of Treatment Interim Analysis). The aim of this analysis is to provide GSK with timely data to inform internal decision making, prior to the end of study.

The following table describes the endpoints that will be analysed/summarised at each interim:

| Interim | Purpose of interim | Endpoints |
|---|---|---|
| Interim Analysis 1 | To inform internal decision making | <ul> <li>Change from baseline in FEV<sub>1</sub> at Days 14, 28, and 56 measured pre- and post-bronchodilator</li> <li>Other spirometry measures (percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio</li> <li>On-treatment exacerbations</li> <li>Proportion of participants achieving EXACT-defined recovery by Days 14, 28, 56 and 84</li> </ul> |
| Interim Analysis 2 | To determine if any adjustments to the randomization ratio would help characterize the dose response profile for nemiralisib | Endpoints listed for Interim Analysis 1 and also: Change from baseline in FEV <sub>1</sub> at Day 84 measured pre- and post-bronchodilator Rate of (on-treatment) exacerbations over the 12-Week Treatment Period Time to next (on-treatment) exacerbation during the 12-Week Treatment Period Proportion of responders using the CAT Change from baseline in CAT Total Score Proportion of responders using the SGRQ Change from baseline in SGRQ Total Score Rescue medication use, as measured in eDiary |
| End of Treatment<br>Interim Analysis | To inform internal decision making | Selected Efficacy and Safety endpoints as defined in Appendix 11: List of Data Displays |

The statistical methods of analyses are described in Section 7.

200879

The Respiratory Data Sciences Group will apply machine learning techniques to the interim data to determine if identifiable phenotypic sub-population(s) of COPD participants are present at baseline, and if they result in different responses to Nemiralisib, to predict which participants will respond to Nemiralisib therapy, and to identify/quantify relationship(s) between different endpoints and response measures. Details of these analyses will be described in a separate RAP and results will be reported separately to the Clinical Study Report (CSR).

The following functions will be unblinded to interim analysis data: Clinical Statistics, Clinical Programming and Respiratory Data Sciences Group. Other member of GSK will be unblinded to group level summary data following the interim analyses (as documented internally).

## 3.1.1. Futility analyses

At least one interim analysis for futility will be performed. The first analysis will occur at Interim Analysis 2, i.e. when 300 participants complete 84 days of treatment, or when approximately 400 participants remain to be randomized, whichever occurs first.

Futility will be assessed in a sequential manner.

- 1) Futility will first be assessed for the primary endpoint of change from baseline in FEV<sub>1</sub> at Day 84 by fitting a suitable dose response model, as described in Section 7.1.2.
- 2) If the posterior predictive probability of declaring success for this endpoint is low across all doses, then futility will be assessed for the rate of (on-treatment) exacerbations endpoint.
- 3) If the posterior predictive probability of declaring success for this endpoint is low, then the study may be stopped.

Any decision to stop will be made after a review of all the data summarised/analysed at the time of the interim, including the proportion of participants achieving the EXACT-defined recovery.

## 3.1.1.1. Futility rules

The decision rules for futility are defined as follows.

## Change from baseline in FEV<sub>1</sub> at Day 84

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, across all doses, where success at the end of the trial for change from baseline in FEV<sub>1</sub> is defined as demonstrating >90% posterior probability that the true difference from placebo for any dose of nemiralisib is greater than 0.

200879

## Rate of on-treatment (moderate/severe) exacerbations

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, where success at the end of the trial for rate of exacerbations is defined as demonstrating >80% posterior probability that the true rate reduction on 750 mcg dose versus placebo >0%.

If a different dose arm appears to be more efficacious than the 750 mcg arm, then futility may be assessed using the rate reduction for this arm versus placebo.

The pre-determined rules will act as guidelines for stopping the study for futility. All of the data summarised/analysed at the time of the interim will be reviewed prior to any decision to stop the study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

200879

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE)<br>Population | All participants who are screened for eligibility. | Study Population |
| Modified Intent<br>To treat (MITT)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment.</li> <li>Participants will be analyzed according to the treatment that they were randomized to.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Per Protocol (PP)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment, excluding any participants with an important protocol deviation.</li> <li>Participants will be analyzed according to the treatment that they were randomized to.</li> </ul> | Sensitivity analyses of efficacy |
| Safety Population | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>Participants will be summarised according to the treatment that they actually received. <ul> <li>If participants receive &gt;1 treatment, then they will be summarised according to the most frequently dosed treatment. In cases where the frequency is equal, the participant will be assigned the lowest dose strength of nemiralisib</li> </ul> </li> </ul> | Safety |
| Pharmacokinetic<br>(PK) Population | <ul> <li>All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values).</li> <li>Participants will be summarised according to the treatment that they actually received</li> </ul> | • PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all
  important deviations and deviations which may lead to exclusion from the
  analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

200879

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Randomization System Data I | | | a Displays for Reporting |
| Code | Description | Description | Order in TLF |
| Α | Placebo | Placebo | 1 |
| В | GSK2269557 12.5 mcg | NEMI 12.5 mcg | 2 |
| С | GSK2269557 25 mcg* | NEMI 25 mcg | 3 |
| D | GSK2269557 50 mcg | NEMI 50 mcg | 4 |
| E | GSK2269557 100 mcg | NEMI 100 mcg | 5 |
| F | GSK2269557 250 mcg | NEMI 250 mcg | 6 |
| G | GSK2269557 500 mcg | NEMI 500 mcg | 7 |
| Н | GSK2269557 750 mcg | NEMI 750 mcg | 8 |

<sup>\*</sup> The nemiralisib dose of 25 mcg may be added following the results of an un-blinded interim analysis if further characterization of the lower end of the dose response curve is required.

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. NEMI 12.5 mcg vs Placebo
- 2. NEMI 25 mcg vs Placebo
- 3. NEMI 50 mcg vs Placebo
- 4. NEMI 100 mcg vs Placebo
- 5. NEMI 250 mcg vs Placebo
- 6. NEMI 500 mcg vs Placebo
- 7. NEMI 750 mcg vs Placebo

## 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Post-bronchodilator Baseline  $FEV_1$  is defined as the latest  $FEV_1$  measured prior to the first dose of study treatment and post-bronchodilator.

200879

Pre-bronchodilator Baseline  $FEV_1$  is defined as the latest  $FEV_1$  measured prior to the first dose of study treatment and pre-bronchodilator.

Baseline CAT Total Score is defined as CAT Total Score measured prior to the first dose of study treatment on Day 1.

Baseline SGRQ Total Score is defined as SGRQ Total Score measured prior to the first dose of study treatment on Day 1.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

A centred baseline will be derived for each participant by subtracting the mean baseline across all participants from each participant's baseline value. The 'centred' baseline may be used instead of Baseline in the statistical analyses to aid convergence.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site and country.

## 5.4. Examination of Covariates and Subgroups

#### 5.4.1. Covariates

The list of covariates may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates of clinical interest may also be considered. The decision to include covariates in the model will be based on their impact on the model fit and will be detailed in the CSR.

A centred covariate will be derived for each participant by subtracting the mean covariate across all participants from each participant's covariate value. The 'centred' covariate may be used in place of the covariate in the statistical analyses to aid convergence.

200879

| Covariate | Details |
|---|---|
| Index exacerbation severity | Categorical variable (Moderate or Severe) derived using the stratification variable from the randomisation system. |
| Age (at screening) | Continuous variable derived as described in Section 13.6.2.1 |
| BMI | Continuous variable derived using Height and Weight variables collected in eCRF: BMI = Weight (kg) / (Height (m)) <sup>2</sup> |
| Gender | Categorical variable (Male or Female), collected in eCRF |
| Country | Categorical variable |
| Smoking status | Categorical variable (Current or Former), collected in eCRF |
| Baseline COPD maintenance therapy type | Categorical variable derived depending on data observed. Possible categories of interest are: Monotherapy vs. Dual therapy vs. Triple therapy |
| Index exacerbation type | Categorical variable: New or Relapse, derived using the question: "Other than the current prescription, for the index exacerbation, has the subject received oral/systemic corticosteroids and/or antibiotics for a COPD exacerbation within the last 7 days?" in the eCRF: New = No Relapse = Yes |
| Number of exacerbations in the previous 12 months | Categorical variable derived from "Total number of COPD exacerbations in the last 12 months" in the eCRF. Possible categories of interest are: 0 vs. 1 vs. ≥2 |

## 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Index exacerbation severity | Moderate vs. Severe |
| Baseline COPD maintenance therapy type | Possible categories of interest are: Monotherapy vs. Dual therapy vs. Triple therapy |
| Index exacerbation type | New vs. Relapse |
| Number of exacerbations in the previous 12 months | Possible categories of interest are: 0 vs. 1 vs. ≥2 |
| Gender | Male vs. Female |
| Smoking status | Current vs. Former |

200879

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 13.2 | Appendix 2: Assessment Windows |
| Section 13.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| Section 13.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 13.5 | Appendix 5: Derived and Transformed Data |
| Section 13.6 | Appendix 6: Reporting Standards for Missing Data |
| Section 13.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "APE" and/or "MITT" populations, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

## 6.1.1. Concomitant medications

Concomitant medications will be summarised by treatment group. Separate summaries of Baseline and On-treatment (Step-up) COPD Maintenance Therapy, and duration of OCS use will also be presented.

Additional summaries or sensitivity analyses of on-treatment COPD maintenance therapy (step-up therapy) may be performed if the data indicate that further investigation is warranted.

200879

## 7. EFFICACY ANALYSES

Details of the outputs are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Further details for use in the endpoint derivations below can be found in Appendix 5: Derived and Transformed Data.

## 7.1. Primary Efficacy Analyses

## 7.1.1. Primary Endpoint

The primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator is defined as:

FEV<sub>1</sub> measured prior to dosing and post-bronchodilator on Day 84 – Post-bronchodilator Baseline FEV<sub>1</sub>

## 7.1.2. Primary Statistical Analyses

The primary endpoint will be analysed by fitting a suitable dose response model. The following models will be fitted, and the one that gives the best fit to the data will be selected: Bayesian 4-parameter  $E_{max}$  dose response model, 3-parameter  $E_{max}$  model and a Log-linear model.

The 4-parameter  $E_{max}$  dose response model will take the form:

Change from baseline FEV<sub>1</sub> = 
$$(E0 + a_1 * baseline) + \frac{(E_{max} + b_1 * baseline) * Dose^{\gamma}}{ED50^{\gamma} + Dose^{\gamma}}$$

The 3-parameter  $E_{max}$  dose response model will take the form:

Change from baseline 
$$FEV_1 = (E0 + a_1 *baseline) + \frac{(E_{max} + b_1 *baseline) *Dose}{ED50 + Dose}$$

Where: E0 =the response at dose = 0 (placebo)

 $E_{max}$  = the maximal response

ED50 =the dose that yields 50% of the maximal response

 $\gamma$  = the slope parameter

a<sub>1</sub>, b<sub>1</sub>, are covariates for explanatory parameters

Initially, normal non-informative priors will be used for the E0,  $a_1$ ,  $a_2$ , and  $E_{max}$  parameters with mean 0 and standard deviation 1E6 L. A functional uniform prior will be used for the ED50 and slope parameters (Bornkamp, 2014), where the prior density for the functional uniform prior is based on all the parameters in the model. An inverse -

200879

gamma prior with shape of 0.001 and scale of 0.001 will be used for the residual variance. However, if a prior distribution appears not to be truly non-informative then alternative prior distributions may be used.

Parameters will be blocked such that the MCMC procedure samples from E0,  $a_1$ ,  $b_1$ , and  $E_{max}$ , first, then the ED50 and slope parameters and then finally the residual variance parameter. For the functional uniform priors, the density will be calculated for values of dose from 0.0001 to 750 in steps of 50 (i.e. 0.0001, 50.0001, 100.0001,..., 750.0001). For the continuous covariates, the density will be calculated from the minimum to the maximum in 10 equal steps. For binary covariates the density will be calculated for values 0 and 1. If the model does not converge including covariates, the model may be fitted with covariates removed.

If the log-linear model is fitted an offset of 1 will be used.

The posterior median change from baseline with 95% Highest Posterior Density (HPD) Credible Intervals, will be presented for each dose along with the adjusted median difference from placebo with 95% HPD, calculated at the mean baseline value across the treatment arms. Posterior probabilities that the true improvement is greater than 0 mL and 75 mL will also be presented. Graphical representation of the dose response across the full dose range will also be produced to allow inference to be made for the non-studied doses based upon the model fit.

#### For the futility analysis:

The predictive probability of success at the end of the study will be calculated (assuming the randomisation ratios remain the same after the interim) for each dose using the formula suggested by Spiegelhalter et al., 2004 as follows:

$$\textit{Predictive probability} = \ 1 - \Phi \Bigg[ \frac{\sqrt{n_1}}{\sqrt{m_1}} \, z_{\text{QS}} - \sqrt{\frac{n_1 + m_1}{m_1}} \, \frac{y_n}{\sigma} \Bigg]$$

Where  $n_1$  is the number of subjects with Day 84 data in the active arm of interest,  $m_1$  is the number of subjects yet to be observed in the active arm of interest,  $y_n$  is the posterior mean difference from placebo from the fitted model, and  $\sigma$  is the standard deviation of the posterior mean difference from placebo.

#### For the possible adaptations at Interim Analysis 2:

If the study is not deemed futile, and either the 4 parameter or 3 parameter  $E_{\text{max}}$  dose response curves has successfully been fitted to the data then adaptation of the randomisation schedule will be considered, to drop, add or amend doses from the randomisation scheme.

The adaptation will be done by comparing the relative information from alternative randomisation schemes with the original randomisation schemes, such to find the design that provides the most information about the dose response relationship. The efficiency ratio (ER) for an alternative scheme comparted to the original, will be calculated as:

200879

$$ER(\theta_{i}) = \left(\frac{|M(\xi_{i},\theta_{i})|}{|M(\xi_{i},\theta_{i})|}\right)^{\frac{1}{p}}, i=1,...,1000$$

Where  $M(\xi, \theta)$  is the information matrix for the design  $\xi$  and model parameters  $\theta = (e\theta, emax, ed50, \gamma, a_1, b_1)^T$ ,  $\xi_1$  is the alternative design one and  $\xi_F$  is the fixed original design, and p is the number of parameters (Dette et al 2008). In order to ensure any adaptation is robust to the variability in the parameter estimates at the interim analysis, 1000 samples will be generated from the posterior distribution of the parameters  $\theta_1, \dots, \theta_{1000}$  and the ER calculated for each set of parameter. Adaptation will then only take place if the median ER is >1.05 and the  $10^{th}$  percentile of the ER is >1. The efficiency ratio will be estimated using the mean baseline value across the population.

The alternative designs that will be considered will depend on the dose response model fitted but could include:

- 1. Add 25mcg dose
- 2. Add 25mcg dose, drop 500mcg dose
- 3. Add 25mcg dose, drop 250 mcg and 500 mcg doses
- 4. Drop 12.5mcg dose
- 5. Drop 12.5 mcg and 50mcg doses

The potential adaption may also be verified in the moderate and severe subgroups to ensure the adaption is beneficial across both groups.

#### 7.1.2.1. Model Checking & Diagnostics

The following list of convergence diagnostics will be applied for each parameter:

- The Monte Carlo Standard Errors (MCSE) should be compared with the standard deviation of the posterior distribution (SD) to ensure that only a fraction of the posterior variability is due to the simulation. The number of samples generated and/or the thinning may be increased to reduce the ratio of the MCSE/SD as deemed necessary.
- The Geweke diagnostic test will be used to assess whether the mean estimates
  have converged by comparing means from the early and latter part of the Markov
  chain using a z-score t-test. Large absolute values of the z-score statistic indicate
  rejection of the null hypothesis of no difference between the mean estimates
  obtained from the early and latter parts of the chain.
- Trace plots of samples versus the simulation index will be visually inspected to assess some aspects of convergence. The centre of the chain should appear stable with very small fluctuations, i.e., the distribution of points should not change as the chain progresses and the posterior mean and variance are relatively constant.
- Autocorrelation plots will be visually inspected to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).

200879

## 7.1.3. Sensitivity and Supportive Analyses

If there are greater than 20% of participants with an important protocol deviation that results in exclusion from the Per Protocol Population, the primary analysis may be repeated using the Per Protocol Population.

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 will also be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant. All post-baseline scheduled visits will be included in the analysis using Day. Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

A further sensitivity analysis may be performed where Baseline  $FEV_1$  is replaced with the  $FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge for participants who were hospitalised for their index exacerbation, i.e. who were randomized with a Severe index exacerbation but kept as Baseline  $FEV_1$  for participants who were randomized with a Moderate index exacerbation.

## 7.1.4. Subgroup Analyses

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will be performed by fitting separate models to each level of the severity subgroup.

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will also be performed by including a treatment-by-severity-by-Day interaction term in the Bayesian Repeated Measures model.

## 7.2. Secondary Efficacy Analyses

#### 7.2.1. Rate of exacerbations

Rate of exacerbation is defined as the frequency of exacerbations (subsequent to the index exacerbation) within the specified time period, for example, the 12-Week Treatment Period or the 24-Week Study Period.

The length of time on treatment or in study, depending on the specified time-period, for each participant will be calculated for each endpoint as follows:

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| Rate of (on-treatment) exacerbations, summarised by: | 12-Week Treatment Period | Time from date of randomisation to date of last dose of study |
| Moderate/severe exacerbations | | treatment |
| Moderate exacerbations | | |
| Severe exacerbations | | |
| All (mild, moderate and | | |

200879

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| severe) exacerbations | | |
| Rate of (on-or off-treatment) exacerbations, summarised by: | 12-Week Treatment Period | Time from date of randomisation to Day 84 (Visit 6) Visit Date. |
| <ul><li>Moderate/severe<br/>exacerbations</li><li>All exacerbations</li></ul> | | For participants who withdraw early from the study: Time from date of randomisation to date of study withdrawal |
| Rate of (off-treatment) exacerbations, summarised by: • Moderate/severe exacerbations • Moderate exacerbations • Severe exacerbations | 12-Week Follow Up Period | Time from date of last dose of study treatment to date of study withdrawal/completion |
| Rate of (on- and off- treatment) exacerbations, summarised by: • Moderate/severe exacerbations • Moderate exacerbations • Severe exacerbations | Full 24-Week Study Period | Time from date of randomisation to date of study withdrawal/completion |

Refer to Section 13.5 for further details regarding the length of time derivation

## 7.2.1.1. Statistical analyses

The rate of exacerbations will be analysed using a Bayesian generalized linear model assuming a negative binomial distribution for the underlying exacerbation rate with a log link function. An offset to account for the length of time on treatment or in study, depending on the specified time-period, for each participant (as described above) will be included in the model as log<sub>e</sub> (length of time).

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The median exacerbation rates for each dose arm per 12 weeks, along with the median ratio in exacerbation rates (nemiralisib/placebo) per 12 weeks for each dose, will be estimated and corresponding 95% HPD credible intervals presented. The probability that the true exacerbation rate ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore estimates of the exacerbation rates for pooled data from 500 mcg plus 750 mcg will also be presented.

200879

#### 7.2.1.2. Subgroup analyses

A subgroup analysis of exacerbation rate by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

## 7.2.1.3. Exploratory analyses

A summary of exacerbation rate by the following groups will be presented and, if feasible, a subgroup analyses may be performed:

- Index exacerbation type (New or Relapse)
- Number of exacerbations in previous 12 months  $(0, 1 \text{ or } \ge 2)$ .

## 7.2.2. Time to next exacerbation

Time to next (on-treatment) exacerbation following index exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation whilst on study treatment. Participants who did not have an exacerbation whilst on study treatment will be censored at the date of their last dose of study treatment.

Time to next (on-or off-treatment) exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation occurring up to Day 84. Participants who have not had an exacerbation during the 12-Week Treatment Period will be censored at Day 84 or the date of study withdrawal, for participants who withdrew from the study prior to Day 84.

Time to next exacerbation following cessation of study treatment is defined as time from the date of last dose of study treatment until the date of onset of the next exacerbation whilst off study treatment during the 12-Week Follow Up Period. Participants who have not had an exacerbation off-treatment will be censored at the date of their last follow up assessment.

Time to next exacerbation will be analysed by severity, as follows:

| Endpoint | Time period |
|---|---|
| Time to next (on-treatment) exacerbation, summarised by: | 12-Week Treatment Period |
| Moderate/severe exacerbations | |
| All (mild, moderate and severe) exacerbations | |
| Time to next (on-or off-treatment) exacerbation, summarised by: | 12-Week Treatment Period |
| Moderate/severe exacerbations | |
| All exacerbations | |
| Time to next exacerbation following cessation of treatment, summarised by: | 12-Week Follow Up Period |
| Moderate/severe exacerbations | |

Refer to Section 13.5 for further details regarding the length of time derivation

200879

#### 7.2.2.1. Statistical analyses

Time to next exacerbation will be analysed using a Bayesian Cox proportional hazards model with the "Efron" method for handling ties.

Kaplan-Meier (KM) estimates of the probability of exacerbation will also be presented.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The hazard ratio and corresponding 95% HPD credible intervals for each nemiralisib dose versus placebo will be presented. The probability that the true hazard ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore an estimate of hazard ratio for pooled data from 500 mcg plus 750 mcg nemiralisib doses versus placebo will also be presented.

## 7.2.2.2. Subgroup analyses

A subgroup analysis of time to exacerbation by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

## 7.2.3. Change from baseline in Clinic Visit trough FEV<sub>1</sub>

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56 measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day X – Post-bronchodilator Baseline  $FEV_1$ 

Where Day X is Day 14, 28, and 56.

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56, 84 measured prebronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day X – Pre-bronchodilator Baseline  $FEV_1$ 

Where Day X is Day 14, 28, 56, and 84.

## 7.2.3.1. Statistical Analyses

Change from baseline in Clinic Visit trough  $FEV_1$  measured post-bronchodilator will be analysed using a dose response model and repeated measures analysis as described for the primary endpoint in Section 7.1.2.

200879

Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured pre-bronchodilator will be analysed using a repeated measures analysis as described in Section 7.1.2

## 7.2.3.2. Subgroup analyses

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will be performed.

## 7.2.4. Change from hospital discharge in clinic visit trough FEV<sub>1</sub>

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> will be derived only for participants who were hospitalised for their index exacerbation and who have been subsequently discharged.

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day  $X - FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day  $X - FEV_1$  measured prior to dosing and post-bronchodilator on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Note, as per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the FEV<sub>1</sub> assessment will be assigned the hospital discharge assessment and the Day 14 assessment will be missing. Refer to Section 13.2.1.1 for further details.

In addition, if discharge takes place after Day 14, the Day 14 assessment will be missing for this analysis.

# 7.2.4.1. Statistical analyses

Change from hospital discharge in clinic visit trough  $FEV_1$  will be analysed using a repeated measures analysis as described in Section 7.1.2 if there are a sufficient number of participants to provide a meaningful analysis, otherwise the data will be summarised.

# 7.2.5. EXAcerbations of Chronic Pulmonary Disease Tool - Patient Reported Outcome (EXACT)

The EXACT is a 14-item daily diary designed to provide a measure of patient-reported symptoms of COPD exacerbation. An EXACT Total Score, ranging from 0 to 100, where

200879

higher scores indicate a more severe condition, will be derived for each day of diary collection according to the instructions in the EXACT User Manual (Version 8.0, Evidera, 2016).

The electronic EXACT diary does not allow a study patient to skip individual items, therefore no missing data are expected for individual items. However, if missing values occur for individual items, the Total Score that contains the item will be set to missing for that day. Moderate-to-severe COPD patients are expected to experience symptom(s) each day, and a score of zero on all 14 EXACT items is likely to represent a situation where in order to complete the diary quickly, the respondent did not accurately report their daily symptom(s), therefore if the EXACT Total Score is 0, it will be set to missing.

A 3-day Rolling Average EXACT Total Score will be calculated for each day, X, as:

(EXACT Total Score on Day X-1 + EXACT Total Score on Day X + EXACT Total Score on Day X+1) / (Number of days with non-missing values)

Note, for Day 1, the Rolling Average EXACT Total Score will be calculated as the average of EXACT Total Score on Days 1 (Randomisation) and 2 only, since no EXACT data is collected prior to randomisation. Similarly, the Rolling Average EXACT Total Score for the last study day will be calculated as the average of EXACT Total Score on the last day and on the day before the last day.

The Rolling Average EXACT Total Score will be calculated for each day as long as at least 1 EXACT total score in the sequence is present. Therefore, only in the case where EXACT total scores are missing for 3 consecutive days in a row (or 2 consecutive days in the case of the first and last day rolling average calculation), will the rolling average score be missing.

The Maximum Observed Value (MOV) is defined as the highest Rolling Average EXACT Total Score observed within the first 14 days of randomisation. Note: this definition differs from the definition in the EXACT User Manual of "the highest rolling average EXACT score observed in the context of an EXACT exacerbation within the first 14 days of the exacerbation", since the date of the index exacerbation is likely to be prior to randomisation.

# 7.2.5.1. Proportion of participants achieving EXACT-defined recovery from index exacerbation

EXACT-defined recovery from the index exacerbation is defined as a decrease in the Rolling Average EXACT Total Score  $\geq 9$  points from the Maximum Observed Value, sustained for  $\geq 7$  days, with the first of the 7 days defined as the recovery day.

The proportion of participants achieving EXACT-defined recovery from the index exacerbation by Days 14, 28, 56, and 84 will be calculated as:

(Number of participants who experience an EXACT-defined recovery on or before Day X) / (Total number of participants in the MITT population)

200879

Where Day X is 14, 28, 56, and 84.

## 7.2.5.2. Time to EXACT-defined recovery from index exacerbation

Time to EXACT-defined recovery from index exacerbation is defined as time from the date of randomisation until date of the first EXACT-defined recovery day during the 12-Week Treatment Period, where EXACT-defined recovery is described in Section 7.2.5.1. Participants who did not experience EXACT-defined recovery during the 12-Week Treatment Period will be censored at the date of their last dose of study treatment.

# 7.2.5.3. Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT is defined as the highest EXACT Total Score (not using the 3-day Rolling Average) during the period from date of onset of the subsequent HCRU-exacerbation until date of EXACT-defined recovery of subsequent exacerbation.

Note, in this case, the Maximum Observed Value and EXACT-defined recovery are derived using the date of onset of the subsequent HCRU-exacerbation.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will only be derived for participants who have had a subsequent exacerbation. If a participant has more than one subsequent exacerbation, severity will be calculated for each subsequent exacerbation.

## 7.2.5.4. Statistical analyses

The proportion of participants achieving EXACT-defined recovery from the index exacerbation will be analysed using a Bayesian logistic regression model. Separate models will be fitted for each time-point.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The results of the analysis will be presented in terms of odds ratios together with its associated 95% HPD credible interval. The probability that the true odds ratio is greater than 1, in addition to other values appropriately selected based on the data, will be presented.

Time to EXACT-defined recovery from index exacerbation will be analysed using the same techniques as described in Section 7.2.2.1.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will be summarised for each treatment group and reported by study period. The severity of subsequent HCRU-defined exacerbation(s) occurring whilst a participant is on treatment will be reported as during the 12-Week Treatment Period and the severity of subsequent HCRU-defined exacerbation(s) occurring after the last dose of study treatment will be reported as during the 12-Week Follow-up Period.

200879

#### 7.2.5.5. Subgroup analyses

A subgroup analysis of the proportion of participants achieving EXACT-defined recovery from the index exacerbation by Index Exacerbation Severity will be performed by including a treatment-by-severity term in the model.

#### 7.2.5.6. Sensitivity and supportive analyses

Sensitivity analyses exploring the impact of any missing data, and changes to the definition of EXACT-defined recovery may be conducted and may be performed post-SAC.

## 7.2.6. COPD Assessment Test (CAT)

The COPD Assessment Test (CAT) is a patient completed questionnaire developed to measure the health status of patients with COPD. The CAT consists of eight items, each on a six-point scale: 0 (no impact) to 5 (high impact). The CAT Score will be calculated for each study day of collection by summing the scores for all questions. The CAT Score ranges from 0 to 40, where higher scores indicate a more severe condition.

## 7.2.6.1. Proportion of responders using the CAT

The proportion of responders using the CAT will only be derived for participants with a baseline CAT Total Score  $\geq 2$ .

The Proportion of responders using the CAT is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq$ 2 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84 and the study day following EXACT-defined recovery from the index exacerbation.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

## **Exploratory – Follow-Up Period**

The Proportion of responders using the CAT at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq$ 2 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is Day 112 and Day 168 and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

#### 7.2.6.2. Change from baseline in CAT Total Score

Change from baseline in CAT Total Score is defined as:

200879

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is 28, 56, 84 and the study day following EXACT defined recovery from the index exacerbation.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

#### Exploratory - Follow-Up Period

The Change from baseline in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is Day 112 and Day 168.

The Change from end of treatment in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – CAT Total Score on Day 84

Where Day X is Day 112 and Day 168.

#### 7.2.6.3. Statistical analyses

The proportion of responders using CAT will be analysed using the same techniques as described in Section 7.2.5.4.

Change from baseline/end of treatment in CAT Total Score will be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant.

All post-baseline scheduled visits will be included in the analysis using Day.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

Adjusted posterior median change from baseline and corresponding 95% HPD credible intervals will be summarised for each treatment by time-point, together with estimated treatment differences (GSK – Placebo) and corresponding 95% HPD credible intervals. The posterior probability that the true treatment difference is less than 0, in addition to other values appropriately selected based on the data, will also be presented.

## 7.2.6.4. Subgroup analyses

A subgroup analysis of the proportion of responders using CAT and the change from baseline in CAT Total Score by Index exacerbation severity will be performed by

200879

including a treatment-by-severity term and a treatment-by-severity-by-Day term in the Bayesian logistic regression and Bayesian Repeated Measures models, respectively.

# 7.2.7. St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)

St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) is a 40-item questionnaire designed specifically to focus on COPD patients. SGRQ-C will be scored to be equivalent to the SGRQ Total Score, ranging from 0 to 100, where higher scores reflect worse health-related quality of life. SGRQ Total Scores will be calculated for each day of collection according to the instructions in SGRQ-C Manual (SGRQ, March 2016).

#### 7.2.7.1. Proportion of responders on the SGRQ Total Score

The proportion of responders on the SGRQ Total Score will only be derived for participants with a baseline SGRQ Total Score  $\geq$ 4.

Proportion of responders on the SGRQ Total Score is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84.

#### Exploratory - Follow-Up Period

The Proportion of responders on the SGRQ Total Score at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is Day 112 and Day 168 and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

#### 7.2.7.2. Change from baseline in SGRQ Total Score

Change from baseline in SGRQ Total Score is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is Day 28, 56, and 84.

## Exploratory - Follow-Up Period

The Change from baseline in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is Day 112 and Day 168.

200879

The Change from end of treatment in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – SGRQ Total Score on Day 84

Where Day X is Day 112 and Day 168.

## 7.2.7.3. Statistical analyses

Change from baseline/end of treatment in SGRQ Total Score and the proportion of responders on the SGRQ Total Score will be analysed using the same techniques as described in Section 7.2.6.3.

#### 7.2.7.4. Subgroup analyses

Subgroup analyses of change from baseline in SGRQ Total Score and the proportion of responders on the SGRQ Total Score by Index exacerbation severity will be conducted as described in Section 7.2.6.4.

#### 7.2.8. Rescue medication use

All participants will record rescue medication use in the eDiary. Rescue medication use will be recorded as the number of occasions of rescue medication use each day.

The Mean Number of Occasions of Rescue Medication Use Per Day is defined as:

(Sum of the number of occasions of rescue medication use each day within the time-period) / (Total number of days with non-missing values within the time-period)

The Percentage of Rescue-Free Days is defined as:

(Sum of the number of days where the number of occasions of rescue medication use is zero within the time-period) / (Total number of days with non-missing values within the time-period)\*100

Where the time-period is defined as follows:

Week 1 of the 12-Week Treatment Period: Day 1 to Day 7

Week 2 of the 12-Week Treatment Period: Day 8 to Day 14

Week 3 of the 12-Week Treatment Period: Day 15 to Day 21

Week 4 of the 12-Week Treatment Period: Day 22 to Day 28

Week 5 of the 12-Week Treatment Period: Day 29 to Day 35

Week 6 of the 12-Week Treatment Period: Day 36 to Day 42

Week 7 of the 12-Week Treatment Period: Day 43 to Day 49

200879

Week 8 of the 12-Week Treatment Period: Day 50 to Day 56

Week 9 of the 12-Week Treatment Period: Day 57 to Day 63

Week 10 of the 12-Week Treatment Period: Day 64 to Day 70

Week 11 of the 12-Week Treatment Period: Day 71 to Day 77

Week 12 of the 12-Week Treatment Period: Day 78 to Day of last dose

Over the 12-Week Treatment Period: Day 1 to Day of last dose.

#### Exploratory - Follow-Up Period

Rescue medication use up to Day 112 will also be summarised by including the timeperiods:

Week 13 (Follow-up Period): (Day of last dose + 1) to (Day of last dose + 1) + 6 days

Week 14 (Follow-up Period): (Day of last dose + 7) to (Day of last dose + 1) + 13 days

Week 15 (Follow-up Period): (Day of last dose + 14) to (Day of last dose + 1) + 20 days

Week 16 (Follow-up Period): (Day of last dose + 21) to (Day of last dose + 1) + 27 days

For a subject to be counted in the time periods for rescue medication use, they must have at least one eDiary entry recorded during that time period.

## 7.2.8.1. Rescue medication use via the clip-on Propeller Sensor for MDI

A subset of participants from countries where the Propeller Sensor for MDI is available will also record rescue medication use via the clip-on Propeller Sensor for MDI. A supportive summary of rescue medication use via the clip-on Propeller Sensor for MDI for these participants will be presented.

Rescue medication use via the clip-on Propeller Sensor for MDI is defined in the same way as rescue medication use via the eDiary, except that the number of actuations will be used instead of the number of occasions in accordance with the way the data is captured.

## 7.2.8.2. Statistical analyses

The Mean Number of (on-treatment) Occasions of Rescue Medication Use Per Day will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

The Percentage of (on-treatment) Rescue-Free Days will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

Rescue medication use via the clip-on Propeller Sensor for MDI will be summarised in the same way as rescue medication use via the eDiary.

200879

# 7.3. Exploratory Efficacy Analyses

## 7.3.1. Change from Day 84 in Clinic Visit trough FEV<sub>1</sub>

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day X – Day 84 post-bronchodilator  $FEV_1$ 

Where Day X is Day112, Day 140 and Day 168.

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day X – Day 84 pre-bronchodilator  $FEV_1$ 

Where Day X is Day 112, Day 140 and Day 168.

Participants who discontinue study treatment prior to Day 84 will be excluded from this analysis.

## 7.3.1.1. Statistical analysis

Change from Day 84 in Clinic Visit trough FEV<sub>1</sub> will be analysed using the same techniques as described for Change from baseline in CAT Total Score in Section 7.2.6.3.

A subgroup analysis of change from Day 84 in FEV<sub>1</sub> will be performed by including a treatment-by-severity-by-Day term in the Bayesian Repeated Measures model.

## 7.3.2. E-RS:COPD (Evaluating Respiratory Symptoms in COPD)

Change from baseline in E-RS: COPD and subscales will be summarised by treatment group. Exploratory analyses related to E-RS: COPD and subscales may be performed post SAC.

#### 7.3.3. Measures of HCRU related to exacerbations

Unscheduled Healthcare Utilisation will be summarised separately for exacerbation-related, COPD-related or non-COPD related; each summary will be presented by all patients (i.e. moderate and severe index exacerbation combined), and separately by index exacerbation severity.

The number of days of hospital admission for the index and subsequent exacerbations will also be summarised by treatment group.

200879

#### 7.3.3.1. Re-hospitalisation within 30 days of index exacerbation

Re-hospitalisation within 30 days of index exacerbation is defined as 30 days from the date of hospital discharge until the date of next hospital admission (+ 1 day, to account for study day derivation), for participants who were hospitalised for their index exacerbation.

Exacerbation-related, COPD-related and Non-COPD-related hospital admissions are collected in separate eCRFs. The date of hospital admission is not collected in the COPD-related eCRF, therefore the date of next hospital admission will be estimated using the earliest of:

- Date of hospital admission for exacerbation-related hospitalisations
- Date of contact for COPD-related hospitalisations, where the number of inpatient hospitalisation days >0
- Date of hospital admission for non-COPD-related hospitalisations.

The proportion of participants who were re-hospitalised within 30 days of the index exacerbation will be summarised by each treatment arm.

#### 7.3.3.2. Time from resolution of index exacerbation to next exacerbation

Time from resolution of index exacerbation to next exacerbation is defined as time from the date of (Investigator-defined) resolution of index exacerbation until the date of onset of the subsequent exacerbation.

A summary of time from resolution of index exacerbation to next exacerbation will be presented. Participants who did not have a subsequent exacerbation or for whom the index exacerbation was not resolved will be excluded from the summary.

Time from resolution of index exacerbation to next exacerbation will only be derived for the first subsequent exacerbation following the index exacerbation.

## 7.3.3.3. Subsequent exacerbation treatment type

A summary of the type of treatment for subsequent exacerbations (OCS, antibiotics, or both) may also be presented.

## 7.3.4. Compliance

Reported compliance for all participants is captured daily in the eDiary from the question "Did you take this morning's dose of study medication"?

Percentage compliance for each participant is calculated as:

(Sum of the number of days where the question was answered with 'Y') / (Number of days from first dose of study treatment to last dose of study treatment)  $\times$  100

Overall percentage compliance will be summarised by each treatment group.

200879

# 7.3.4.1. Number of actuations of double-blind study treatment measured by the clip-on Propeller Sensor

Percentage compliance via the clip-on Propeller Sensor for ELLIPTA in the subset of participants from countries where the Propeller Sensor for ELLIPTA is available is calculated as:

(Sum of the number of days with actuation > 0) / (Number of days from first dose of study treatment to last dose of study treatment) x 100

Overall percentage compliance will be summarised by each treatment group.

# 7.3.5. Inflammatory/infective markers in blood and sputum in relation to acute exacerbation of COPD

Results of the analysis of blood/spontaneous sputum samples of eosinophil counts and inflammatory/infective mediators/markers will be summarised by treatment group.

Further analyses of inflammatory/infective markers may be performed, for example split by CRP high, CRP low, Procalcitonin high, etc. categories.

### 7.3.6. Other spirometry measurements

Percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio will be summarised by treatment group.

## 7.3.7. Other symptoms suggestive of exacerbation

Responses to questions in the eDiary related to symptoms of sputum purulence (colour), fever, sore throat, wheezing and colds collected in the eDiary will be listed by treatment group.

# 7.3.8. Classification of exacerbating COPD participants and prediction of response to nemiralisib using machine learning techniques

Exploratory analysis of endpoints using machine learning techniques will be performed which will include classification of COPD participants, identification of parameters which describe a responder, and prediction of response to nemiralisib using baseline data. Details of these analyses will be described in a separate RAP and results may be reported separately to the CSR.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. The details of the planned displays will be provided in Appendix 11: List of Data Displays.

200879

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards.

## 8.1.1. Adverse Events of Special Interest

#### 8.1.1.1. Post-inhalation Cough Immediately Following Dosing

Post-inhalation cough immediately following dosing is an Adverse Event of Special Interest (AESI).

Post-inhalation cough immediately following dosing will be evaluated during study Visits 2-6 in the 12-Week Double-Blind Treatment Period. Investigators (or medically qualified designees) will monitor participants for potential study treatment tolerability issues, including post-inhalation cough, within 5 minutes immediately following dosing.

The percentage of patients experiencing post-inhalation cough following dosing, regardless of whether it was also reported as an AE, overall and by each visit will be summarised for each treatment group. The type of cough, time to onset and duration of cough, and severity will also be summarised.

In addition, any post-inhalation cough immediately following dosing reported as an adverse event during the clinic visit observation or during the course of the study will be summarised by treatment group.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and liver function tests will be based on GSK Core Data Standards.

## 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

## 8.4. Mortality

A summary of all-cause mortality by treatment will be presented.

## 9. PHARMACOKINETIC ANALYSES

## 9.1. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

200879

## 9.2. Drug Concentration Measures

Plasma nemiralisib concentrations of GSK2269557 will be listed and summarised by dose, day and time. Drug levels will be summarised by day (14, 28), dose and time intervals (trough, 0-<1h, 1-6h).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 13.4.3 Reporting Standards for Pharmacokinetic).

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

## 10. POPULATION PK ANALYSIS

A dataset for population PK analysis will be provided by Statistics and Programming based on the NONMEM data specifications in Section 13.8.2.

Conduct of the population PK analyses will be based on the current guidance which contains specific recommendations for working practices, processes and standards for population PK and PK/PD analysis conducted by Clinical Pharmacology Modelling and Simulation (CPMS) [Analysis & Reporting, 2017].

The sparse PK samples will be subjected to a validated population PK model for nemiralisib currently under development.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR. Analyses and reporting of the population PK model will be in accordance with the FDA and EMEA guidance on population PK, PK-PD analyses.

## 10.1. Derived Pharmacokinetic Parameters

The exposure parameters (e.g. AUC, C<sub>max</sub>) will be derived from the individual post-hoc estimates from the POP PK model. These will be summarized across dose treatments, subgroups (e.g., gender, race) or as a function of a continuous variable (e.g., age).

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

If statistical analyses suggest an effect of nemiralisib on primary and other key clinical endpoints, an integrated longitudinal population dose/exposure versus clinical response on analysis key parameters including  $FEV_1$  and exacerbation rate will be undertaken. Participant characteristics influencing the relationship will be evaluated.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

200879

## 12. REFERENCES

Bornkamp, B. (2014). Practical considerations for using functional uniform prior distributions for dose-response estimation in clinical trials. Biometrical Journal, 56(6), 947-962. doi: 10.1002/bimj.201300138.

Dette, H., Bretz, F., Pepelyshev, A. & Pinheiro, J., (2008). Optimal Designs for Dose-Finding Studies. Journal of the American Statistical Association, 103:483, 1255-1237. doi: 10.1198/016214508000000427.

Evidera. (2016). The Exacerbations of Chronic Pulmonary Disease Tool (EXACT®) Patient-Reported Outcome (PRO) USER MANUAL (Version 8.0).

SGRQ-C Manual (2016). St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Manual (Version 1.3).

Spiegelhalter, D.J., Abrams, K.R. & Myles, J.P., (2004). Bayesian Approaches to Clinical Trials and Health-Care Evaluation. John Wiley & Sons, Ltd.

200879

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 13.1.1. Exclusions from Per Protocol Population

Protocol deviations will be reviewed regularly throughout the course of the study, as described in Protocol Deviation Management Plan (PDMP). Deviations which will result in exclusion from the Per Protocol population will be assigned on a case-by-case basis prior to database freeze (DBF).

Decisions on whether or not the subject should be excluded from the PP population because the incorrect treatment was taken, due to the incorrect container being dispensed, will be identified after unblinding (i.e. post DBF). A PD of "incorrect treatment" will be added to the reporting dataset.

200879

## 13.2. Appendix 2: Assessment Windows

# 13.2.1. Definitions of Assessment Windows for Analyses

#### 13.2.1.1. Hospital discharge

As per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the FEV<sub>1</sub> assessment will be assigned the hospital discharge FEV<sub>1</sub> assessment and the Day 14 assessment will be missing.

For all other analyses and summaries that include participants who were hospitalised for their index exacerbation, an additional Analysis Timepoint of "HOSPTIAL DISCHARGE" will be derived. However, in the cases where discharge takes place between Day 11 and Day 17 (inclusive), participants will be summarised under DAY 14 and a footnote to say that participants who were discharged at Day 14 are summarised under DAY 14 will be included.

## 13.2.1.2. EXACT-Defined Recovery for CAT Trigger

Due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery from the index exacerbation is not derived according to the EXACT User Manual. Instead, it has been derived using a 3-day Rolling Average that is calculated as the mean EXACT score [Day X-2, Day X-1, Day X].

200879

# 13.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

#### 13.3.1. Study Periods

## 13.3.1.1. 12-Week Treatment Period

The 12-Week Treatment Period is assigned from Study Day 1 to Study Day 84.

#### 13.3.1.2. 12-Week Follow-Up Period

The 12-Week Follow-up Period is assigned from Study Day 85 to Study Day 168.

## 13.3.2. Study Phases

Exacerbation events during the 12-Week Treatment Period will be classified according to their occurrence from randomisation until treatment discontinuation/study withdrawal days, as detailed below.

| Study Phase | Occurring from randomisation until |
|---|---|
| On-Treatment during the 12-Week Treatment Period | Treatment Stop Day |
| On- or Off-Treatment during the 12-Week Treatment | Day 84 or Study Withdrawal Day if Treatment Stop |
| Period | Day is < Day 84 |

# 13.3.2.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before Randomisation Date |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 13.3.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date plus 10 days. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.
200879

#### 13.4. Appendix 4: Data Display Standards & Handling Conventions

#### 13.4.1. **Reporting Process**

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | : \arprod\gsk2269557\mid200879 |
| Analysis Datasets | |
| For all interim analyses, except for the End of Treatment Interim Analysis, datasets will be created according to Legacy GSK A&R dataset standards. | |

- For the End of Treatment Interim Analysis and the final reporting effort, datasets will be created according to current CDISC standards

#### **Generation of RTF Files**

RTF files will be generated for the final reporting effort.

#### 13.4.2. **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
  - Figures will be produced using PROC SGPLOT in SAS

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
- For lab parameters results that contain a character value of '<', or '>', e.g. '<X' or '>X', the parameter value will be imputed with X.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

200879

| Unscheduled Visits | |
|---|---|
| Unscheduled visits will be included in summary tables of the worst-case results by potential clinical importance criteria only. | |
| All unscheduled vi | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

# 13.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 13.8.2 Population Pharmacokinetic (PopPK) Dataset Specification. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in the CPMS RAP. |

200879

### 13.5. Appendix 5: Derived and Transformed Data

#### 13.5.1. General

### Multiple Measurements at One Analysis Time Point

 Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Randomisation Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### Time from date of randomisation and time from date of last dose of study treatment

- For endpoints that use the time from the date of randomisation to a reference date, time will be calculated as
  - (Ref Date Randomisation Date) + 1
- For endpoints that use the time from the date of last dose of study treatment to a reference date, time will be calculated as
  - (Ref Date (Last Dose Date + 1)) +1

### 13.5.2. Study Population

### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- The cumulative dose will be based on the formula:

**Cumulative Dose = Sum of (Number of Days x Total Daily Dose)** 

### 13.5.3. Safety

#### **Adverse Events**

### **AE'S of Special Interest**

 Post-inhalation cough is an AE of special interest. The lower level term (LLT) to be included is "coughing after drug inhalation"

200879

# 13.6. Appendix 6: Reporting Standards for Missing Data

## 13.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) is defined as completing all phases of the study including the last scheduled study visit |
| | A participant is considered to have completed the Treatment Period, if he/she has completed the last on-treatment study visit (Visit 6) |
| | Withdrawn subjects were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will not be summarised (and will be listed only). |

# 13.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 13.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> </ul> |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |
| Age | <ul> <li>The eCRF collects year of birth only. Day and Month will be imputed by Data Management using a PP for the day and PPD for the month</li> <li>Age will then be derived referenced to the Screening Date</li> <li>A footnote to say that age has been imputed will be included in any outputs containing</li> </ul> |
| | age. |

200879

# 13.7. Appendix 7: Values of Potential Clinical Importance

# 13.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male 18-64 years | 7.1 | 19.9 |
| Haemoglobin | G/DL | Male 65+ years | 7.1 | 19.9 |
| Tidemoglobin | | Female 18-64 years | 7.1 | 19.9 |
| | | Female 65+ years | 7.1 | 19.9 |
| Lymphocytes | GI/L | | 0.85 | 4.1 |
| Total Absolute Neutrophil Count | GI/L | | 1.5 | 8 |
| Platelet Count | GI/L | | 31 | 1499 |
| White Blood Cell count | 01/1 | 18-64 years | 1.1 | 10.8 |
| Write blood Cell Court | GI/L | 65+ years | 1.1 | 10.8 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 32 | 50 |
| Calcium | mmol/L | | 1.5 | 3.24 |
| | | Male 40-49 years | 69 | 160 |
| | | Male 50-59 years | 67.2 | 160 |
| | | Male 60-69 years | 67.2 | 160 |
| Creatinine | | Male 70+ years | 59.2 | 160 |
| Creatifile | | Female 40-49 years | 52.2 | 160 |
| | | Female 50-59 years | 53 | 160 |
| | | Female 60-69 years | 53 | 160 |
| | | Female 70+ years | 55.7 | 160 |
| | mmol/L | 13-49 years | 2.2 | 27.8 |
| Glucose | IIIIIIOI/L | 50+ years | 2.2 | 27.8 |
| Potassium | tassium mmol/L | | 2.8 | 6.5 |
| Sodium | mmol/L | | 120 | 160 |
| | mmol/l | 13-64 years | 2.5 | 15 |
| Urea/BUN | mmol/L | 65+ years | 2.5 | 15 |

200879

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 2x ULN |
| T. Bilirubin + ALT | µmol/L<br>U/L | High | 2xULN T.Bilirubin + ≥ 3x ULN ALT |
| Direct Bilirubin | μmol/L | | 0 – 6 |

## 13.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 530 |
| Absolute PR Interval | msec | < 110 | > 240 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 13.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 90 | > 140 |
| Diastolic Blood Pressure | mmHg | < 60 | > 90 |
| Heart Rate | bpm | < 40 | > 110 |

200879

### 13.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

### 13.8.1. Population Pharmacokinetic (PopPK) Methodology

All analysis will be performed in the validated Modelling and Analysis Platform (MAP). MAP consists of a Linux desktop containing various modelling applications, including NONMEM, PsN, Pirana, R and RStudio. All software versions used will be documented.

The population PK analysis will be performed in the following sequence of steps:

- 1. Exploratory data analysis/data check out.
- 2. Base structural model development.
- 3. Covariate analysis.
- 4. Model refinement.
- 5. Model evaluation.
- 6. Model application using simulation

The above analysis and reporting steps follow EMEA (http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC500003067.pdf) and FDA population PK guidances (https://www.fda.gov/downloads/drugs/guidances/UCM072137.pdf)

Key components of these regulatory guidelines on population PK are also included in the Global CPMS guidance for pop pk RAP (https://connect.gsk.com/sites/cpms/TandD/Guidances).

#### 13.8.2. Population Pharmacokinetic (PopPK) Dataset Specification

Statistics & Programming, in discussion with CPMS, will provide a NONMEM dataset.

Column headings in NONMEM-ready datasets and specifications should be consistent to minimise the programming process, and facilitate a smooth transfer of projects between users as needed. IDSL standards will be followed where possible.

A list of most common standardised variable names for NONMEM datasets can be found in Table below.

200879

## List of Variable Names for NONMEM-Ready Datasets for PopPK Analysis

| Variable | Label (Variable description) |
|---|---|
| С | NONMEM line exclusion identifier |
| ID | NONMEM subject identifier |
| STUD | Study ID |
| SUBJID | Subject identifier for study |
| SITEID | Unique identifier for a study site |
| AMT | NONMEM Amount of drug administered then EVID =1- dose event record |
| UAMT | Unit of AMT (mg) |
| ADDL | NONMEM Additional dose |
| CONC | Drug Concentration |
| UCONC | Unit of CONC (ng/mL) |
| LNCONC | Natural log of CONC column |
| ANALYTE | Drug label e.g 557 |
| LLQ | Lower Limit of quantification |
| LNLLQ | Natural log of LLQ column |
| DAY | Study day number of record or of dosing |
| TIME | Plasma sample time after last dose |
| UTIME | Unit of TIME (h) |
| DOSE | Dose amount |
| EVID | NONMEM Event ID If row has dose then EVID=1 else EVID=0 |
| | If EVID=1 then this is a dose event record |
| п | If EVID = 0 then this is an observation record |
| II<br>SS | NONMEM Inter-dose interval II=24 – dose every day |
| MDV | Steady state item SS= 1 refers to steady state |
| AGE | NONMEM Missing data value then MDV=1 else MDV=0 |
| _ | Subject Age (yrs) |
| SEX | Subject gender 0 = Male 1 = Female |
| SEXTEXT | Subject gender text Male or Female |
| BMI | Baseline Body Mass Index |
| WT | Baseline Subject weight |
| CONMED1 | Identifier for inhibitor CYP3A4 1 =Yes, 0 = No |
| CONMED1TXT | Inhibitor Name |
| CONMED2 | Identifier for inducer CYP3A4 1 =Yes, 0 = No |
| CONMED2TXT | Inducer Name |
| - | 00101 (010) (010) (110) |

If observation record e.g CONC has "NA" or "NS" then assign CONC cell as "."

If observation record e.g CONC has "NQ" or "BQL" then assign CONC cell as "." and MDV = 1 -this means value can be estimated by model

Missing covariate data should be imputed as "-99.

200879

### 13.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

### 13.9.1. Pharmacokinetic/Pharmacodynamic Methodology

PK-PD analysis of Nemiralisib will be guided by the results of the formal statistical analyses on the key clinical endpoints. The aims of the PK-PD analyses will contribute towards the dose selection in future studies using an integrated longitudinal analysis framework.

The objective is to explore an integrated modelling framework to characterise the longitudinal FEV1 response versus dose (average systemic exposure) during on- & off-treatment phases

$$FEV1_i(t_{ij}) = FEV1_{i,base} \cdot (1 + f(t_{ij}, dose_i, x_i) + \varepsilon_{ij} \text{ with } \varepsilon_{ij} \sim N(0, \sigma 2)$$

A longitudinal nonlinear mixed-effects model will be used to describe the FEV1 response over time measured for each patient (i) at each visit (tij) with  $\varepsilon$  denoting the normal distributed residual variability with mean 0 and variance  $\sigma$ 2. The function f() describes the relative change from observed FEV1 at baseline (FEV1,<sub>base</sub>) and any influence of patient characteristics on FEV1 response will be assessed.

Joint relationship between time to first exacerbation and FEV1 change as function of dose/exposure and patient covariates will be assessed.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

200879

# 13.10. Appendix 10: Abbreviations & Trade Marks

## 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SGRQ | St. George's Respiratory Questionnaire |
| SGRQ-C | St. George's Respiratory Questionnaire for COPD Patients |
| SOP | Standard Operation Procedure |

200879

| IFL | TFL | Tables, Figures & Listings |
|-----|-----|----------------------------|
|-----|-----|----------------------------|

## 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| COPD Assessment Test (CAT) |
| ELLIPTA |
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| E-RS: COPD |
| EXACT-PRO |
| NONMEM |
| Propeller Sensor |
| SAS |
| SGRQ |

200879

## 13.11. Appendix 11: List of Data Displays

## 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays for SAC:

| Section | Tables | Figures |
|------------------|--------------|----------------|
| Study Population | 1.1 to 1.28 | Not applicable |
| Efficacy | 2.1 to 2.100 | 2.1 to 2.20 |
| Safety | 3.1 to 3.31 | 3.1 to 3.3 |
| Pharmacokinetic | 4.1 to 4.2 | Not applicable |
| Section | Listings | |
| ICH Listings | 1 to 27 | |
| Other Listings | 28 to 30 | |

## 13.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

### 13.11.3. Deliverables

| Delivery | Description |
|---|---|
| IA | Interim Analysis (except the End of treatment Phase Interim Analysis) |
| EOT | End of Treatment Phase Interim Analysis |
| SAC | Statistical Analysis Complete |

200879

## 13.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | MITT | ES8 | Summary of Subject Status and Reason for Study Withdrawal | | EOT, SAC |
| 1.2. | MITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | EOT, SAC |
| 1.3. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| 1.4. | APE | NS1 | Summary of Number of Participants by Country and Site ID | | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | MITT | DV1 | Summary of Important Protocol Deviations | | SAC |
| 1.6. | MITT | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tion Analysed | | | | |
| 1.7. | MITT | SP1 | Summary of Study Populations | | SAC |
| 1.8. | MITT | SP2 | Summary of Exclusions from the Per Protocol/Safety Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | 1 |
| 1.9. | MITT | DM1 | Summary of Demographic Characteristics | Use the following ranges for the Age<br>Group row: ≤64; 65-74; ≥75 | EOT, SAC |
| 1.10. | APE | DM11 | Summary of Age Ranges | | SAC |
| 1.11. | MITT | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.12. | MITT | MH4 | Summary of Past Medical Conditions | | EOT, SAC |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.13. | MITT | MH4 | Summary of Current Medical Conditions | | EOT, SAC |
| 1.14. | MITT | FH1 | Summary of Family History of Cardiovascular Risk Factors | | EOT, SAC |
| 1.15. | MITT | SU1 | Summary of Smoking History at Screening | | EOT, SAC |
| 1.16. | MITT | SU1 | Summary of Smoking Status Over the 12-Week Treatment Period | | EOT, SAC |
| 1.17. | MITT | SU1 | Summary of Smoking Status Over the 12-Week Follow-Up Period | | SAC |
| 1.18. | MITT | Example 7 | Summary of COPD Duration at Screening | | EOT, SAC |
| 1.19. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening | Use categories 0;1;2;3;≥3. Summarise moderate/severe, moderate; severe Include 7-Day History of COPD Exacerbations | EOT, SAC |
| 1.20. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening by Country | | EOT, SAC |
| Conco | mitant Medicati | ons | | | |
| 1.21. | MITT | Example 14 | Summary of Baseline COPD Maintenance Therapy | | EOT, SAC |
| 1.22. | MITT | Example 15 | Summary of On-Treatment COPD Maintenance (Step-up) Therapy | | EOT, SAC |
| 1.23. | MITT | CM1 | Summary of Concomitant Medications During 12-Week<br>Treatment Period | | EOT, SAC |
| 1.24. | MITT | Example 16 | Summary of OCS Use | | EOT, SAC |
| 1.25. | MITT | CM1 | Summary of Concomitant Medications During 12-Week Follow-<br>Up Period | | SAC |

200879

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.26. | MITT | EX1 | Summary of Exposure to Study Treatment | | EOT, SAC |
| 1.27. | MITT | Example 2 | Summary of Treatment Compliance | | EOT, SAC |
| 1.28. | MITT | Example 2 | Summary of Actuations of Study Treatment Measured by the Clip-on Propeller Sensor | | SAC |

## 13.11.5. Efficacy Tables

## 13.11.5.1. Efficacy tables for Interim Analysis 1

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV <sub>1</sub> | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | IA1 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | IA1 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator (Dose Response Model) | | IA1 |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator (Dose Response Model) | | IA1 |
| 2.7. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.8. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.9. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Post-bronchodilator (Repeated Measures Model) | | IA1 |
| 2.10. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Pre-bronchodilator (Repeated Measures Model) | | IA1 |
| 2.11. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| 2.12. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Pre-bronchodilator by Index Exacerbation Severity<br>(Repeated Measures Model) | | IA1 |
| Rate of | Exacerbations | | | | |
| 2.13. | MITT | Example 5 | Summary of On-treatment Exacerbations | | IA1 |
| 2.14. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Severity | | IA1 |
| EXAcer | bations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.15. | MITT | Example 9 | Summary of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | Exclude statistical analysis information (summary only) | IA1 |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | MITT | Example 9 | Summary of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | Exclude statistical analysis information (summary only) | IA1 |
| Other S | pirometry Mea | sures | | | |
| 2.17. | MITT | Example 3 | Summary of Spirometry Measurements | | IA1 |
| 2.18. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA1 |

200879

## 13.11.5.2. Efficacy tables for Interim Analysis 2

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | IA2 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator.<br>Include additional row for hospital<br>discharge visit for Severe group | IA2 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator (Dose Response Model) | | IA2 |
| 2.9. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.10. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.12. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.13. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.14. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.15. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | IA2 |
| 2.16. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | IA2 |
| 2.17. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Post-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.18. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Pre-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.19. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.20. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) Measured Pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| 2.21. | MITT | Example 32 | Summary of Efficiency Ratio for Possible Adaptions to Randomization Ratio | | IA2 |
| Rate of | Exacerbations | 1 | | | |
| 2.22. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations | | IA2 |
| 2.23. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent<br>Exacerbations by Index Exacerbation Severity | | IA2 |
| 2.24. | MITT | Example 6 | Statistical Analysis of On-treatment (Moderate/Severe)<br>Subsequent Exacerbations | | IA2 |
| 2.25. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | IA2 |
| EXAce | rbations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | • |
| 2.26. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | IA2 |
| 2.27. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | IA2 |
| COPD | Assessment Te | st (CAT) | | | |
| 2.28. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score | | IA2 |
| 2.29. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the CAT Total Score by Visit | | IA2 |
| 2.30. | MITT | Example 11 | Statistical Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) | | IA2 |

200879

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) | | |
| 2.31. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score | | IA2 |
| 2.32. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the SGRQ Total Score by Visit | | IA2 |
| 2.33. | MITT | Example 11 | Statistical Analysis of Change from Baseline in SGRQ Total Score (Repeated Measures Model) | | IA2 |
| Rescue | Medication Us | e | | | |
| 2.34. | MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | IA2 |
| 2.35. | MITT | RM1 | Summary of Percentage of Rescue-Free Days | | IA2 |
| Other S | Other Spirometry Measures | | | | |
| 2.36. | MITT | Example 3 | Summary of Spirometry Measurements | | IA2 |
| 2.37. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA2 |

## 13.11.5.3. Efficacy tables for End of Treatment Interim Analysis and SAC

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | EOT, SAC |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.9. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | EOT, SAC |
| 2.10. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | EOT, SAC |
| 2.11. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | EOT, SAC |
| 2.12. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | EOT, SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | EOT, SAC |
| 2.14. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | EOT, SAC |
| 2.15. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate (Dose Response Model) | | EOT, SAC |
| 2.16. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe (Dose Response Model) | | EOT, SAC |
| 2.17. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.18. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L)<br>Measured Post-bronchodilator by Index Exacerbation Severity<br>(Repeated Measures Model) | | EOT, SAC |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV <sub>1</sub> | | |
| 2.19. | MITT | Example 3 | Summary of Change from Hospital Discharge in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.20. | MITT | Example 11 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.21. | MITT | Example 11 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) Measured Pre-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| Change | from Day 84 in | n Clinic Visit troug | jh FEV₁ | | |
| 2.22. | MITT | Example 3 | Summary of Change from Day 84 in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Post-bronchodilator (Repeated Measures Model) | | SAC |
| 2.24. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Pre-bronchodilator (Repeated Measures Model) | | SAC |
| 2.25. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | SAC |
| 2.26. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) Measured Pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | SAC |
| Rate of | Exacerbations | | | | |
| 2.27. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.28. | MITT | Example 5 | Summary of On-treatment (Mild/Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.29. | MITT | Example 5 | Summary of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.30. | MITT | Example 6 | Statistical Analysis of On-treatment (Moderate/Severe)<br>Subsequent Exacerbations | | EOT, SAC |
| 2.31. | MITT | Example 6 | Statistical Analysis of On-treatment (Mild/Moderate/Severe)<br>Subsequent Exacerbations | | EOT, SAC |
| 2.32. | MITT | Example 6 | Subgroup Analysis of On-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.33. | MITT | Example 5 | Summary of On-treatment Subsequent Exacerbations by Index Exacerbation Type | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | MITT | Example 5 | Summary of On-treatment Subsequent Exacerbations by Number of Exacerbations in Previous 12 Months | | EOT, SAC |
| 2.35. | MITT | Example 5 | Summary of On-or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | EOT, SAC |
| 2.36. | MITT | Example 5 | Summary of On-or Off-treatment (Mild/Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | EOT, SAC |
| 2.37. | MITT | Example 5 | Summary of On-or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |
| 2.38. | MITT | Example 6 | Statistical Analysis of On- or Off-treatment (Moderate/Severe)<br>Subsequent Exacerbations During the 12-Week Treatment<br>Period | | EOT, SAC |
| 2.39. | MITT | Example 6 | Statistical Analysis of On- or Off-treatment (Mild/Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period | | EOT, SAC |
| 2.40. | MITT | Example 6 | Subgroup Analysis of On- or Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 12-Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |
| 2.41. | MITT | Example 5 | Summary of Off-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |
| 2.42. | MITT | Example 5 | Summary of Off-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.43. | MITT | Example 6 | Statistical Analysis of Off-treatment (Moderate/Severe) Subsequent Exacerbations | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.44. | MITT | Example 6 | Subgroup Analysis of Off-treatment (Moderate/Severe) Subsequent Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.45. | MITT | Example 5 | Summary of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period | | EOT, SAC |
| 2.46. | MITT | Example 5 | Summary of On- and Off-treatment (Moderate/Severe) Subsequent Exacerbations During the 24-Week Study Period by Index Exacerbation Severity | | EOT, SAC |
| 2.47. | MITT | Example 6 | Statistical Analysis of On- and Off-treatment (Moderate/Severe)<br>Subsequent Exacerbations During the 24-Week Study Period | | EOT, SAC |
| 2.48. | MITT | Example 6 | Subgroup Analysis of On- and Off-treatment (Moderate/Severe)<br>Subsequent Exacerbations During the 24-Week Study Period by<br>Index Exacerbation Severity | | EOT, SAC |
| Time to | Next Exacerba | ation | | | |
| 2.49. | MITT | Example 8 | Statistical Analysis of Time to next On-treatment Exacerbation | | EOT, SAC |
| 2.50. | MITT | Example 8 | Subgroup Analysis of Time to next On-treatment Exacerbation by Index Exacerbation Severity | | EOT, SAC |
| 2.51. | MITT | Example 8 | Statistical Analysis of Time to next On- or Off-treatment Exacerbation During the 12-Week Treatment Period | | EOT, SAC |
| 2.52. | MITT | Example 8 | Statistical Analysis of Time to next On- or Off-treatment Exacerbation During the 12-Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |
| 2.53. | MITT | Example 8 | Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment | | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.54. | MITT | Example 8 | Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment by Index Exacerbation Severity | | SAC |
| EXAce | bations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.55. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | EOT, SAC |
| 2.56. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | EOT, SAC |
| 2.57. | MITT | Example 8 | Summary and Statistical Analysis of Time to EXACT-defined Recovery | | EOT, SAC |
| 2.58. | MITT | Example 10 | Summary of Severity of Subsequent HCRU-defined<br>Exacerbation During 12-Week Treatment Period | Also split by moderate and severe | EOT, SAC |
| 2.59. | MITT | Example 10 | Summary of Severity of Subsequent HCRU-Defined<br>Exacerbation During 12-Week Follow-up Period | Also split by moderate and severe | EOT, SAC |
| COPD | Assessment Te | st (CAT) | | | |
| 2.60. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score | | EOT, SAC |
| 2.61. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.62. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the CAT Total Score by Visit | | EOT, SAC |
| 2.63. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders Using the CAT Total Score by Visit by Index Exacerbation Severity | | EOT, SAC |
| 2.64. | MITT | Example 11 | Statistical Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.65. | MITT | Example 11 | Subgroup Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.66. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score | | EOT, SAC |
| 2.67. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.68. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.69. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) | | |
| 2.70. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score | | EOT, SAC |
| 2.71. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.72. | MITT | Example 9 | Statistical Analysis of Proportion of Responders on the SGRQ<br>Total Score by Visit | | EOT, SAC |
| 2.73. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders on the SGRQ<br>Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.74. | MITT | Example 11 | Statistical Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.75. | MITT | Example 11 | Subgroup Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |
| 2.76. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score | | EOT, SAC |
| 2.77. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score by Index Exacerbation Severity | | EOT, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.78. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in SGRQ Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.79. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in SGRQ<br>Total Score (Repeated Measures Model) by Index Exacerbation<br>Severity | | EOT, SAC |
| E-RS: C | COPD | | | | |
| 2.80. | MITT | Example 3 | Summary of Change from Baseline in E-RS: COPD and Subscales | | SAC |
| Rescue | Medication Us | se | | | |
| 2.81. | MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | EOT, SAC |
| 2.82. | MITT | RM1 | Summary of Percentage of Rescue-Free Days | | EOT, SAC |
| 2.83. | MITT | RM1 | Summary of Mean Number of Actuations of Rescue Medication Use Per Day Via the Clip-on Propeller Sensor for MDI | | EOT, SAC |
| 2.84. | MITT | RM1 | Summary of Percentage of Rescue-Free Days Via the Clip-on Propeller Sensor for MDI | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Compli | ance | | | | |
| 2.85. | MITT | IP1 | Summary of Overall IP Compliance | | EOT, SAC |
| 2.86. | MITT | IP1 | Summary of Overall IP Compliance Via the Clip-on Propeller Sensor for ELLIPTA | | EOT, SAC |
| Health | care Resource I | Utilisation | | | |
| 2.87. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilisation | | EOT, SA |
| 2.88. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilization by Index Exacerbation Severity | | EOT, SA |
| 2.89. | MITT | Example 21 | Summary of Exacerbation Related Hospitalizations | | EOT, SAC |
| 2.90. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation | | EOT, SAC |
| 2.91. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | EOT, SAC |
| 2.92. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation | | EOT, SAC |
| 2.93. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | EOT, SAC |
| 2.94. | MITT | Example 22 | Summary of Re-hospitalization Within 30 days of Index Exacerbation | | EOT, SAC |
| 2.95. | MITT | Example 24 | Summary of Time from Resolution of Index Exacerbation to Next Exacerbation | | EOT, SAC |
| 2.96. | MITT | Example 23 | Summary of Subsequent Exacerbation Treatment | | EOT, SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Other S | Other Spirometry Measures | | | | |
| 2.97. | MITT | Example 3 | Summary of Spirometry Measurements | | EOT, SAC |
| 2.98. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | EOT, SAC |
| Inflamn | Inflammatory/infective Markers in Blood and Sputum | | | | |
| 2.99. | MITT | Example 3 | Summary of Inflammatory Markers in Blood | | SAC |
| 2.100. | MITT | Example 3 | Summary of Inflammatory Markers in Sputum | | SAC |

200879

## 13.11.6. Efficacy Figures

## 13.11.6.1. Efficacy Figures for Interim Analysis 1

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | IA1 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | IA1 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 measured post-bronchodilator | | IA1 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |

200879

## 13.11.6.2. Efficacy Figures for Interim Analysis 2

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | IA2 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | IA2 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator | | IA2 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator | | IA2 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.13. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator | | IA2 |
| 2.14. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.15. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| Time to | Time to Next Exacerbation | | | | |
| 2.16. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Moderate/Severe) Exacerbation | | IA2 |
| 2.17. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Mild/Moderate/Severe) Exacerbation | | IA2 |

200879

## 13.11.6.3. Efficacy Figures for End of Treatment Interim Analysis and SAC

| Efficacy | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator | | EOT, SAC | |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator | | EOT, SAC | |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator | | EOT, SAC | |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator | | EOT, SAC | |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC | |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC | |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC | |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC | |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC | |
| Efficac | Efficacy: Figures | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC | | | |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC | | | |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC | | | |
| 2.13. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator | | EOT, SAC | | | |
| 2.14. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC | | | |
| 2.15. | MITT | Example 31 | Plot of Repeated Measures Model of Change from Baseline in FEV <sub>1</sub> Measured Post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC | | | |
| Time to | Next Exacerba | ation | | | | | | |
| 2.16. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Moderate/Severe) Exacerbation | | EOT, SAC | | | |
| 2.17. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-treatment (Mild/Moderate/Severe) Exacerbation | | EOT, SAC | | | |
| 2.18. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-or Off-treatment (Moderate/Severe) Exacerbation During the 12-Week Treatment Period | | EOT, SAC | | | |

200879

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next On-or Off-treatment (Mild/Moderate/Severe) Exacerbation During the 12-Week Treatment Period | | EOT, SAC |
| 2.20. | MITT | Example 30 | Kaplan-Meier Plot of Time to Next (Moderate/Severe) Exacerbation Following Cessation of Study Treatment | | SAC |

# 13.11.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term | | EOT, SAC |
| 3.2. | Safety | AE1 | Summary of Post-Treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Treatment Emergent Adverse Events by Overall Frequency | | EOT, SAC |
| 3.4. | Safety | AE1 | Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term | | EOT, SAC |
| 3.5. | Safety | AE15 | Summary of Common (>=5%) Non-serious Treatment Emergent<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | AE1 | Summary of Treatment Emergent Adverse Events for<br>Participants with Absolute Neutrophil Count Below Lower Value of PCI | | SAC |
| Serious | and Other Sig | nificant Adverse I | Events | | |
| 3.7. | Safety | AE16 | Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | | EOT, SAC |
| 3.8. | Safety | AE16 | Summary of Fatal Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | Only with subcategory: Number of Fatal SAEs | EOT, SAC |
| 3.9. | Safety | AE1 | Summary of Serious Treatment Emergent Drug-related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.10. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | EOT, SAC |
| 3.11. | Safety | AE1 | Summary of Post-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.12. | Safety | AE1 | Summary of Treatment Emergent Adverse Events of Special Interest by Lower Level Term | | EOT, SAC |
| 3.13. | Safety | Example 17 | Summary of Post-Inhalation Cough by Visit | | EOT, SAC |
| 3.14. | Safety | Example 28 | Summary of Post-Inhalation Cough by Visit and Cough Type | | EOT, SAC |
| 3.15. | Safety | Example 33 | Summary of Post-Inhalation (PI) Cough at Any Visit | | EOT, SAC |
| Labora | tory: Chemistry | 1 | | | |
| 3.16. | Safety | LB1 | Summary of Chemistry Data | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.17. | Safety | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.18. | Safety | LB1 | Summary of Hematology Data | | SAC |
| 3.19. | Safety | LB1 | Summary of Change from Baseline in Hematology | Only for WBC, lymphocytes, neutrophils | SAC |
| 3.20. | Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.21. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC |
| 3.22. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC |
| ECG | • | | | | |
| 3.23. | Safety | EG1 | Summary of ECG Findings | | EOT, SAC |
| 3.24. | Safety | EG2 | Summary of ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | EOT, SAC |
| 3.25. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | SAC |
| 3.26. | Safety | Example 27 | Summary of QTcF Categories | | SAC |
| 3.27. | Safety | Example 27 | Summary of QTcB Categories | | SAC |
| 3.28. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.29. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.30. | Safety | Example 25 | Summary of ECG Abnormalities for Participants with Any Abnormal ECG Interpretation | | EOT, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | gns | | | | |
| 3.31. | Safety | VS1 | Summary of Vital Signs | | SAC |
| 3.32. | Safety | VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | | EOT, SAC |

200879

## 13.11.8. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory | | | | |
| 3.1. | Safety | LB7 | LFT Shift from Baseline to Maximum | | EOT, SAC |
| 3.2. | Safety | Example 13 | Median (range) Absolute Neutrophil Count by Time and Treatment | | SAC |
| ECG | ECG | | | | |
| 3.3. | Safety | EG8 | Distribution of QTcF Change by Time and Treatment | | SAC |

## 13.11.9. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic Cond | centration-Time D | ata | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK2269557 Pharmacokinetic Concentration-Time Data | | SAC |
| 4.2. | PK | PK05 | Summary of Log-Transformed Plasma GSK2269557<br>Pharmacokinetic Concentration-Time Data | | SAC |

200879

## 13.11.10. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | MITT | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | MITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 4. | MITT | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | | SAC |
| 5. | MITT | TA1 | Listing of Planned and Actual Treatments | | SAC |
| Protoc | ol Deviations | | | | |
| 6. | MITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 7. | MITT | IE3 | Listing of Participants with Inclusion/Exclusion Criteria<br>Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 8. | MITT | SP3 | Listing of Participants Excluded from Per Protocol Population | For participants excluded from MITT population (i.e. participants in the MITT but not in PP) | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | MITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 10. | MITT | DM9 | Listing of Race | | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | MITT | CP_CM3 | Listing of Concomitant Medications | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ure and Treatme | ent Compliance | | | • |
| 12. | Safety | EX3 | Listing of Exposure Data | | SAC |
| Advers | e Events | | | | |
| 13. | Safety | AE8 | Listing of All Adverse Events | | SAC |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | • |
| 16. | Safety | AE8 | Listing of Fatal Serious Adverse Events | | SAC |
| 17. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 18. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping<br>Events | | SAC |
| All Lab | oratory | | | | • |
| 22. | Safety | LB5 | Listing of All Chemistry Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 23. | Safety | LB14 | Listing of Chemistry Data with Character Results | | SAC |

200879

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Safety | LB5 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 25. | Safety | LB14 | Listing of all Hematology Data with Character Results | | SAC |
| ECG | | | | | |
| 26. | Safety | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | | SAC |
| 27. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal Finding | | SAC |

## 13.11.11. Non-ICH Listings

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 28. | MITT | Example 29 | Listing of Subjects who Received Incorrect Medication | | SAC |
| 29. | PK | PK07 | Listing of Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 30. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC |

200879

### 13.12. Appendix 12: Example Mock Shells for Data Displays

### 13.12.1. Example shell 1

Example Shell X
Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of COPD Exacerbation History at Screening

| | Treatment A (N=100) | Treatment B (N=100) | Total (N=200) |
|---|---|---|---|
| Moderate COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Severe COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Total number of moderate/severe COPD exacerbations | | | |
| n | 911 | 899 | 1810 |
| 0 | 313 (34%) | 317 (35%) | 630 (35%) |
| 1 | 252 (28%) | 253 (28%) | 505 (28%) |
| >=2 | 346 (38%) | 329 (37%) | 675 (37%) |

Note: Number of COPD exacerbations reported in the 12 months prior to the Screening Visit.

200879

## 13.12.2. Example Shell 2

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific
Table X

Summary of Treatment Compliance

| | Treatment $P$ (N=100) | A Treatment B (N=100) | Total (N=200) |
|---|---|---|---|
| Overall compliance (%) | | | |
| n | XX | XX | XX |
| Mean | xx | XX | XX |
| SD | xx | XX | XX |
| Median | xx | XX | XX |
| Min. | xx | XX | XX |
| Max. | xx | XX | XX |
| Compliance interval | | | |
| < 80% | xx (x%) | xx (x%) | xx (x%) |
| 80% - < 100% | xx (x%) | xx (x%) | xx (x%) |
| 100% - < 120% | xx (x%) | xx (x%) | xx (x%) |
| >=120% | xx (x%) | xx (x%) | xx (x%) |

200879

## 13.12.3. Example shell 3

Example Shell X Protocol: ABC123456


Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of Change from Baseline in FEV1 (L)  $\begin{tabular}{ll} Measured post-bronchodilator \end{tabular}$ 

| Visit | N | Treatment Arm | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| Day 1 | 200 | Placebo | 200 | 0.111 | 0.1111 | 0.100 | -0.11 | 1.11 |
| _ | 200 | GSK2269557 12.5 mc | g 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | 200 | GSK2269557 50 mc | g 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | 200 | GSK2269557 100 mc | g 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | 200 | GSK2269557 250 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 500 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 750 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| Day 14 | 200 | Placebo | 200 | 0.111 | 0.1111 | 0.100 | -0.11 | 1.11 |
| | 200 | GSK2269557 12.5 mc | g 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | 200 | GSK2269557 50 mc | g 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | 200 | GSK2269557 250 mc | g 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | 200 | GSK2269557 500 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 750 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |

200879

### 13.12.4. Example Shell 4

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Statistical Analysis of Change from Baseline in FEV1 (ml)
Measured post-bronchodilator

| Visit | N | Treatmen | t Arm | l | n | Posterior<br>Median | 95% Credible<br>Interval |
|---|---|---|---|---|---|---|---|
| Day 14 | Х | Placebo | | | Х | X.XX | (x.xx, x.xx) |
| | X | GSK2269557 | 12.5 | mcg | X | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 50 | mcg | X | x.xx | (x.xx, x.xx) |
| | Х | GSK2269557 | 100 | mcg | X | x.xx | (x.xx, x.xx) |
| | Х | GSK2269557 | 250 | mcg | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 500 | mcg | X | x.xx | (x.xx, x.xx) |
| | X | GSK2269557 | 750 | mcg | Х | X.XX | (x.xx, x.xx) |
| Day 28 | Х | Placebo | | | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 12.5 | mcg | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 50 | mcg | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 100 | mcg | X | x.xx | (x.xx, x.xx) |
| | Х | GSK2269557 | 250 | mcg | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 500 | mcg | Х | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 | 750 | mcg | Х | X.XX | (x.xx, x.xx) |

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Statistical Analysis of Change from Baseline in FEV1 (ml)
Measured post-bronchodilator

| Visit | Treatment | Compariso | on | Adjusted<br>Median<br>Difference | Std Dev | 95% Credible<br>Interval | Prob Treat. Diff >0 (%) |
|---|---|---|---|---|---|---|---|
| Day 14 | GSK2269557<br>Placebo | 12.5 mg | VS | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557<br>Placebo | 50 mg | vs | x.xx | x.xx | (x.xx, x.xx) | X.XX |
| | GSK2269557<br>Placebo | 100 mg | vs | x.xx | x.xx | (x.xx, x.xx) | X.XX |
| | GSK2269557<br>Placebo | 250 mg | vs | x.xx | x.xx | (x.xx, x.xx) | X.XX |
| | GSK2269557<br>Placebo | 500 mg | vs | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557<br>Placebo | 750 mg | vs | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| Day 28 | GSK2269557<br>Placebo | 12.5 mg | vs | x.xx | X.XX | (x.xx, x.xx) | x.xx |
| | GSK2269557<br>Placebo | 50 mg | VS | x.xx | X.XX | (x.xx, x.xx) | X.XX |
| | GSK2269557<br>Placebo | 100 mg | vs | X.XX | x.xx | (x.xx, x.xx) | X.XX |

200879

## 13.12.5. Example Shell 5

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Number of moderate/severe exacerbations per subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |
| 4 | 0 | 2 (2%) |
| 5 | 0 | 1 (1%) |
| >5 | 0 | 1 (1%) |
| Subjects with >=1 moderate/severe exacerbation | 13 (13%) | 28 (28%) |
| Total Number of moderate/severe exacerbations | 21 | 49 |
| Number of moderate exacerbations per Subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |

200879

### 13.12.6. Example Shell 6

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Statistical Analysis of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Moderate/severe exacerbations Annual exacerbation rate (95% CrI) Active vs. Placebo Ratio Pr Diff <1 Percent reduction in rate (95% CrI) | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx)<br>0.85 (x.xx, x.xx)<br>x.xx<br>15% (x.xx, x.xx) |
| Predictive probability (%) [1] [only when required] | | xx% |
| Moderate exacerbations | | |
| Annual exacerbation rate (95% CrI) | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx) |
| Active vs. Placebo | | |
| Ratio | | 0.85 (x.xx, x.xx) |
| Pr Diff <1 | | x.xx |
| Percent reduction in rate (95% CrI) | | 15% (x.xx, x.xx) |

<sup>[1]</sup> Predictive posterior probability of success at end of study, where success is Pr(Reduction>0%)>80%

200879

## 13.12.7. Example Shell 7

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Duration at Screening

| | Treatme (N=100) | | Treatme<br>(N=100) | | Total (N=200) | |
|---|---|---|---|---|---|---|
| Duration of COPD: | | | | | | |
| n | 100 | | 99 | | 199 | |
| <1 year | XX | (x%) | XX | (x%) | XX | (x%) |
| >=1 to <5 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=5 to <10 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=10 to <15 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=15 to <20 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=20 to <25 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=25 years | XX | (x%) | XX | (x%) | XX | (x%) |

200879

### 13.12.8. Example Shell 8

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary and Analysis of Time to Next On-treatment Moderate/Severe Exacerbation (days)

up to Day 84

| | Treatment A (N=100) | Treatment B (N=100) |
|-------------------------------|---------------------|---------------------|
| Number of Subjects with Event | 10 (10%) | 14 (14%) |
| Number of Subjects Censored | 90 (90%) | 86 (86%) |

Treatment A vs. Placebo Hazard Ratio 95% Credible Interval

X.XX (x.xx, x.xx)

Note: Hazard ratio and 95% Credible Interval are from a Bayesian Cox proportional hazards model

200879

### 13.12.9. Example Shell 9

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Statistical Analysis of Proportion of Participants Achieving EXACT-definition of Response

| | Treatment A (N=100) | |
|---------------------------|---------------------|-------------------------|
| Day 14 | | |
| n | x.xx | x.xx |
| Responder | x.xx (x%) | x.xx (x%) |
| Non-responder | x.xx (x%) | x.xx (x%) |
| Active vs. Placebo | | |
| Odds Ratio (OR) (95% CrI) | x.xx (x.xx, | x.xx) x.xx (x.xx, x.xx) |
| Pr OR >1 x. | XX X. | xx |
| Day 28 | | |
| n | x.xx | x.xx |
| Responder | x.xx (x%) | x.xx (x%) |
| Non-responder | x.xx (x%) | x.xx (x%) |
| Active vs. Placebo | | |
| Odds Ratio (95% CrI) | x.xx (x.xx, x.x | (x) x.xx (x.xx, x.xx) |
| Pr Diff >1 | X.XX | x.xx |

200879

### 13.12.10. Example Shell 10


Population: Intent-to-Treat/Safety/Other study specific

Table

Summary of severity of subsequent HCRU-defined exacerbation during 12-Week Treatment Period

| Treatment | N | n | Mean | SD | Median | Min. | Max. |
|-----------|----|----|-------|-------|--------|-------|-------|
| Placebo | 30 | 30 | xx.xx | XX.XX | XX.XX | xx.xx | XX.XX |
| Trt A | 30 | 30 | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| Trt B | 30 | 30 | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |

200879

## 13.12.11. Example Shell 11

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Mixed Model Repeated Measures Analysis of CAT Total Score

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Day 28 | | |
| n | X.XX | x.xx |
| Adjusted mean score change (SE)<br>Active - Placebo | x.xx (x) | x.xx (x) |
| Difference (SE) | x.xx (x.xx) | x.xx (x.xx) |
| 95% (CrI) | X.XX | x.xx |
| Pr Diff >0 | x.xx | X.XX |
| Day 56 | | |
| n | X.XX | X.XX |
| Adjusted mean score change (SE)<br>Active - Placebo | x.xx (x) | x.xx (x) |
| Difference (SE) | x.xx (x.xx) | x.xx (x.xx) |
| 95% (CrI) | X.XX | X.XX |
| Pr Diff >0 | X.XX | x.xx |

200879

### 13.12.12. Example Shell 12

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | | | atment B<br>100) |
|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | , | 7%) 19<br>3%) 81 | (19%)<br>(81%) |
| Number of Home Visits (day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | | 100<br>0%) 92<br>4%) 4<br>0<br>0<br>2 | (92%)<br>(4%)<br>(<1%) |
| Number of Home Visits (night) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>100 (10<br>0<br>0<br>0<br>0 | 100<br>0%) 100<br>0<br>0<br>0 | (100%) |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Office/Practice Visits | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 911<br>846 (93%)<br>42 (5%)<br>13 (1%)<br>7 (<1%)<br>3 (<1%) | 899<br>808 (90%)<br>58 (6%)<br>23 (3%)<br>8 (<1%)<br>2 (<1%)<br>140 |
| Number of Urgent Care/Outpatient Visits | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 911<br>886 (97%)<br>15 (2%)<br>3 (<1%)<br>3 (<1%)<br>4 (<1%)<br>54 | 899<br>882 (98%)<br>10 (1%)<br>2 (<1%)<br>3 (<1%)<br>2 (<1%)<br>37 |
| Number of Emergency Room Visits | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 911<br>906 (>99%)<br>5 (<1%)<br>0<br>0<br>0<br>5 | 899<br>893 (>99%)<br>5 (<1%)<br>1 (<1%)<br>0<br>0 |

<sup>[1]</sup> Total number of contacts across all subjects.

PPD

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table 2.159

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Days in Intensive Care | n | 911 | 899 |
| | 1<br>2 | 910 (>99%)<br>0 | 894 (>99%)<br>0<br>1 (<1%) |
| | 3<br>>3 | 0<br>1 (<1%) | 0<br>4 (<1%) |
| | Total [2] | 12 | 40 (<1%) |
| Number of Days in General Ward | n | 911 | 899 |
| | 0<br>1 | 896 (98%)<br>0 | 878 (98%)<br>2 (<1%) |
| | 2 3 | 1 (<1%)<br>0 | 1 (<1%)<br>0 |
| | >3<br>Total [2] | 14 (2%)<br>119 | 18 (2%)<br>258 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

## 13.12.13. Example shell 13

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific



200879


# 13.12.14. Example Shell 14

Protocol: XYZ100001
Population: Intent-to-Treat/Safety/Other study specific

paracion: income to freat/barety/other beday specific

Summary of Baseline COPD Maintenance Therapy

| Therapy category | Treatment A (N=81) | A Treatment B (N=79) |
|---|---|---|
| Any medication at baseline | 70 (86%) | 50 (63%) |
| Monotherapy<br>LAMA only | X (x%)<br>x (x%) | X (x%)<br>x (x%) |
| Dual therapy<br>ICS/LABA<br>Dual bronchodilator | x (x%)<br>x (x%)<br>xx (xx%) | xx (x%)<br>x (x%) |
| Triple therapy LAMA/ICS/LABA | X (x%)<br>x (x%) | X (x%) |

200879

## 13.12.15. Example Shell 15


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of On-Treatment COPD Maintenance (Step-up) Therapy

| | Treatment A | Treatment B |
|---------------------|-------------|-------------|
| Therapy category | (N=81) | (N=79) |
| | | _ |
| Any Step-up Therapy | 70 (86%) | 50 (63%) |

200879

## 13.12.16. Example shell 16


Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of OCS use

| | Treatment A (N=81) | Treatment B (N=79) |
|---------------------------------|--------------------|--------------------|
| OCS use for index exacerbation | 81 (100%) | 79 (100%) |
| Total number of Days of OCS use | 01 (100%) | 75 (100%) |
| Mean | Xx | XX |
| SD | Xx | XX |
| Median | Xx | XX |
| Min. | Xx | XX |
| Max. | Xx | xx |
| On-treatment OCS use | xx (xx%) | xx (xx%) |
| Total number of Days of OCS use | | |
| Mean | Xx | xx |
| SD | Xx | XX |
| Median | Xx | XX |
| Min. | Xx | XX |
| Max. | Xx | XX |

200879

## 13.12.17. Example Shell 17


Population: Safety

Table X
Summary of Post-Inhalation Cough by Visit

Visit: VISIT 2 (RANDOMISATION)

| · · · | | acebo | 50 | K2269557<br>mcg<br>i=14) | 10 | K2269557<br>0 mcg<br>=15) | 25 | K2269557<br>0 mcg<br>=16) | 50 | SK2269557<br>)0 mcg<br>J=14) | 750 | (2269557<br>) mcg<br>=42) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Did subject experience PI cough? [1] | | | | | | | | | | | | |
| n | 20 | | 10 | | 12 | | 15 | | 1 | .2 | 35 | 5 |
| Yes | 7 | (35%) | 4 | (40%) | 6 | (50%) | 3 | (20%) | | 6 (50%) | 12 | 2 (34%) |
| No | 13 | (65%) | 6 | (60%) | 6 | (50%) | 12 | (80%) | | 6 (50%) | 23 | 8 (66%) |
| Type of cough | | | | | | | | | | | | |
| Single cough | 4 | (57%) | 2 | (50%) | 1 | (17%) | 1 | (33%) | 1 | (17%) | 2 | (17%) |
| Intermittent cough | 2 | (29%) | 2 | (50%) | 5 | (83%) | 1 | (33%) | 4 | (67%) | 5 | (42%) |
| Continuous cough | 1 | (14%) | 0 | | 0 | | 1 | (33%) | 1 | (17%) | 5 | (42%) |
| Severity of cough | | | | | | | | | | | | |
| Mild | 5 | (71%) | 3 | (75%) | 3 | (50%) | 2 | (67%) | 1 | (17%) | 6 | (50%) |
| Moderate | 2 | (29%) | 1 | (25%) | 2 | (33%) | 1 | (33%) | 5 | (83%) | 4 | (33%) |
| Severe | 0 | | 0 | | 1 | (17%) | 0 | | 0 | | 2 | (17%) |
| Time to onset of PI cough (minutes) | | | | | | | | | | | | |
| 0-1 | 6 | (86%) | 3 | (75%) | 6 | (100%) | 3 | (100%) | 6 | (100%) | 12 | (100%) |
| >1-2 | 1 | (14%) | 1 | (25%) | 0 | | 0 | | 0 | | 0 | |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| Duration of PI cough (minutes) | | | | | | | | | | | | |
| <=1 | 6 | (86%) | 3 | (75%) | 5 | (83%) | 3 | (100%) | 5 | (83%) | 11 | (92%) |
| >1-2 | 1 | (14%) | 1 | (25%) | 1 | (17%) | 0 | | 1 | (17%) | 1 | (8%) |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |

# 2019N398117\_00

200879

### CONFIDENTIAL

| >5-10 | Х | | Х | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| >10-30 | Х | | X | | | | | | | | |
| >30 | Х | | Х | | | | | | | | |
| Number of subjects reporting cough as AE/SAE Mild | 2<br>x | (29%)<br>(x%) | 1<br>x | (25%) | 4 | (67%) | 0 | 2 | (33%) | 3 | (25%) |
| Moderate | Х | (x%) | Х | | | | | | | | |
| Severe | Х | (x%) | Х | | | | | | | | |

<sup>[1]</sup> Percentages are calculated using the number of subjects evaluated at visit as the denominator.

All other percentages are calculated using the number of subjects with a PI cough at visit as the denominator.

200879


### 13.12.18. Example shell 18

Protocol: ABC123456

Population: Intent-to-Treat/Safety/Other study specific

Figure

Plot of Dose Response Model of Change from Baseline in FEV1



[Footnote to describe the fitted model]

200879

### 13.12.19. Example Shell 19

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | A Treatment B (N=100) |
|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | 97 (97%)<br>3 (3%) | |
| Number of Home Visits (day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>90 (90%)<br>4 (4%)<br>0<br>0<br>0<br>4 | 100<br>92 (92%)<br>4 (4%)<br>0<br>0<br>2 (<1%) |
| Number of Home Visits (night) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>100 (100%)<br>0<br>0<br>0<br>0 | 100<br>100 (100%)<br>0<br>0<br>0<br>0 |

<sup>[1]</sup> Total number of contacts across all subjects.

PPC

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Office/Practice Visits | n | 911 | 899 |
| | 0 | 846 (93%) | 808 (90%) |
| | 1 | 42 (5%) | 58 (6%) |
| | 2 | 13 (1%) | 23 (3%) |
| | 3 | 7 (<1%) | 8 (<1%) |
| | >3 | 3 (<1%) | 2 (<1%) |
| | Total [1] | 103 | 140 |
| Number of Urgent Care/Outpatient Visits | n | 911 | 899 |
| | 0 | 886 (97%) | |
| | 1 | | 10 (1%) |
| | 2 | | 2 (<1%) |
| | 3 | | 3 (<1%) |
| | >3 | 4 (<1%) | 2 (<1%) |
| | Total [1] | 54 | 37 |
| Number of Emergency Room Visits | n | 911 | 899 |
| | 0 | 906 (>99%) | |
| | 1 | 5 (<1%) | |
| | 2 | 0 | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 0 | 0 |
| | Total [1] | 5 | 7 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Days in Intensive Care | n | 911 | 899 |
| | 0 | 910 (>99%) | 894 (>99%) |
| | 1 | 0 | 0 |
| | 2 | 0 | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 1 (<1%) | 4 (<1%) |
| | Total [2] | 12 | 40 |
| Number of Days in General Ward | n | 911 | 899 |
| | 0 | 896 (98%) | 878 (98%) |
| | 1 | 0 | 2 (<1%) |
| | 2 | 1 (<1%) | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 14 (2%) | 18 (2%) |
| | Total [2] | 119 | 258 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

## 13.12.20. Example Shell 20


Population: Intent-to-Treat/Safety/Other study specific

Summary of Non-COPD Related Unscheduled Healthcare Resource Utilization

| | | | ment A<br>0) | Treatment B (N=100) | |
|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | | (97%)<br>(3%) | 19<br>81 | (19%)<br>(81%) |
| Number of Days in Accident and emergency | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>90<br>4<br>0<br>0<br>0 | (90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2<br>4 | (92%)<br>(4%)<br>(<1%) |
| Number of Days in General Ward | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>100 (<br>0<br>0<br>0 | 100%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) |

200879

# 13.12.21. Example Shell 21

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of Exacerbation Related Hospitalizations

| | Treatment A (N=100) | |
|-----------------------------------|---------------------|------|
| Index exacerbation | | |
| Participants with hospitalization | x.xx | x.xx |
| Number of hospitalizations | x.xx | x.xx |
| Mean duration (days) | X.XX | x.xx |
| SD | X.XX | x.xx |
| Median duration (days) | X.XX | x.xx |
| Minimum duration (days) | x.xx | X.XX |
| Maximum duration (days) | X.XX | X.XX |
| Subsequent exacerbations | | |
| Participants with hospitalization | X.XX | x.xx |
| Number of hospitalizations | X.XX | x.xx |
| Mean duration (days) | X.XX | x.xx |
| SD | X.XX | x.xx |
| Median duration (days) | X.XX | x.xx |
| Minimum duration (days) | X.XX | x.xx |
| Maximum duration (days) | X.XX | X.XX |
200879

# 13.12.22. Example Shell 22

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Re-hospitalization Within 30 days of Index Exacerbation

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Re-hospitalization Within 30 days | Yes | 97 (97%) | 19 (19%) |
| | No | 3 (3%) | 81 (81%) |

200879

# 13.12.23. Example Shell 23


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Subsequent Exacerbation Treatment

| | Treatment A (N=81) | Treatment B (N=79) |
|-------------------------|--------------------|--------------------|
| Subsequent exacerbation | 70 (86%) | 50 (63%) |
| ocs | X (x%) | X (x%) |
| Antibiotics | x (x%) | x (x%) |
| OCS and antibiotics | X (x%) | X (x%) |

200879

# 13.12.24. Example Shell 24

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Time from Resolution of Index Exacerbation to Next Exacerbation

| | Treatment A (N=100) | Treatment B (N=100) |
|-------------------------|---------------------|---------------------|
| Subsequent exacerbation | X.XX | X.XX |
| Mean duration (days) | x.xx | x.xx |
| SD | X.XX | x.xx |
| Median duration (days) | x.xx | x.xx |
| Minimum duration (days) | X.XX | x.xx |
| Maximum duration (days) | x.xx | X.XX |

200879

# 13.12.25. Example Shell 25


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of ECG Abnormalities for Participants with Any Abnormal Clinically Significant ECG Interpretation

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Visit 2 (Day 1) | | |
| Abnormal - Clinically significant | 10 (10%) | 15 (15%) |
| Any finding | 5 (50%) | 5 (33%) |
| ST depression | 5 (50%) | 5 (33%) |
| Short PR Interval | 0 | 5 (33%) |
| T wave inversion | 0 | 5 (33%) |

Includes Scheduled, unscheduled and Early Withdrawal visits. Participants may have more than one abnormality at each visit.

200879

# 13.12.26. Example Shell 26


Population: Intent-to-Treat/Safety/Other study specific

Table X

Statistical Analysis of Change from Baseline in FEV1 (mL) (Dose Response Model)  $\qquad \qquad \text{Measured post-bronchodilator}$ 

| | Placebo<br>(N=xx) | DNX 5mg (N=xx) | DNX 10mg<br>(N=xx) | DNX 25mg<br>(N=xx) | DNX 35mg<br>(N=xx) | DNX 50mg (N=xx) |
|---|---|---|---|---|---|---|
| n [1] | xx | xx | xx | xx | xx | xx |
| Posterior Adj. Median Change<br>95% HPD Credible Interval | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) | x.xx<br>(x.xx,x.xx) |
| Active - Placebo<br>Posterior Adj. Median<br>Difference | | x.xx | x.xx | x.xx | x.xx | x.xx |
| 95% HPD Credible Interval | | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) | (x.xx,<br>x.xx) |
| <pre>Prob(Difference&gt;0) Predictive probability (%) [2] [only if required]</pre> | | xx%<br>xx% | xx%<br>xx% | xx%<br>xx% | xx%<br>xx% | xx% |

<sup>[2]</sup> Predictive posterior probability of success at end of study, where success is Pr(Difference>0)>90%. Note: Model fitted was a....[insert as appropriate].



<sup>[1]</sup> Number of subjects with data contributing to the analysis.

200879

# 13.12.27. Example Shell 27

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of QTc(F) (msec) Categories

| | Treatment A (N=100) | Treatment B (N=100) |
|------------------|---------------------|---------------------|
| Screening | | |
| n | XX | xx |
| <=450 | xx (xx%) | xx (xx%) |
| >450 to <=480 | xx (xx%) | xx (xx%) |
| >480 to <=500 | xx (xx%) | xx (xx%) |
| >500 | xx (xx%) | xx (xx%) |
| Day 1 (Baseline) | | |
| n | xx | xx |
| <=450 | xx (xx%) | xx (xx%) |
| >450 to <=480 | xx (xx%) | xx (xx%) |
| >480 to <=500 | xx (xx%) | xx (xx%) |
| >500 | xx (xx%) | xx (xx%) |
| Day 14 | | |
| n | xx | xx |
| <=450 | xx (xx%) | xx (xx%) |
| >450 to <=480 | xx (xx%) | xx (xx%) |
| >480 to <=500 | xx (xx%) | xx (xx%) |
| >500 | xx (xx%) | xx (xx%) |

200879

# 13.12.28. Example Shell 28


Population: Safety

| Visit 2 | (Day 1) |
|---------|---------------------|
| mrma af | asuah. Cinala asuah |

>30

| Type of cough: Single cough | Treatment A (N=100) |
|-------------------------------------|---------------------|
| Did subject experience event [1]? | 12 (24%) |
| Cough severity | |
| Mild | 6 (50%) |
| Moderate | 5 (42%) |
| Severe | 1 (8%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 2 (17%) |
| >1-2 | 3 (25%) |
| >2-3 | 4 (33%) |
| >3-4 | 3 (25%) |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 7 (58%) |
| >1 - 2 | 2 (17%) |
| >2 - 3 | 3 (25%) |
| >3 - 4 | 0 |
| >4 - 5 | 0 |
| >5 - 10 | 0 |
| >10 - 30 | 0 |

<sup>[1]</sup> Percentages are calculated using the number of subjects evaluated at visit as the denominator.

All other percentages are calculated using the number of subjects with particular cough type at visit as the denominator.

# 2019N398117\_00


200879

Protocol: ABC123456
Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

Visit 2 (Day 1)
Type of cough: Single cough

Number of subjects reporting cough as AE/SAE

Mild

Moderate

Severe

Treatment A

(N=100)

2 (17%)
2 (17%)

200879

Protocol: ABC123456

Population: Safety


#### 

| Visit 2 (Day 1) Type of cough: Intermittent cough | Treatment A (N=100) |
|---------------------------------------------------|---------------------|
| Did subject experience event [1]? | 11 (22%) |
| Cough severity | |
| Mild | 2 (18%) |
| Moderate | 6 (55%) |
| Severe | 3 (27%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 1 (9%) |
| >1-2 | 4 (36%) |
| >2-3 | 6 (55%) |
| >3-4 | 0 |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 0 |
| >1 - 2 | 3 (27%) |
| >2 - 3 | 6 (55%) |
| >3 - 4 | 1 (9%) |
| >4 - 5 | 0 |
| >5 - 10 | 0 |
| >10 - 30 | 1 (9%) |
| >30 | 0 |

200879


Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

| Visit 2 (Day 1) Type of cough: Intermittent cough | Treatment A<br>(N=100) |
|---|---|
| Number of subjects reporting cough as AE/SAE<br>Mild<br>Moderate | 5 (45%)<br>1 (9%)<br>2 (18%) |
| Severe | 2 (18%) |

200879

Protocol: ABC123456
Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

| Visit 2 (Day 1) Type of cough: Continuous cough | Treatment A (N=100) |
|---|---|
| Did subject experience event [1]? | 4 (8%) |
| Cough severity Mild Moderate Severe | 1 (25%)<br>2 (50%)<br>1 (25%) |
| Time to onset of PI cough (minutes) 0-1 >1-2 >2-3 >3-4 >4-5 >5 | 3 (75%)<br>1 (25%)<br>0<br>0<br>0 |
| Duration of PI cough (minutes) <=1 >1 - 2 >2 - 3 >3 - 4 >4 - 5 >5 - 10 >10 - 30 >30 | 0<br>0<br>0<br>1 (25%)<br>1 (25%)<br>0<br>1 (25%)<br>1 (25%) |

200879


Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

Visit 2 (Day 1)

| Type of cough: Continuous cough | Treatment A (N=100) |
|---|---|
| Number of subjects reporting cough as AE/SAE Mild Moderate Severe | 2 (50%)<br>1 (25%)<br>1 (25%)<br>0 |

REPEAT FOR EACH VISIT

200879

# 13.12.29. Example Shell 29

Protocol: MID200879

Population: Intent-to-Treat

| Randomized<br>Treatment | Centre/<br>Subj | Start<br>Date of<br>Dosing | End<br>Date of<br>Dosing | Duration<br>(Days) | Dispense Visit | Dispense<br>Date | Actual<br>Treatment<br>Dispensed |
|---|---|---|---|---|---|---|---|
| GSK2269557 500 mcg | PPD | xxxxxxxx | xxxxxxxx | XX | Visit 3 (Week 0) | XXFEB2013 | GSK2269557 500 mcg |
| | | XXXXXXXXX<br>XXXXXXXXX | XXXXXXXXX<br>XXXXXXXXX | XX<br>XX | Visit 5 (Week 4)<br>Visit 6 (Week 8) | | GSK2269557 100 mcg<br>GSK2269557 500 mcg |

200879

# 13.12.30. Example Shell 30


Population: Intent-to-Treat/Safety/Other study specific

 $Figure \ X \\ Kaplan-Meier \ Plot \ of \ Time \ to \ Next \ On-treatment \ Exacerbation \ During \ the \ 12-Week \ Treatment \ Period$ 



200879

# 13.12.31. Example Shell 31


Population: Intent-to-Treat/Safety/Other study specific

 $Figure \ X \\ Plot \ of \ Repeated \ Measures \ Model \ of \ Change \ from \ Baseline \ in \ FEV1 \ Measured \ Post-bronchodilator \\$ 



200879

# 13.12.32. Example Shell 32

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Efficiency Ratio for Possible Adaptions to Randomization Ratio

| | Median | 10 <sup>th</sup> Percentile |
|---|---|---|
| Design 1: Add 25mcg dose | xx | xx |
| Design 2: Add 25mcg dose, drop 500mcg dose | XX | XX |
| Design 3: Add 25mcg dose, drop 250 mcg and 500 mcg doses | XX | XX |
| Design 4: Drop 12.5mcg dose | XX | XX |
| Design 5: Drop 12.5mcg and 50mcg doses | XX | XX |

200879

# 13.12.33. Example Shell 33


Population: Safety

Table X
Summary of Post-Inhalation (PI) Cough at Any Visit

| | | acebo<br>=43) | 50 | mcg | 10 | K2269557<br>0 mcg<br>=15) | 250 | (2269557<br>) mcg<br>=16) | 500 | 2269557<br>mcg<br>14) | 750 | (2269557<br>) mcg<br>=42) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Did subject experience PI cough at any vi<br>Yes | | ?<br>(xx%) | Х | (xx%) | Х | (xx%) | Х | (xx%) | Х | (xx%) | X | (xx%) |
| No | Χ | . , | Χ | (xx%) | Χ | , , | Χ | (xx%) | | (xx%) | Χ | (xx%) |
| Maximum Severity of cough | | | | | | | | | | | | |
| Mild | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Χ | (xx%) | Х | (xx%) |
| Moderate | Χ | (xx%) | X | (xx%) | Χ | (xx%) | Χ | (xx) | Χ | (xx%) | Χ | (xx%) |
| Severe | 0 | | 0 | | Χ | (xx%) | 0 | | 0 | | Χ | (xx%) |
| Maximum Duration of PI cough (minutes)[1 | ] | | | | | | | | | | | |
| Mean | Х | | Х | | Х | | Х | | Х | | Х | |
| SD | Х | | X | | Х | | Х | | Х | | Х | |
| Median | Х | | Х | | Х | | Х | | Х | | Х | |
| Minimum | Х | | X | | Х | | Х | | Х | | Х | |
| Maximum | X | | Х | | Х | | Х | | Х | | Х | |
| Number of occurrences of PI cough | | | | | | | | | | | | |
| 0 | Х | | Х | | Х | | Х | | Х | | Х | |
| 1 | Х | | Х | | Х | | Х | | Х | | Х | |
| 2 | Х | | Х | | Х | | Х | | Х | | Х | |
| 3 | Х | | Х | | Х | | Х | | Х | | Х | |
| 4 | Х | | Х | | Х | | Х | | Х | | Х | |

[1] Duration from the maximum severity cough

#### The GlaxoSmithKline group of companies

200879

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Phase IIb, Randomized (Stratified), Double-Blind (Sponsor Open), Parallel-Group, Placebo-Controlled, Dose-Finding Study of Nemiralisib (GSK2269557) Added to Standard of Care (SoC) Versus SoC Alone in Participants Diagnosed with an Acute Moderate or Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD) |
|---|---|---|
| <b>Compound Number</b> | : | GSK2269557 |
| <b>Effective Date</b> | : | 08-MAR-2018 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200879 and at the planned interim analyses.
- This RAP is intended to describe the efficacy, safety and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

RAP Author(s): PPD

Statistics Leader, (Respiratory Clinical Statistics)

| Approver | Date | Approval Method |
|---|---|---|
| TA Director (Respiratory Clinical Statistics) | 07-MAR-2018 | Email |
| PPD | | |
| Programming Manager (Respiratory Clinical Programming) | 08-MAR-2018 | Email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

200879

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Programmer (Respiratory Clinical Programming) | 07-MAR-2018 | Email |
| PPD Clinical Development Director (Respiratory) | 07-MAR-2018 | Email |
| Clinical Development Manager (Respiratory) | 06-MAR-2018 | Email |
| Medical Director (Global Clinical Safety and Pharmacovigilance) | 06-MAR-2018 | Email |
| PPD Manager, Clinical Pharmacology (Clinical Pharmacology Modelling and Simulation) | 06-MAR-2018 | Email |
| Director, Patient Centred Outcomes (Value Evidence & Outcomes) | 02-MAR-2018 | Email |

200879

# **TABLE OF CONTENTS**

| 2. SUMMARY OF KEY PROTOCOL INFORMATION 8 2.1. Study Objective(s) and Endpoint(s). 8 2.2. Study Design 11 3. PLANNED ANALYSES 11 3.1. Interim Analyses 13 3.1.1. Futility analyses 13 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING 16 CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4.1. Covariates and Subgroups 17 5.4.2. Examination of Covariates and Subgroups 17 5.5. Other Considerations for Data Analyses and Data Handling 18 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 | | | | | PAGE |
|---|---|---|---|---|---|
| 2.1. Study Objective(s) and Endpoint(s) | 1. | INTRO | ODUCTIO | N | 8 |
| 2.1. Study Objective(s) and Endpoint(s) | 2 | CLIMA | | KEY PROTOCOL INFORMATION | Q |
| 2.2. Study Design 11 3. PLANNED ANALYSES 11 3.1. Interim Analyses 11 3.1.1. Futility analyses 13 3.1.1.1. Futility rules 14 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.2.1. Statistical Analyses 22 7.2.1.1. Statistical analyses 22 7.2.1.2. Subgroup analyses 24 7.2.1.3. Ex | ۷. | | | | |
| 3. PLANNED ANALYSES 11 3.1. Interim Analyses 13 3.1.1. Futility analyses 13 3.1.1.1. Futility rules 14 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Statistical Analyses 22 7.1.3. Sensitivity and Supportive Analyses 22 7.2.1. Rate of exacerbations | | | Study D | Design | 0<br>11 |
| 3.1.1 Interim Analyses 11 3.1.1.1 Futility analyses 13 3.1.1.1 Futility rules 14 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING 16 CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 18 Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1 Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Endpoint 20 7.1.2.1 Model Checking & Diagnostics 20 7.1.2.1 Primary Statistical Analyses 20 7.1.2.1 Subgroup Analyses 22 7.1.3. Sessitivity and Supportiv | | ۷.۷. | Study D | /esigit | 11 |
| 3.1.1 Interim Analyses 11 3.1.1.1 Futility analyses 13 3.1.1.1 Futility rules 14 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING 16 CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 18 Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1 Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Endpoint 20 7.1.2.1 Model Checking & Diagnostics 20 7.1.2.1 Primary Statistical Analyses 20 7.1.2.1 Subgroup Analyses 22 7.1.3. Sessitivity and Supportiv | 3. | PLAN | NED ANA | ALYSES | 11 |
| 3.1.1. Futility analyses 3.1.1.1. Futility rules 14 3.2. Final Analyses 14 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.1.5. Secondary Efficacy Analyses 22 7.1.1. Rate of exacerbations 23 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 24 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 7.2.3. Subgroup analyses 26 7.2.3. Subgroup analyses | | | | | |
| 3.1.1.1 Futility rules 14 3.2 Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1 Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1 Study Treatment & Sub-group Display Descriptors 16 5.1 Study Treatment & Sub-group Display Descriptors 16 5.2 Baseline Definitions 16 5.3 Multicentre Studies 17 5.4 Examination of Covariates and Subgroups 17 5.4.1 Covariates 17 5.4.2 Examination of Subgroups 18 5.5 Other Considerations for Data Analyses and Data Handling Conventions 19 6 STUDY POPULATION ANALYSES 19 6.1 Overview of Planned Study Population Analyses 19 6.1.1 Concomitant medications 19 7 EFFICACY ANALYSES 20 7.1 Primary Efficacy Analyses 20 7.1.1 Primary Endpoint 20 7.1.2 Primary Statistical Analyses 20 | | | | | |
| 3.2. Final Analyses 14 4. ANALYSIS POPULATIONS 15 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Gradical Analyses 20 7.1.2. Secondary Efficacy Analyses 22 7.2. Secondary Efficacy Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Statistical analyses 24 7.2.1. Statistical analyses 24 7.2.1. Exploratory a | | | | | |
| 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.4. Subgroup Analyses 22 7.1.1. Statistical analyses 22 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.1. Statistical analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from bas | | 3.2. | Final Ar | | |
| 4.1. Protocol Deviations 15 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.4. Subgroup Analyses 22 7.1.1. Statistical analyses 22 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.1. Statistical analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from bas | 4 | A N I A I | VOIC DO | DI II ATIONIC | 4.5 |
| 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING 16 CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Vis | 4. | | | | |
| CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.1.2. Secondary Efficacy Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1. Subgroup analyses 24 7.2.1. Subgroup analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 | | 4.1. | Protoco | i Deviations | 15 |
| CONVENTIONS 16 5.1. Study Treatment & Sub-group Display Descriptors 16 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.1.2. Secondary Efficacy Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1. Subgroup analyses 24 7.2.1. Subgroup analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 | 5. | CONS | SIDERAT | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Statistical Analyses 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 < | | | | | 16 |
| 5.2. Baseline Definitions 16 5.3. Multicentre Studies 17 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1.1. Primary Efficacy Analyses 20 7.1.2. Primary Statistical Analyses 20 7.1.2. Primary Statistical Analyses 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 < | | | | | |
| 5.4. Examination of Covariates and Subgroups 17 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 22 7.1.2. Primary Statistical Analyses 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. | | 5.2. | Baseline | e Definitions | 16 |
| 5.4.1. Covariates 17 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 22 7.1.2. Primary Statistical Analyses 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.1. Statistical analyses 24 7.2.2. Time to next exacerbation 25 7.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 | | 5.3. | | | |
| 5.4.2. Examination of Subgroups 18 5.5. Other Considerations for Data Analyses and Data Handling Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 22 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | 5.4. | Examin | | |
| 5.5. Other Considerations for Data Analyses and Data Handling Conventions | | | | | |
| Conventions 19 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.1. Statistical analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | 18 |
| 6. STUDY POPULATION ANALYSES 19 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | 5.5. | | | 40 |
| 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | Conven | itions | 19 |
| 6.1. Overview of Planned Study Population Analyses 19 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | 6. | STUD | Y POPUI | LATION ANALYSES | 19 |
| 6.1.1. Concomitant medications 19 7. EFFICACY ANALYSES 20 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1. Statistical analyses 24 7.2.1.1. Statistical analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses < | | | | | |
| 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | |
| 7.1. Primary Efficacy Analyses 20 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | |
| 7.1.1. Primary Endpoint 20 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | 7. | | | | |
| 7.1.2. Primary Statistical Analyses 20 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2.1. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.1. Statistical analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | 7.1. | • | | |
| 7.1.2.1. Model Checking & Diagnostics 22 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | |
| 7.1.3. Sensitivity and Supportive Analyses 22 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | 7.1.2. | | |
| 7.1.4. Subgroup Analyses 22 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | <b>-</b> 4 0 | | |
| 7.2. Secondary Efficacy Analyses 23 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | |
| 7.2.1. Rate of exacerbations 23 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | 7.0 | | | |
| 7.2.1.1. Statistical analyses 24 7.2.1.2. Subgroup analyses 24 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | 7.2. | | | |
| 7.2.1.2. Subgroup analyses | | | 7.2.1. | | |
| 7.2.1.3. Exploratory analyses 24 7.2.2. Time to next exacerbation 25 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | | | |
| 7.2.2. Time to next exacerbation | | | | | |
| 7.2.2.1. Statistical analyses 25 7.2.2.2. Subgroup analyses 26 7.2.3. Change from baseline in Clinic Visit trough FEV1 26 7.2.3.1. Statistical Analyses 26 7.2.3.2. Subgroup analyses 26 | | | 7 2 2 | | |
| 7.2.2.2. Subgroup analyses | | | 1.2.2. | | |
| 7.2.3. Change from baseline in Ćlinic Visit trough FEV <sub>1</sub> | | | | <b>,</b> | |
| 7.2.3.1. Statistical Analyses | | | 722 | | |
| 7.2.3.2. Subgroup analyses26 | | | 1.2.3. | | |
| | | | 724 | | |

200879

| | | | 7.2.4.1. | Statistical analyses | 27 |
|---|---|---|---|---|---|
| | | 7.2.5. | EXAcerba | tions of Chronic Pulmonary Disease Tool - | |
| | | | | eported Outcome (EXACT) | 27 |
| | | | 7.2.5.1. | Proportion of participants achieving EXACT- | |
| | | | | defined recovery from index exacerbation | 28 |
| | | | 7.2.5.2. | Time to EXACT-defined recovery from index | |
| | | | | exacerbation | 28 |
| | | | 7.2.5.3. | Severity of subsequent HCRU-defined | |
| | | | | exacerbation(s) defined by EXACT | 28 |
| | | | 7.2.5.4. | Statistical analyses | 29 |
| | | | 7.2.5.5. | Subgroup analyses | |
| | | | 7.2.5.6. | Sensitivity and supportive analyses | |
| | | 7.2.6. | | sessment Test (CAT) | |
| | | | 7.2.6.1. | Proportion of responders using the CAT | |
| | | | 7.2.6.2. | Change from baseline in CAT Total Score | |
| | | | 7.2.6.3. | Statistical analyses | |
| | | | 7.2.6.4. | Subgroup analyses | 31 |
| | | 7.2.7. | | e's Respiratory Questionnaire for COPD | |
| | | | | SGRQ-C) | 31 |
| | | | 7.2.7.1. | Proportion of responders on the SGRQ Total | |
| | | | | Score | |
| | | | 7.2.7.2. | Change from baseline in SGRQ Total Score | |
| | | | 7.2.7.3. | Statistical analyses | |
| | | | 7.2.7.4. | Subgroup analyses | |
| | | 7.2.8. | | nedication use | 33 |
| | | | 7.2.8.1. | Rescue medication use via the clip-on | |
| | | | | Propeller Sensor for MDI | 34 |
| | | | 7.2.8.2. | Statistical analyses | |
| | 7.3. | | | / Analyses | |
| | | 7.3.1. | - | om Day 84 in Clinic Visit trough FEV <sub>1</sub> | |
| | | | 7.3.1.1. | Statistical analysis | |
| | | 7.3.2. | | PD (Evaluating Respiratory Symptoms in COPD) | |
| | | 7.3.3. | | of HCRU related to exacerbations | 35 |
| | | | 7.3.3.1. | Re-hospitalisation within 30 days of index | |
| | | | | exacerbation | 36 |
| | | | 7.3.3.2. | Time from resolution of index exacerbation to | |
| | | | | next exacerbation | |
| | | | 7.3.3.3. | Subsequent exacerbation treatment type | |
| | | 7.3.4. | Complian | ce | 36 |
| | | | 7.3.4.1. | Number of actuations of double-blind study | |
| | | | | treatment measured by the clip-on Propeller | |
| | | | | Sensor | 37 |
| | | 7.3.5. | | ory/infective markers in blood and sputum in | |
| | | | | acute exacerbation of COPD | |
| | | 7.3.6. | | ometry measurements | |
| | | 7.3.7. | Other PR | O symptoms suggestive of exacerbation | 37 |
| _ | | | | | |
| 8. | | | | | |
| | 8.1. | | | alyses | |
| | | 8.1.1. | | Events of Special Interest | 37 |
| | | | 8.1.1.1. | Post-inhalation Cough Immediately Following | |
| | | | | Dosing | 37 |

| | | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | 200879 |
|---|---|---|---|
| | 8.2.<br>8.3.<br>8.4. | Clinical Laboratory Analyses Other Safety Analyses Mortality | 38 |
| 9. | PHARI<br>9.1.<br>9.2. | MACOKINETIC ANALYSES Population of Interest Drug Concentration Measures | 38 |
| 10. | | LATION PK ANALYSIS Derived Pharmacokinetic Parameters | |
| 11. | PHARI | MACOKINETIC / PHARMACODYNAMIC | ANALYSES39 |
| 12. | REFER | RENCES | 40 |
| 13. | APPEN<br>13.1. | NDICES Appendix 1: Protocol Deviation Managen Protocol Population | nent and Definitions for Per |
| | 13.2. | <ul><li>13.1.1. Exclusions from Per Protocol P</li><li>Appendix 2: Assessment Windows</li><li>13.2.1. Definitions of Assessment Windows</li><li>13.2.1.1. Hospital discharge</li></ul> | opulation41 |
| | 13.3. | 13.3.1.1. 12-Week Treatment<br>13.3.1.2. 12-Week Follow-Up<br>13.3.2. Study Phases | t Emergent Adverse |
| | 13.4. | Appendix 4: Data Display Standards & H. 13.4.1. Reporting Process | dverse Events 44 andling Conventions 45 |
| | 13.5. | Appendix 5: Derived and Transformed Da 13.5.1. General | ata |
| | 13.6. | Appendix 6: Reporting Standards for Mis 13.6.1. Premature Withdrawals | |
| | 13.7. | Appendix 7: Values of Potential Clinical II<br>13.7.1. Laboratory Values<br>13.7.2. ECG | |
| | 13.8. | Appendix 8: Population Pharmacokinetic 13.8.1. Population Pharmacokinetic (Population | (PopPK) Analyses |
| | 13.9. | Appendix 9: Pharmacokinetic / Pharmacokinetic | |

| | | | 200879 |
|---|---|---|---|
| | 13.9.1. | Pharmacokinetic/Pharmacodynamic Methodology | 54 |
| 13.10. | | x 10: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 13 11 | | 11: List of Data Displays | |
| 10.11. | 13 11 1 | Data Display Numbering | 57 |
| | 13 11 2 | Mock Example Shell Referencing | 57<br>57 |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | 13.11.5. | 13.11.5.1. Efficacy tables for Interim Analysis 1 | |
| | | 13.11.5.2. Efficacy tables for Interim Analysis 2 | 03 |
| | | 13.11.5.3. Efficacy tables for End of Treatment Interim Analysis and SAC | 67 |
| | 40 44 0 | | |
| | 13.11.0. | Efficacy Figures | |
| | | 13.11.6.1. Efficacy Figures for Interim Analysis 1 | |
| | | 13.11.6.2. Efficacy Figures for Interim Analysis 2 | 80 |
| | | 13.11.6.3. Efficacy Figures for End of Treatment Interim | 00 |
| | | Analysis and SAC | |
| | | Safety Tables | |
| | 13.11.8. | Safety Figures | 87 |
| | | Pharmacokinetic Tables | |
| | | .ICH Listings | |
| | | .Non-ICH Listings | |
| 13.12. | | 12: Example Mock Shells for Data Displays | |
| | | Example shell 1 | |
| | | Example Shell 2 | |
| | | Example shell 3 | |
| | 13.12.4. | Example Shell 4 | 94 |
| | 13.12.5. | Example Shell 5 | 96 |
| | 13.12.6. | Example Shell 6 | 97 |
| | 13.12.7. | Example Shell 7 | 98 |
| | | Example Shell 8 | |
| | 13.12.9. | Example Shell 9 | 100 |
| | | .Example Shell 10 | |
| | | .Example Shell 11 | |
| | | .Example Shell 12 | |
| | 13.12.13 | .Example shell 13 | 106 |
| | 13.12.14 | .Example Shell 14 | 107 |
| | | Example Shell 15 | |
| | | Example shell 16 | |
| | | Example Shell 17 | |
| | | Example shell 18 | |
| | | Example Shell 19 | |
| | | Example Shell 20 | |
| | | Example Shell 21 | |
| | | Example Shell 22 | |
| | | Example Shell 23 | |
| | | Example Shell 24 | |
| | | Example Shell 25 | |
| | | Example Shell 26 | |
| | | Example Shell 27 | |
| | 10.14.41 | . LAGITING STICIT 41 | 143 |

| | 200879 |
|---------------------------|--------|
| 13.12.28.Example Shell 28 | 124 |
| 13.12.29.Example Shell 29 | |

200879

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 200879.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterise the dose response of<br>nemiralisib administered in addition to<br>SoC compared with placebo and SoC<br>in participants diagnosed with an<br>acute moderate or severe<br>exacerbation of COPD | Change from baseline in Clinic Visit trough forced expiratory volume in one second (FEV <sub>1</sub> ) at Day 84 measured post-bronchodilator |
| Secondary Objectives | Secondary Endpoints |
| To characterise the dose response and efficacy of nemiralisib administered in addition to SoC compared with placebo and SoC in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>Rate of moderate and severe exacerbations over the 12-Week Treatment Period</li> <li>Time to next moderate/severe exacerbation following index exacerbation</li> <li>Change from baseline in Clinic Visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days 14, 28, 56, and 84 (Day 84: post-bronchodilator is the primary endpoint; pre-bronchodilator is a secondary endpoint) and at hospital discharge (only for participants who are hospitalized for the index exacerbation)</li> <li>Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre- and post-bronchodilator at Days, 14, 28, 56, and 84 (in participants hospitalized for index exacerbation only)</li> </ul> |
| To evaluate the treatment effect of nemiralisib in addition to SoC compared with placebo and SoC on symptoms indicative of an exacerbation and on health status using Patient-Reported Outcomes (PROs) in participants diagnosed with an acute moderate or severe exacerbation of COPD | <ul> <li>EXAcerbations of Chronic Pulmonary Disease Tool (EXACT-PRO)</li> <li>Proportion of participants achieving the EXACT definition of recovery from the index exacerbation by Days 14, 28, 56, and 84</li> <li>Time to recovery from index exacerbation</li> <li>Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT</li> <li>COPD Assessment Test (CAT)</li> <li>Proportion of responders using the CAT at Treatment Days 28, 56, and 84, and following EXACT defined recovery from the index exacerbation</li> <li>Change from baseline (Day 1) in CAT total score at Days 28, 56, and 84 and following EXACT defined recovery from the index exacerbation</li> </ul> |

200879

| Objectives | Endpoints |
|---|---|
| To evaluate the usage of rescue<br>medication in patients diagnosed with<br>an acute moderate or severe<br>exacerbation of COPD | St. George's Respiratory Questionnaire (SGRQ) Total Score Proportion of responders on the SGRQ total score as measured by the SGRQ for COPD Patients (SGRQ-C) at Days 28, 56, and 84 Change from baseline (Day 1) in SGRQ total score at Days 28, 56, and 84 Rescue medication use (occasions/day), averaged over each week of treatment and over the 84-day treatment period The percentage of rescue-free days (24-hour periods) during each week of treatment and over the 84-day treatment period |
| To evaluate the population pharmacokinetics of nemiralisib in participants diagnosed with an acute moderate or severe exacerbation of COPD | Plasma nemiralisib concentrations and derived PK parameters (e.g., area under the curve [AUC (0-24) and AUC(0-t)], maximum concentration [Cmax], time at maximum concentration [Tmax], Ctrough) as appropriate will be collected in a subset of randomized participants (approximately 300) at selected sites as follows: trough (pre-dose) for the study treatment and post-dose for the study treatment from 0-1 hour and >1 to 6 hours on Days 14 and 28 of the 12-Week Treatment Period |
| To assess the safety and tolerability of<br>nemiralisib and placebo in participants<br>diagnosed with an acute moderate or<br>severe exacerbation of COPD | <ul> <li>Incidence of adverse events (AEs; including serious AEs and AE of Special Interest [AESI])</li> <li>Vital signs (pulse rate, systolic and diastolic blood pressure) (measured at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>12-lead electrocardiogram (ECG) assessments (performed at clinic Visits 1 [Screening], 3 [Day 14], 6 [Day 84], and 7 [Day 112] or Early Withdrawal Visit)</li> <li>Clinical laboratory tests (hematology and chemistry; performed at each clinic visit up through Visit 7 [Day 112] or Early Withdrawal Visit)</li> <li>Incidence of COPD exacerbations</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To further characterize the dose<br>response, and efficacy, of nemiralisib<br>administered in addition to SoC<br>compared with placebo and SoC in<br>participants diagnosed with an acute<br>moderate or severe exacerbation of<br>COPD | <ul> <li>Rate of mild exacerbations over the 12-Week Treatment Period</li> <li>Rate of all exacerbations (mild, moderate and severe combined) over the 12-Week Treatment Period</li> <li>Time to next exacerbation (mild, moderate and severe combined)</li> </ul> |

200879

| Objectives | Endpoints |
|---|---|
| To evaluate the treatment effect of nemiralisib in addition to SoC compared with placebo and SoC on symptom stability following an exacerbation using Patient-Reported Outcomes in participants diagnosed with an acute moderate or severe exacerbation of COPD | Stability of symptoms post recovery measured using E-RS:COPD (Evaluating Respiratory Symptoms in COPD) and subscales from Randomization (Visit 2) to Day 84 (Visit 6) |
| To explore the PK/PD relationship for<br>nemiralisib | Relationship between drug exposure and<br>Pharmacodynamic responses (e.g. efficacy, heart rate,<br>clinical laboratory analytes and blood biomarkers) in the<br>PK subset of participants (approximately 300) at selected<br>sites |
| To evaluate the treatment effect of<br>nemiralisib in addition to SoC<br>compared with placebo and SoC on<br>HCRU in participants who experience<br>a severe exacerbation of COPD | Measures of HCRU related to severe exacerbations (e.g., hospitalizations, length of hospital stay, re-hospitalization within 30 days, number of Emergency Room [ER] visits, etc.) |
| To evaluate compliance with study treatment | Number of actuations of the double-blind study treatment<br>as measured by the clip-on Propeller Sensor (for<br>countries where the Propeller Sensor for ELLIPTA is<br>available) |
| To evaluate inflammatory markers in<br>blood in relation to acute exacerbation<br>of COPD | <ul> <li>Blood samples collected at Screening through Visit 7 (as part of the clinical laboratory blood samples) for analysis of blood eosinophil counts and inflammatory mediators</li> <li>Blood samples for analysis of inflammatory biomarkers (including but not limited to: high sensitivity C-reactive protein [hs-CRP], chemokine interferon-γ inducible protein 10 kDa (CXCL10)], and procalcitonin) collected at Visit 1 (Screening)</li> </ul> |
| To evaluate inflammatory and infective markers in sputum in relation to acute exacerbation of COPD | Spontaneous sputum sample for analysis of inflammatory<br>and infective markers collected at Screening/Day 1 (pre-<br>dose) and Day 56 in participants who are willing and able<br>to provide a sample |
| To evaluate the potential post-<br>treatment impact of double-blind study<br>treatment during the 12-Week Post-<br>Treatment Follow-Up Period | <ul> <li>Change from baseline (Day 84) in Clinic Visit trough FEV1 measured pre- and postbronchodilator at Day 112, 140 and 168</li> <li>Rate of moderate and severe COPD exacerbation(s) during the 12-Week Follow-Up Period</li> <li>Rate of moderate and severe COPD exacerbation(s) over the 24 week study duration</li> <li>Time to next exacerbation following cessation of double blind study treatment</li> <li>Proportion of responders using the CAT at Days 112 and 168</li> <li>Change from baseline (Day 1) in CAT Total score at Days 112 and 168</li> <li>Proportion of responders on the SGRQ Total Score as measured by the SGRQ-C at Days 112 and 168</li> <li>Change from baseline (Day 1) in SGRQ total score at</li> </ul> |

200879

| Objectives | En | dpoints |
|------------|----|-----------------------------------------------------|
| | | Days 112 and 168 |
| | • | Severity of subsequent HCRU exacerbation defined by |
| | | EXACT |
| | • | E-RS: COPD and subscales from last dose of double- |
| | | blind study treatment |
| | • | Rescue medication use up to Day 112 |

# 2.2. Study Design

This is a Phase IIb, multicenter, randomized, stratified (by index COPD exacerbation severity [moderate or severe] and by whether or not the participant is in the PK Subgroup), double-blind (Sponsor Open), placebo-controlled, parallel-group study in participants who present with an acute moderate or severe exacerbation of COPD requiring Standard of Care (SoC).

This study consists of a Screening Period, a 12-Week Treatment Period and a 12-Week Post-Treatment Follow-Up Period. Randomization and the first dose of the double-blind study treatment administration (Visit 2/Day 1) should take place in the morning, as soon as possible following determination of eligibility and completion of the baseline measures, including the EXACT-PRO questionnaire for the day of randomization, and FEV<sub>1</sub> measurement and no later than 48 hours after the start of SoC.

PK Subgroup: Sparse PK sampling will be conducted in a subgroup of participants at selected sites. The PK Subgroup will be identical to the main study in terms of the study population, design, and conduct, with the exception of blood draws (3 per visit on Days 14 and 28) for PK analysis.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

Ongoing data reviews of unblinded safety data, conducted by an Internal Safety Review Committee (iSRC), will be performed throughout the trial. Details will be documented in the iSRC charter.

Interim analyses of the primary endpoint and key secondary endpoints to inform internal decision making will be conducted periodically throughout the trial. The first analysis (Interim Analysis 1) is planned to occur when approximately 170 participants complete 28 days of treatment, where approximately 50 of the 170 participants have an index exacerbation defined as severe. A change that could arise from this interim analysis is a specification of the stratification proportions by index exacerbation severity status (moderate or severe). This decision will be based on inspection of all available endpoints at the interim analysis.

Further interim analyses will be performed, depending on the observed recruitment rate. At least one interim analysis of the primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator will be performed to

200879

determine whether or not any adjustments to the randomization ratio across doses would help optimize the characterization of the dose response profile for nemiralisib. This analysis (Interim Analysis 2) is planned to occur when approximately 300 participants complete 84 days of treatment or when approximately 400 participants remain to be randomised, whichever occurs first. Adjustments could include ceasing randomization to an existing dose(s) of nemiralisib and/or modification of the allocation ratios for the existing nemiralisib doses and/or addition of a 25mcg dose. Other changes may include specification of the stratification proportions by index exacerbation severity status.

An interim analysis of efficacy data collected during the Double-Blind Treatment Period will be conducted when the last participant in the study has completed the 12-week Double-Blind Treatment Period (End of Treatment Interim Analysis). The aim of this analysis is to provide GSK with timely data to inform internal decision making, prior to the end of study.

The following table describes the endpoints that will be analysed/summarised at each interim:

| Interim | Purpose of interim | Endpoints |
|---|---|---|
| Interim Analysis 1 | To inform internal decision making | <ul> <li>Change from baseline in FEV<sub>1</sub> at Days 14, 28, 56 and 84 measured pre- and post-bronchodilator</li> <li>Change from hospital discharge in FEV<sub>1</sub> at Day 14, 28, 56 and 84 measured pre- and post-bronchodilator in participants hospitalized for the index exacerbation</li> <li>Other spirometry measures (percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio</li> </ul> |
| | | Summary of on-treatment exacerbations Summary of proportion of participants achieving EXACT-defined recovery by |
| | | Days 14, 28, 56 and 84 |

200879

| Interim | Purpose of interim | Endpoints |
|---|---|---|
| Interim Analysis 2 | To determine if any adjustments to the randomization ratio would help characterize the dose response profile for nemiralisib | Endpoints listed for Interim Analysis 1 and also: Rate of (on-treatment) exacerbations over the 12-Week Treatment Period Time to next (on-treatment) exacerbation during the 12-Week Treatment Period Analysis of proportion of participants achieving the EXACT-defined recovery by Days 14, 28, 56, and 84 Rescue medication use, as measured in eDiary |
| End of Treatment<br>Interim Analysis | To inform internal decision making | All endpoints to be reported as per<br>Statistical Analysis Complete (SAC)<br>deliverable |

The statistical methods of analyses are described in Section 7.

The Respiratory Data Sciences Group will apply machine learning techniques to the interim data to determine if identifiable phenotypic sub-population(s) of COPD participants are present at baseline, and if they result in different responses to Nemiralisib, to predict which participants will respond to Nemiralisib therapy, and to identify/quantify relationship(s) between different endpoints and response measures. Details of these analyses will be described in a separate RAP and results will be reported separately to the Clinical Study Report (CSR).

The following functions will be unblinded to interim analysis data: Clinical Statistics, Clinical Programming and Respiratory Data Sciences Group. Other member of GSK will be unblinded to group level summary data following the interim analyses (as documented internally).

#### 3.1.1. Futility analyses

At least one interim analysis for futility will be performed. The first analysis will occur at Interim Analysis 2, i.e. when 300 participants complete 84 days of treatment, or when approximately 400 participants remain to be randomised, whichever occurs first.

Futility will be assessed in a sequential manner.

- 1) Futility will first be assessed for the primary endpoint of change from baseline in FEV<sub>1</sub> at Day 84 by fitting a suitable dose response model, as described in Section 7.1.2.
- 2) If the posterior predictive probability of declaring success for this endpoint is low across all doses, then futility will be assessed for the rate of (on-treatment) exacerbations endpoint.
- 3) If the posterior predictive probability of declaring success for this endpoint is low, then the study may be stopped.

200879

Any decision to stop will be made after a review of all the data summarised/analysed at the time of the interim, including the proportion of participants achieving the EXACT-defined recovery.

#### 3.1.1.1. Futility rules

The decision rules for futility are defined as follows.

### Change from baseline in FEV<sub>1</sub> at Day 84

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, across all doses, where success at the end of the trial for change from baseline in FEV<sub>1</sub> is defined as demonstrating >90% posterior probability that the true difference from placebo for any dose of nemiralisib is greater than 0.

#### Rate of on-treatment exacerbations

Stop study for futility if the predictive probability of success at the end of the trial, given the data at the interim is <20%, where success at the end of the trial for rate of exacerbations is defined as demonstrating >80% posterior probability that the true rate reduction on 750 mcg dose versus placebo >0%.

If a different dose arm appears to be more efficacious than the 750 mcg arm, then futility may be assessed using the rate reduction for this arm versus placebo.

The pre-determined rules will act as guidelines for stopping the study for futility. All of the data summarised/analysed at the time of the interim will be reviewed prior to any decision to stop the study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

200879

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE)<br>Population | All participants who are screened for eligibility. | Study Population |
| Modified Intent<br>To treat (MITT)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment.</li> <li>Participants will be analyzed according to the treatment that they were randomised to.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Per Protocol (PP)<br>Population | <ul> <li>All randomized participants who receive at least one dose of study treatment, excluding any participants with an important protocol deviation.</li> <li>Participants will be analyzed according to the treatment that they were randomised to.</li> </ul> | Sensitivity analyses of efficacy |
| Safety Population | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>Participants will be summarised according to the treatment that they actually received. <ul> <li>If participants receive &gt;1 treatment, then they will be summarised according to the most frequently dosed treatment. In cases where the frequency is equal, the participant will be assigned the lowest dose strength of nemiralisib</li> </ul> </li> </ul> | Safety |
| Pharmacokinetic<br>(PK) Population | <ul> <li>All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values).</li> <li>Participants will be summarised according to the treatment that they actually received</li> </ul> | • PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

# 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

200879

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Randomization System Data Displays for Reporting | | Reporting | |
| Code | Description | Description | Order in TLF |
| Α | Placebo | Placebo | 1 |
| В | GSK2269557 12.5 mcg | NEMI 12.5 mcg | 2 |
| С | GSK2269557 25 mcg* | NEMI 25 mcg | 3 |
| D | GSK2269557 50 mcg | NEMI 50 mcg | 4 |
| Е | GSK2269557 100 mcg | NEMI 100 mcg | 5 |
| F | GSK2269557 250 mcg | NEMI 250 mcg | 6 |
| G | GSK2269557 500 mcg | NEMI 500 mcg | 7 |
| Н | GSK2269557 750 mcg | NEMI 750 mcg | 8 |

<sup>\*</sup> The nemiralisib dose of 25 mcg may be added following the results of an un-blinded interim analysis if further characterization of the lower end of the dose response curve is required.

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. NEMI 12.5 mcg vs Placebo
- 2. NEMI 25 mcg vs Placebo
- 3. NEMI 50 mcg vs Placebo
- 4. NEMI 100 mcg vs Placebo
- 5. NEMI 250 mcg vs Placebo
- 6. NEMI 500 mcg vs Placebo
- 7. NEMI 750 mcg vs Placebo

#### 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Baseline  $FEV_1$  is defined as  $FEV_1$  measured prior to the first dose of study treatment and post-bronchodilator on Day 1.

200879

Baseline CAT Total Score is defined as CAT Total Score measured prior to the first dose of study treatment on Day 1.

Baseline SGRQ Total Score is defined as SGRQ Total Score measured prior to the first dose of study treatment on Day 1.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

Prior to use in any statistical model, Baseline will be 'centred'. A centred baseline will be derived for each participant by subtracting the mean baseline across all participants from each participant's baseline value.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site and country.

# 5.4. Examination of Covariates and Subgroups

#### 5.4.1. Covariates

The list of covariates may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates of clinical interest may also be considered. The decision to include covariates in the model will be based on their impact on the model fit and will be detailed in the CSR.

Any continuous covariates will be 'centred' prior to use in statistical models. A centred covariate will be derived for each participant by subtracting the mean covariate across all participants from each participant's covariate value.

200879

| Covariate | Details |
|---|---|
| Index exacerbation severity | Categorical variable (Moderate or Severe), collected in eCRF. The stratification variable from the randomisation system may be used at the interim analyses if data in eCRF is sparse. |
| Age (at screening) | Continuous variable derived as described in Section 13.6.2.1 |
| ВМІ | Continuous variable derived using Height and Weight variables collected in eCRF: BMI = Weight (kg) / (Height (m)) <sup>2</sup> |
| Gender | Categorical variable (Male or Female), collected in eCRF |
| Country | Categorical variable |
| Smoking status | Categorical variable (Current or Former), collected in eCRF |
| Baseline COPD maintenance therapy type | Categorical variable derived depending on data observed |
| Index exacerbation type | Categorical variable: New or Relapse, derived using the question: "Other than the current prescription, for the index exacerbation, has the subject received oral/systemic corticosteroids and/or antibiotics for a COPD exacerbation within the last 7 days?" in the eCRF: New = No Relapse = Yes |
| Number of exacerbations in the previous 12 months | Categorical variable derived from "Total number of COPD exacerbations in the last 12 months" in the eCRF |

# 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Index exacerbation severity | Moderate vs. Severe |
| Baseline COPD maintenance therapy type | Possible categories of interest are: Monotherapy vs. Dual therapy vs. Triple therapy |
| Index exacerbation type | New vs. Relapse |
| Number of exacerbations in the previous 12 months | Possible categories of interest are: 0 vs. 1 vs. ≥2 |
| Gender | Male vs. Female |
| Smoking status | Current vs. Former |

200879

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 13.2 | Appendix 2: Assessment Windows |
| Section 13.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| Section 13.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 13.5 | Appendix 5: Derived and Transformed Data |
| Section 13.6 | Appendix 6: Reporting Standards for Missing Data |
| Section 13.7 | Appendix 7: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "APE" and/or "MITT" populations, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

#### 6.1.1. Concomitant medications

Concomitant medications will be summarised by treatment group. Separate summaries of Baseline and On-treatment (Step-up) COPD Maintenance Therapy, and duration of OCS use will also be presented.

Additional summaries or sensitivity analyses of on-treatment COPD maintenance therapy (step-up therapy) may be performed if the data indicate that further investigation is warranted.
200879

### 7. EFFICACY ANALYSES

Details of the outputs are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Details of Study Day calculations, including protocol-defined time windows, for use in the endpoint derivations below can be found in Section 13.2.

## 7.1. Primary Efficacy Analyses

## 7.1.1. Primary Endpoint

The primary endpoint of change from baseline in clinic visit trough FEV<sub>1</sub> at Day 84 measured post-bronchodilator is defined as:

FEV<sub>1</sub> measured prior to dosing and post-bronchodilator on Day 84 – Baseline FEV<sub>1</sub>

## 7.1.2. Primary Statistical Analyses

The primary endpoint will be analysed, by first intent, using a Bayesian 4-parameter  $E_{max}$  dose response model. Should the data not allow for a suitable model fit, then the following Bayesian models will be attempted in this sequential order: a 3-parameter  $E_{max}$  model and a Log-linear model.

The 4-parameter  $E_{max}$  dose response model will take the form:

Change from baseline FEV<sub>1</sub> = 
$$(E0 + a_1 * baseline) + \frac{(E_{max} + b_1 * baseline) * Dose^{\gamma}}{ED50^{\gamma} + Dose^{\gamma}}$$

Where: E0 =the response at dose = 0 (placebo)

 $E_{max}$  = the maximal response

ED50 =the dose that yields 50% of the maximal response

 $\gamma$  = the slope parameter

a<sub>1</sub>, b<sub>1</sub>, are covariates for explanatory parameters

Initially, normal non-informative priors will be used for the E0,  $a_1$ ,  $a_2$ , and  $E_{max}$  parameters with mean 0 and standard deviation 1E6 L. A functional uniform prior will be used for the ED50 and slope parameters (Bornkamp, 2014), where the prior density for the functional uniform prior is based on all the parameters in the model. An inverse - gamma prior with shape of 0.001 and scale of 0.001 will be used for the residual variance. However, if a prior distribution appears not to be truly non-informative then alternative prior distributions may be used.

Parameters will be blocked such that the MCMC procedure samples from E0,  $a_1$ ,  $b_1$ , and  $E_{max}$ , first, then the ED50 and slope parameters and then finally the residual variance

200879

parameter. For the functional uniform priors, the density will be calculated for values of dose from 0.0001 to 750 in steps of 50 (i.e. 0.0001, 50.0001, 100.0001,..., 750.0001). For the continuous covariates, the density will be calculated from the minimum to the maximum in 10 equal steps. For binary covariates the density will be calculated for values 0 and 1. If the model does not converge including covariates, the model may be fitted with covariates removed.

If the log-linear model is fitted an offset of 1 will be used.

The posterior median change from baseline with 95% Highest Posterior Density (HPD) Credible Intervals, will be presented for each dose along with the adjusted median difference from placebo with 95% HPD. Posterior probabilities that the true improvement is greater than 0 mL, 50 mL and 100 mL will also be presented. Graphical representation of the dose response across the full dose range will also be produced to allow inference to be made for the non-studied doses based upon the model fit.

#### For the futility analysis:

The predictive probability of success at the end of the study will be calculated for each dose using the formula suggested by Spiegelhalter et al., 2004 as follows:

Predictive probability (%) = 
$$\Phi\left[\frac{\sqrt{(m+n)}(my_m)}{\sqrt{mn}} + \sqrt{\frac{m}{n}}z_{0.9}\right]$$

Where m is the average number of subjects with Day 84 data in the placebo and dose arm of interest, n is the average number of subjects yet to be observed,  $y_m$  is the posterior mean difference from placebo from the fitted model,  $\sigma$  is the standard deviation of the posterior mean difference from placebo.

#### For the possible adaptations at Interim Analysis 2:

If the study is not deemed futile, and either the 4 parameter or 3 parameter  $E_{max}$  dose response curves has successfully been fitted to the data then adaptation of the randomisation schedule will be considered, to drop, add or amend doses from the randomisation scheme.

The adaptation will be done by comparing the relative information from alternative randomisation schemes with the original randomisation schemes, such to find the design that provides the most information about the dose response relationship. The efficiency ratio (ER) for an alternative scheme comparted to the original, will be calculated as:

$$ER(\theta_i) = \left(\frac{|M(\xi_i,\theta_i)|}{|M(\xi_i,\theta_i)|}\right)^{\frac{1}{p}}, i=1,...,1000$$

Where  $M(\xi, \theta)$  is the information matrix for the design  $\xi$  and model parameters  $\theta = (e0, emax, ed50, \gamma)^T$ ,  $\xi_1$  is the alternative design one and  $\xi_F$  is the fixed original design. In order to ensure any adaptation is robust to the variability in the parameter estimates at the interim analysis, 1000 samples will be generated from the posterior distribution of the parameters  $\theta_1, \dots, \theta_{1000}$  and the ER calculated for each set of

200879

parameter. Adaptation will then only take place if the median ER is >1.05 and the  $10^{th}$  percentile of the ER is >1.

### 7.1.2.1. Model Checking & Diagnostics

The following list of convergence diagnostics will be applied for each parameter:

- The Monte Carlo Standard Errors (MCSE) should be compared with the standard deviation of the posterior distribution (SD) to ensure that only a fraction of the posterior variability is due to the simulation. The number of samples generated and/or the thinning may be increased to reduce the ratio of the MCSE/SD as deemed necessary.
- The Geweke diagnostic test will be used to assess whether the mean estimates have converged by comparing means from the early and latter part of the Markov chain using a z-score t-test. Large absolute values of the z-score statistic indicate rejection of the null hypothesis of no difference between the mean estimates obtained from the early and latter parts of the chain.
- Trace plots of samples versus the simulation index will be visually inspected to
  assess some aspects of convergence. The centre of the chain should appear stable
  with very small fluctuations, i.e., the distribution of points should not change as
  the chain progresses and the posterior mean and variance are relatively constant.
- Autocorrelation plots will be visually inspected to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).

## 7.1.3. Sensitivity and Supportive Analyses

If there are greater than 20% of participants with an important protocol deviation that results in exclusion from the Per Protocol Population, the primary analysis may be repeated using the Per Protocol Population.

Change from baseline in clinic visit trough  $FEV_1$  at Day 84 will also be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant. All post-baseline scheduled visits will be included in the analysis using Day. Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

A further sensitivity analysis may be performed where Baseline  $FEV_1$  is replaced with the  $FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge for participants who were hospitalised for their index exacerbation, i.e. who were randomised with a Severe index exacerbation but kept as Baseline  $FEV_1$  for participants who were randomised with a Moderate index exacerbation

## 7.1.4. Subgroup Analyses

A subgroup analysis of change from baseline in clinic visit trough FEV<sub>1</sub> by index exacerbation severity will be performed by including the severity covariate term in the

200879

model, if possible. For the Bayesian 4-parameter  $E_{max}$  dose response model this would take the form:

Change from baseline  $FEV_1 =$ 

$$(E0 + a_1 * baseline + a_2 severity) + \frac{(E_{\max} + b_1 * baseline + b_2 * severity) * Dose^{\gamma}}{ED50^{\gamma} + Dose^{\gamma}}$$

Where  $a_1$ ,  $a_2$ ,  $b_1$ ,  $b_2$  are covariates for explanatory parameters.

If there are convergence issues, then the model for the primary endpoint may be fitted separately to each level of the subgroup.

A subgroup analysis of change from baseline in clinic visit trough  $FEV_1$  by index exacerbation severity will also be performed by including a treatment-by-severity-by-Day interaction term in the Bayesian Repeated Measures model.

## 7.2. Secondary Efficacy Analyses

### 7.2.1. Rate of exacerbations

Rate of exacerbation is defined as the frequency of exacerbations (subsequent to the index exacerbation) within the specified time period, for example, the 12-Week Treatment Period or the 24-Week Study Period.

The length of time on treatment or in study, depending on the specified time-period, for each participant will be calculated for each endpoint as follows:

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| Rate of (on-treatment) exacerbations, summarised by: • Moderate and severe exacerbations | 12-Week Treatment Period | Time from date of randomisation to date of last dose of study treatment |
| Moderate exacerbations | | |
| Severe exacerbations | | |
| All (mild, moderate and severe) exacerbations | | |
| Rate of (on-or off-treatment) exacerbations, summarised by: | 12-Week Treatment Period | Time from date of randomisation to Day 84. |
| Moderate and severe exacerbations | | For participants who withdraw early from the study: Time from |
| All exacerbations | | date of randomisation to date of study withdrawal |
| Rate of (off-treatment) exacerbations, summarised by: | 12-Week Follow Up Period | Time from date of last dose of study treatment to date of last |
| Moderate and severe exacerbations | | follow up assessment |
| Moderate exacerbations | | |

200879

| Endpoint | Time period | Length of time derivation |
|---|---|---|
| Severe exacerbations | | |
| Rate of (on- and off- treatment) exacerbations, summarised by: • Moderate and severe exacerbations | Full 24-Week Study Period | Time from date of randomisation to date of last follow up assessment |
| Moderate exacerbations | | |
| Severe exacerbations | | |

Refer to Section 13.5 for further details regarding the length of time derivation

## 7.2.1.1. Statistical analyses

The rate of exacerbations will be analysed using a Bayesian generalized linear model assuming a negative binomial distribution for the underlying exacerbation rate with a log link function. An offset to account for the length of time on treatment or in study, depending on the specified time-period, for each participant (as described above) will be included in the model as log<sub>e</sub> (length of time).

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The median exacerbation rates for each dose arm per 12 weeks, along with the median ratio in exacerbation rates (nemiralisib/placebo) per 12 weeks for each dose, will be estimated and corresponding 95% HPD credible intervals presented. The probability that the true exacerbation rate ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore estimates of the exacerbation rates for pooled data from 500 mcg plus 750 mcg will also be presented.

## 7.2.1.2. Subgroup analyses

A subgroup analysis of exacerbation rate by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

#### 7.2.1.3. Exploratory analyses

A summary of exacerbation rate by the following groups will be presented and, if feasible, a subgroup analyses may be performed:

- Index exacerbation type (New or Relapse)
- Number of exacerbations in previous 12 months  $(0, 1 \text{ or } \ge 2)$ .

200879

#### 7.2.2. Time to next exacerbation

Time to next (on-treatment) exacerbation following index exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation whilst on study treatment. Participants who did not have an exacerbation whilst on study treatment will be censored at the date of their last dose of study treatment.

Time to next (on-or off-treatment) exacerbation during the 12-Week Treatment Period is defined as time from the date of randomisation until the date of onset of the first exacerbation occurring up to Day 84. Participants who have not had an exacerbation during the 12-Week Treatment Period will be censored at Day 84 or the date of study withdrawal, for participants who withdrew from the study prior to Day 84.

Time to next exacerbation following cessation of study treatment is defined as time from the date of last dose of study treatment until the date of onset of the next exacerbation whilst off study treatment during the 12-Week Follow Up Period. Participants who have not had an exacerbation off-treatment will be censored at the date of their last follow up assessment.

Time to next exacerbation will be analysed by severity, as follows:

| Endpoint | Time period |
|---|---|
| Time to next (on-treatment) exacerbation, summarised by: | 12-Week Treatment Period |
| Moderate and severe exacerbations | |
| Moderate exacerbations | |
| Severe exacerbations | |
| All (mild, moderate and severe) exacerbations | |
| Time to next (on-or off-treatment) exacerbation, summarised by: | 12-Week Treatment Period |
| Moderate and severe exacerbations | |
| All exacerbations | |
| Time to next exacerbation following cessation of treatment, summarised by: | 12-Week Follow Up Period |
| Moderate and severe exacerbations | |
| Moderate exacerbations | |
| Severe exacerbations | |

Refer to Section 13.5 for further details regarding the length of time derivation

## 7.2.2.1. Statistical analyses

Time to next exacerbation will be analysed using a Bayesian Cox proportional hazards model with the "Efron" method for handling ties. Kaplan-Meier (KM) estimates of the probability of exacerbation will also be presented.

200879

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The hazard ratio and corresponding 95% HPD credible intervals for each nemiralisib dose versus placebo will be presented. The probability that the true hazard ratio is less than 1, in addition to other values appropriately selected based on the data, will be presented.

Based on pharmacological predictions, the 500 mcg and 750 mcg doses are expected to result in similar levels of target inhibition and thus potentially translate to similar clinical benefit, therefore an estimate of hazard ratio for pooled data from 500 mcg plus 750 mcg nemiralisib doses versus placebo will also be presented.

#### 7.2.2.2. Subgroup analyses

A subgroup analysis of time to exacerbation by Index exacerbation severity will be performed by including a treatment-by-severity term in the model.

## 7.2.3. Change from baseline in Clinic Visit trough FEV<sub>1</sub>

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56 measured post-bronchodilator is defined as:

FEV<sub>1</sub> measured prior to dosing and post-bronchodilator on Day X – Baseline FEV<sub>1</sub>

Where Day X is Day 14, 28, and 56.

Change from baseline in clinic visit trough FEV<sub>1</sub> at Day 14, 28, 56, 84 measured prebronchodilator is defined as:

FEV<sub>1</sub> measured prior to dosing and pre-bronchodilator on Day X – Baseline FEV<sub>1</sub>

Where Day X is Day 14, 28, 56, and 84.

#### 7.2.3.1. Statistical Analyses

Change from baseline in Clinic Visit trough FEV<sub>1</sub> will be analysed using a dose response model and repeated measures analysis as described for the primary endpoint in Section 7.1.2.

## 7.2.3.2. Subgroup analyses

A subgroup analysis of change from baseline in clinic visit trough  $FEV_1$  by index exacerbation severity will be performed.

### 7.2.4. Change from hospital discharge in clinic visit trough FEV<sub>1</sub>

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> will be derived only for participants who were hospitalised for their index exacerbation and who have been subsequently discharged.

200879

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day  $X - FEV_1$  measured post-bronchodilator and prior to dosing on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Change from hospital discharge in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day  $X - FEV_1$  measured prior to dosing and post-bronchodilator on day of hospital discharge.

Where Day X is 14, 28, 56 and 84.

Note, as per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the FEV<sub>1</sub> assessment will be assigned the hospital discharge assessment and the Day 14 assessment will be missing. Refer to Section 13.2.1.1 for further details.

In addition, if discharge takes place after Day 14, the Day 14 assessment will be missing for this analysis.

#### 7.2.4.1. Statistical analyses

Change from hospital discharge in clinic visit trough  $FEV_1$  will be analysed using a dose response model and repeated measures analysis as described for the primary endpoint in Section 7.1.2 if there are a sufficient number of participants to provide a meaningful analysis, otherwise the data will be summarised.

# 7.2.5. EXAcerbations of Chronic Pulmonary Disease Tool - Patient Reported Outcome (EXACT)

The EXACT is a 14-item daily diary designed to provide a measure of patient-reported symptoms of COPD exacerbation. An EXACT Total Score, ranging from 0 to 100, where higher scores indicate a more severe condition, will be derived for each day of diary collection according to the instructions in the EXACT User Manual (Version 8.0, Evidera, 2016).

The electronic EXACT diary does not allow a study patient to skip individual items, therefore no missing data are expected for individual items. However, if missing values occur for individual items, the Total Score that contains the item will be set to missing for that day. Moderate-to-severe COPD patients are expected to experience symptom(s) each day, and a score of zero on all 14 EXACT items is likely to represent a situation where in order to complete the diary quickly, the respondent did not accurately report their daily symptom(s), therefore if the EXACT Total Score is 0, it will be set to missing.

A 3-day Rolling Average EXACT Total Score will be calculated for each day, X, as:

200879

(EXACT Total Score on Day X-1 + EXACT Total Score on Day X + EXACT Total Score on Day X+1) / (Number of days with non-missing values)

Note, for Day 1, the Rolling Average EXACT Total Score will be calculated as the average of EXACT Total Score on Days 1 (Randomisation) and 2 only, since no EXACT data is collected prior to randomisation. Similarly, the Rolling Average EXACT Total Score for the last study day will be calculated as the average of EXACT Total Score on the last day and on the day before the last day.

The Rolling Average EXACT Total Score will be calculated for each day as long as at least 1 EXACT total score in the sequence is present. Therefore, only in the case where EXACT total scores are missing for 3 consecutive days in a row (or 2 consecutive days in the case of the first and last day rolling average calculation), will the rolling average score be missing.

The Maximum Observed Value (MOV) is defined as the highest Rolling Average EXACT Total Score observed within the first 14 days of randomisation. Note: this definition differs from the definition in the EXACT User Manual of "the highest rolling average EXACT score observed in the context of an EXACT exacerbation within the first 14 days of the exacerbation", since the date of the index exacerbation is likely to be prior to randomisation.

# 7.2.5.1. Proportion of participants achieving EXACT-defined recovery from index exacerbation

EXACT-defined recovery from the index exacerbation is defined as a decrease in the Rolling Average EXACT Total Score  $\geq 9$  points from the Maximum Observed Value, sustained for  $\geq 7$  days, with the first of the 7 days defined as the recovery day.

The proportion of participants achieving EXACT-defined recovery from the index exacerbation by Days 14, 28, 56, and 84 will be calculated as:

(Number of participants who experience an EXACT-defined recovery on or before Day X) / (Total number of participants in the MITT population)

Where Day X is 14, 28, 56, and 84.

#### 7.2.5.2. Time to EXACT-defined recovery from index exacerbation

Time to EXACT-defined recovery from index exacerbation is defined as time from the date of randomisation until date of the first EXACT-defined recovery day during the 12-Week Treatment Period, where EXACT-defined recovery is described in Section 7.2.5.1. Participants who did not experience EXACT-defined recovery during the 12-Week Treatment Period will be censored at the date of their last dose of study treatment.

# 7.2.5.3. Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT is defined as the highest EXACT Total Score (not using the 3-day Rolling Average) during the period

200879

from date of onset of the subsequent HCRU-exacerbation until date of EXACT-defined recovery of subsequent exacerbation.

Note, in this case, the Maximum Observed Value and EXACT-defined recovery are derived using the date of onset of the subsequent HCRU-exacerbation.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will only be derived for participants who have had a subsequent exacerbation. If a participant has more than one subsequent exacerbation, severity will be calculated for each subsequent exacerbation.

## 7.2.5.4. Statistical analyses

The proportion of participants achieving EXACT-defined recovery from the index exacerbation will be analysed using a Bayesian logistic regression model. Separate models will be fitted for each time-point.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.

The results of the analysis will be presented in terms of odds ratios together with its associated 95% HPD credible interval. The probability that the true odds ratio is greater than 1, in addition to other values appropriately selected based on the data, will be presented.

Time to EXACT-defined recovery from index exacerbation will be analysed using the same techniques as described in Section 7.2.2.1.

Severity of subsequent HCRU-defined exacerbation(s) defined by EXACT will be summarised for each treatment group and reported by study period. The severity of subsequent HCRU-defined exacerbation(s) occurring whilst a participant is on treatment will be reported as during the 12-Week Treatment Period and the severity of subsequent HCRU-defined exacerbation(s) occurring after the last dose of study treatment will be reported as during the 12-Week Follow-up Period.

## 7.2.5.5. Subgroup analyses

A subgroup analysis of the proportion of participants achieving EXACT-defined recovery from the index exacerbation by Index Exacerbation Severity will be performed by including a treatment-by-severity term in the model.

### 7.2.5.6. Sensitivity and supportive analyses

Sensitivity analyses exploring the impact of any missing data, and changes to the definition of EXACT-defined recovery may be conducted and may be performed post-SAC.

200879

### 7.2.6. COPD Assessment Test (CAT)

The COPD Assessment Test (CAT) is a patient completed questionnaire developed to measure the health status of patients with COPD. The CAT consists of eight items, each on a six-point scale: 0 (no impact) to 5 (high impact). The CAT Score will be calculated for each study day of collection by summing the scores for all questions. The CAT Score ranges from 0 to 40, where higher scores indicate a more severe condition.

## 7.2.6.1. Proportion of responders using the CAT

The proportion of responders using the CAT will only be derived for participants with a baseline CAT Total Score  $\geq 2$ .

The Proportion of responders using the CAT is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq$ 2 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84, and the study day following EXACT-defined recovery from the index exacerbation.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

## **Exploratory – Follow-Up Period**

The Proportion of responders using the CAT at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in CAT Total Score  $\geq$ 2 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is FU Day 28 and FU Day 56, as defined in Section 13.2.1, and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

#### 7.2.6.2. Change from baseline in CAT Total Score

Change from baseline in CAT Total Score is defined as:

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is 28, 56, 84, and the study day following EXACT defined recovery from the index exacerbation.

Note: due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery is not derived according to the EXACT User Manual, see Section 13.2.1.2 for further details.

200879

## **Exploratory – Follow-Up Period**

The Change from baseline in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – Baseline CAT Total Score

Where Day X is FU Day 28 and FU Day 84, as defined in Section 13.2.1.

The Change from end of treatment in CAT Total Score at Day 112 and 168 is defined as:

CAT Total Score on Day X – CAT Total Score on Day 84

Where Day X is FU Day 28 and FU Day 84, as defined in Section 13.2.1.

## 7.2.6.3. Statistical analyses

The proportion of responders using CAT will be analysed using the same techniques as described in Section 7.2.5.4.

Change from baseline in CAT Total Score will be compared between treatment groups using a Bayesian Repeated Measures analysis with covariates for baseline-by-Day interaction and treatment-by-Day interaction. Day will be fitted as a repeated effect within each participant.

All post-baseline scheduled visits will be included in the analysis using Day.

Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised. An unstructured covariance matrix will be used to model the within-subject error.

Adjusted posterior median change from baseline and corresponding 95% HPD credible intervals will be summarised for each treatment by time-point, together with estimated treatment differences (GSK – Placebo) and corresponding 95% HPD credible intervals. The posterior probability that the true treatment difference is less than 0, in addition to other values appropriately selected based on the data, will also be presented.

## 7.2.6.4. Subgroup analyses

A subgroup analysis of the proportion of responders using CAT and the change from baseline in CAT Total Score by Index exacerbation severity will be performed by including a treatment-by-severity term and a treatment-by-severity-by-Day term in the Bayesian logistic regression and Bayesian Repeated Measures models, respectively.

# 7.2.7. St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C)

St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) is a 40-item questionnaire designed specifically to focus on COPD patients. SGRQ-C will be scored to be equivalent to the SGRQ Total Score, ranging from 0 to 100, where higher scores reflect worse health-related quality of life. SGRQ Total Scores will be calculated for each

200879

day of collection according to the instructions in SGRQ-C Manual (Version 1.3, March 2016).

### 7.2.7.1. Proportion of responders on the SGRQ Total Score

The proportion of responders on the SGRQ Total Score will only be derived for participants with a baseline SGRQ Total Score  $\geq$ 4.

Proportion of responders on the SGRQ Total Score is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is 28, 56, and 84.

## **Exploratory – Follow-Up Period**

The Proportion of responders on the SGRQ Total Score at Day 112 and 168 is defined as:

(Number of participants with a decrease from baseline in SGRQ Total Score  $\geq$ 4 on or before Day X)/(Total number of participants in the MITT population)

Where Day X is FU Day 28 and FU Day 84, as defined in Section 13.2.1 and the study day following EXACT defined recovery, if it occurs during the Follow-up period.

#### 7.2.7.2. Change from baseline in SGRQ Total Score

Change from baseline in SGRQ Total Score is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is Day 28, 56, and 84.

### Exploratory - Follow-Up Period

The Change from baseline in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – Baseline SGRQ Total Score

Where Day X is FU Day 28 and FU Day 84, as defined in Section 13.2.1.

The Change from end of treatment in SGRQ Total Score at Day 112 and 168 is defined as:

SGRQ Total Score on Day X – SGRQ Total Score on Day 84

Where Day X is FU Day 28 and FU Day 84, as defined in Section 13.2.1.

200879

#### 7.2.7.3. Statistical analyses

Change from baseline in SGRQ Total Score and the proportion of responders on the SGRQ Total Score will be analysed using the same techniques as described in Section 7.2.6.3.

#### 7.2.7.4. Subgroup analyses

Subgroup analyses of change from baseline in SGRQ Total Score and the proportion of responders on the SGRQ Total Score by Index exacerbation severity will be conducted as described in Section 7.2.6.4.

#### 7.2.8. Rescue medication use

All participants will record rescue medication use in the eDiary. Rescue medication use will be recorded as the number of occasions of rescue medication use each day.

The Mean Number of (on-treatment) Occasions of Rescue Medication Use Per Day is defined as:

(Sum of the number of occasions of rescue medication use each day within the time-period) / (Total number of days with non-missing values within the time-period)

The Percentage of (on-treatment) Rescue-Free Days is defined as:

(Sum of the number of days where the number of occasions of rescue medication use is zero within the time-period) / (Total number of days with non-missing values within the time-period)\*100

Where the time-period is defined as follows:

Week 1 of the 12-Week Treatment Period: Day 1 to Day 7

Week 2 of the 12-Week Treatment Period: Day 8 to Day 14

Week 3 of the 12-Week Treatment Period: Day 15 to Day 21

Week 4 of the 12-Week Treatment Period: Day 22 to Day 28

Week 5 of the 12-Week Treatment Period: Day 29 to Day 35

Week 6 of the 12-Week Treatment Period: Day 36 to Day 42

Week 7 of the 12-Week Treatment Period: Day 43 to Day 49

Week 8 of the 12-Week Treatment Period: Day 50 to Day 56

Week 9 of the 12-Week Treatment Period: Day 57 to Day 63

Week 10 of the 12-Week Treatment Period: Day 64 to Day 70

200879

Week 11 of the 12-Week Treatment Period: Day 71 to Day 77

Week 12 of the 12-Week Treatment Period: Day 78 to Day of last dose

Over the 12-Week Treatment Period: Day 1 to Day of last dose.

#### Exploratory - Follow-Up Period

Rescue medication use up to Day 112 will also be summarised by including the time-periods:

Week 13 (Follow-up Period): (Day of last dose + 1) to (Day of last dose + 1) + 6 days

Week 14 (Follow-up Period): (Day of last dose + 7) to (Day of last dose + 1) + 13 days

Week 15 (Follow-up Period): (Day of last dose + 14) to (Day of last dose + 1) + 20 days

Week 16 (Follow-up Period): (Day of last dose + 21) to (Day of last dose + 1) + 27 days

For a subject to be counted in the time periods for rescue medication use, they must have at least one eDiary entry recorded during that time period.

## 7.2.8.1. Rescue medication use via the clip-on Propeller Sensor for MDI

A subset of participants from countries where the Propeller Sensor for MDI is available will also record rescue medication use via the clip-on Propeller Sensor for MDI. A supportive summary of rescue medication use via the clip-on Propeller Sensor for MDI for these participants will be presented.

Rescue medication use via the clip-on Propeller Sensor for MDI is defined in the same way as rescue medication use via the eDiary, except that the number of actuations will be used instead of the number of occasions in accordance with the way the data is captured.

#### 7.2.8.2. Statistical analyses

The Mean Number of (on-treatment) Occasions of Rescue Medication Use Per Day will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

The Percentage of (on-treatment) Rescue-Free Days will be summarised between each treatment group using means, standard deviations, medians, minimum and maximum.

The Percentage of Participants Taking (on-treatment) Rescue Medication By Day for each treatment group will also be presented.

Rescue medication use via the clip-on Propeller Sensor for MDI will be summarised in the same way as rescue medication use via the eDiary.

200879

## 7.3. Exploratory Efficacy Analyses

## 7.3.1. Change from Day 84 in Clinic Visit trough FEV<sub>1</sub>

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured post-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and post-bronchodilator on Day X – Day 84 post-bronchodilator  $FEV_1$ 

Where Day X is FU Day 28, FU Day 56 and FU Day 84, as defined in Section 13.2.1.

Change from Day 84 in clinic visit trough FEV<sub>1</sub> measured pre-bronchodilator is defined as:

 $FEV_1$  measured prior to dosing and pre-bronchodilator on Day X – Day 84 post-bronchodilator  $FEV_1$ 

Where Day X is FU Day 28, FU Day 56 and FU Day 84, as defined in Section 13.2.1.

Participants who discontinue study treatment prior to Day 84 will be excluded from this analysis.

## 7.3.1.1. Statistical analysis

Change from Day 84 in Clinic Visit trough FEV<sub>1</sub> will be analysed using the same techniques as described for Change from baseline in CAT Total Score in Section 7.2.6.3.

A subgroup analysis of change from Day 84 in FEV<sub>1</sub> will be performed by including a treatment-by-severity-by-Day term in the Bayesian Repeated Measures model.

### 7.3.2. E-RS:COPD (Evaluating Respiratory Symptoms in COPD)

Change from baseline in E-RS: COPD and subscales will be summarised by treatment group. Exploratory analyses related to E-RS: COPD and subscales may be performed post SAC.

#### 7.3.3. Measures of HCRU related to exacerbations

Unscheduled Healthcare Utilisation will be summarised separately for exacerbation-related, COPD-related or non-COPD related; each summary will be presented by all patients (i.e. moderate and severe index exacerbation combined), and separately by index exacerbation severity.

The number of days of hospital admission for the index and subsequent exacerbations will also be summarised by treatment group.

200879

#### 7.3.3.1. Re-hospitalisation within 30 days of index exacerbation

Re-hospitalisation within 30 days of index exacerbation is defined as 30 days from the date of hospital discharge until the date of next hospital admission (+ 1 day, to account for study day derivation), for participants who were hospitalised for their index exacerbation.

Exacerbation-related, COPD-related and Non-COPD-related hospital admissions are collected in separate eCRFs. The date of hospital admission is not collected in the COPD-related eCRF, therefore the date of next hospital admission will be estimated using the earliest of:

- Date of hospital admission for exacerbation-related hospitalisations
- Date of contact for COPD-related hospitalisations, where the number of inpatient hospitalisation days >0
- Date of hospital admission for non-COPD-related hospitalisations.

The proportion of participants who were re-hospitalised within 30 days of the index exacerbation will be summarised by each treatment arm.

#### 7.3.3.2. Time from resolution of index exacerbation to next exacerbation

Time from resolution of index exacerbation to next exacerbation is defined as time from the date of (Investigator-defined) resolution of index exacerbation until the date of onset of the subsequent exacerbation.

A summary of time from resolution of index exacerbation to next exacerbation will be presented. Participants who did not have a subsequent exacerbation or for whom the index exacerbation was not resolved will be excluded from the summary.

Time from resolution of index exacerbation to next exacerbation will only be derived for the first subsequent exacerbation following the index exacerbation.

### 7.3.3.3. Subsequent exacerbation treatment type

A summary of the type of treatment for subsequent exacerbations (OCS, antibiotics, or both) may also be presented.

## 7.3.4. Compliance

Reported compliance for all participants is captured daily in the eDiary from the question "Did you take this morning's dose of study medication"?

Percentage compliance for each participant is calculated as:

(Sum of the number of days where the question was answered with 'Y') / (Number of days from first dose of study treatment to last dose of study treatment)  $\times$  100

Overall percentage compliance will be summarised by each treatment group.

200879

# 7.3.4.1. Number of actuations of double-blind study treatment measured by the clip-on Propeller Sensor

Percentage compliance via the clip-on Propeller Sensor for ELLIPTA in the subset of participants from countries where the Propeller Sensor for ELLIPTA is available is calculated as:

(Sum of the total number of actuations) / (Number of days from first dose of study treatment to last dose of study treatment) x 100

Overall percentage compliance will be summarised by each treatment group.

# 7.3.5. Inflammatory/infective markers in blood and sputum in relation to acute exacerbation of COPD

Results of the analysis of blood/spontaneous sputum samples of eosinophil counts and inflammatory/infective mediators/markers will be summarised by treatment group.

Further analyses of inflammatory/infective markers may be performed, for example split by CRP high, CRP low, Procalcitonin high, etc. categories.

### 7.3.6. Other spirometry measurements

Percent predicted FEV<sub>1</sub>, Forced Vital Capacity (FVC), percent predicted FVC and FEV/FVC ratio will be summarised by treatment group.

### 7.3.7. Other PRO symptoms suggestive of exacerbation

Responses to questions related to PRO symptoms of sputum purulence (colour), fever, sore throat, wheezing and colds collected in the eDiary will be listed by treatment group.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. The details of the planned displays will be provided in Appendix 11: List of Data Displays.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards.

#### 8.1.1. Adverse Events of Special Interest

#### 8.1.1.1. Post-inhalation Cough Immediately Following Dosing

Post-inhalation cough immediately following dosing is an Adverse Event of Special Interest (AESI).

200879

Post-inhalation cough immediately following dosing will be evaluated during study Visits 2-6 in the 12-Week Double-Blind Treatment Period. Investigators (or medically qualified designees) will monitor participants for potential study treatment tolerability issues, including post-inhalation cough, within 5 minutes immediately following dosing.

The percentage of patients experiencing post-inhalation cough following dosing, regardless of whether it was also reported as an AE, overall and by each visit will be summarised for each treatment group. The type of cough, time to onset and duration of cough, and severity will also be summarised.

In addition, any post-inhalation cough immediately following dosing reported as an adverse event during the clinic visit observation or during the course of the study will be summarised by treatment group.

## 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and liver function tests will be based on GSK Core Data Standards.

## 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

## 8.4. Mortality

A summary of all-cause mortality by treatment will be presented.

## 9. PHARMACOKINETIC ANALYSES

## 9.1. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 9.2. Drug Concentration Measures

Plasma nemiralisib concentrations of GSK2269557 will be listed and summarised by dose, day and time. Drug levels will be summarised by day (14, 28), dose and time intervals (trough, 0-<1h, 1-6h).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 13.4.3 Reporting Standards for Pharmacokinetic).

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

200879

### 10. POPULATION PK ANALYSIS

A dataset for population PK analysis will be provided by Statistics and Programming based on the NONMEM data specifications in Section 13.8.2.

Conduct of the population PK analyses will be based on the current guidance which contains specific recommendations for working practices, processes and standards for population PK and PK/PD analysis conducted by Clinical Pharmacology Modelling and Simulation (CPMS) [Analysis & Reporting, 2017].

The sparse PK samples will be subjected to a validated population PK model for nemiralisib currently under development.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR. Analyses and reporting of the population PK model will be in accordance with the FDA and EMEA guidance on population PK, PK-PD analyses.

#### 10.1. Derived Pharmacokinetic Parameters

The exposure parameters (e.g. AUC,  $C_{max}$ ) will be derived from the individual post-hoc estimates from the POP PK model. These will be summarized across dose treatments, subgroups (e.g., gender, race) or as a function of a continuous variable (e.g., age).

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

If statistical analyses suggest an effect of nemiralisib on primary and other key clinical endpoints, an integrated longitudinal population dose/exposure versus clinical response on analysis key parameters including  $FEV_1$  and exacerbation rate will be undertaken. Participant characteristics influencing the relationship will be evaluated.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

200879

## 12. REFERENCES

Bornkamp, B. (2014). Practical considerations for using functional uniform prior distributions for dose-response estimation in clinical trials. Biometrical Journal, 56(6), 947-962. doi: 10.1002/bimj.201300138

Evidera. (2016). The Exacerbations of Chronic Pulmonary Disease Tool (EXACT®) Patient-Reported Outcome (PRO) USER MANUAL (Version 8.0).

Spiegelhalter, D.J., Abrams, K.R. & Myles, J.P., (2004). Bayesian Approaches to Clinical Trials and Health-Care Evaluation. John Wiley & Sons, Ltd.

200879

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 13.1.1. Exclusions from Per Protocol Population

Protocol deviations will be reviewed regularly throughout the course of the study, as described in Protocol Deviation Management Plan (PDMP). Deviations which will result in exclusion from the Per Protocol population will be assigned on a case-by-case basis prior to database freeze (DBF).

Decisions on whether or not the subject should be excluded from the PP population because the incorrect treatment was taken, due to the incorrect container being dispensed, will be identified after unblinding (i.e. post DBF). A PD of "incorrect treatment" will be added to the reporting dataset.

200879

## 13.2. Appendix 2: Assessment Windows

### 13.2.1. Definitions of Assessment Windows for Analyses

The target Study Day and Analysis Timepoint for summaries and analyses for participants who do not discontinue treatment prior to the Day 84 (+window) is shown in the table below:

| Target | Analysis Window | | Analysis Timepoint |
|---------------|---------------------|------------------|--------------------|
| | Beginning Timepoint | Ending Timepoint | |
| Study Day 1 | Day 1 | Day 1 | DAY 1 |
| Study Day 14 | Day 11 | Day 17 | DAY 14 |
| Study Day 28 | Day 25 | Day 31 | DAY 28 |
| Study Day 56 | Day 52 | Day 59 | DAY 56 |
| Study Day 84 | Day 80 | Day 87 | DAY 84 |
| Study Day 112 | Day 108 | Day 115 | FU DAY 28 |
| Study Day 140 | Day 136 | Day 143 | FU DAY 56 |
| Study Day 168 | Day 164 | Day 171 | FU DAY 84 |

FU = Follow Up

For participants who discontinue treatment prior to Day 84 (+window), a follow-up (FU) Study Day will be derived as:

FU Study Day = (Date of follow-up assessment – Date of last dose of study treatment) +1

The FU Study Day will then be used to assign Study Days and Analysis Timepoints for summaries and analyses as shown in the table below:

| Derived follow-up (FU) | Analysis Window | | Analysis Timepoint |
|---|---|---|---|
| Study day | Beginning Timepoint | Ending Timepoint | |
| FU Study Day 28 | FU Study Day 24 | FU Study Day 31 | FU DAY 28 |
| FU Study Day 56 | FU Study Day 52 | FU Study Day 59 | FU DAY 56 |
| FU Study Day 84 | FU Study Day 80 | FU Study Day 87 | FU DAY 84 |

#### 13.2.1.1. Hospital discharge

For the change from hospital discharge in clinic visit trough  $FEV_1$  endpoint, the assessment on the day of hospital discharge can be derived using the date of hospital discharge for the index exacerbation from the eCRF. As per Section 5.1 of the Protocol, if discharge takes place between Day 11 and Day 17 (inclusive), the assessments planned for Day 14 may be completed on the day of discharge. In these cases, for this endpoint only, the  $FEV_1$  assessment will be assigned the hospital discharge  $FEV_1$  assessment and the Day 14 assessment will be missing.

200879

For all other analyses and summaries that include participants who were hospitalised for their index exacerbation, an additional Analysis Timepoint of "HOSPTIAL DISCHARGE" will be derived. However, in the cases where discharge takes place between Day 11 and Day 17 (inclusive), participants will be summarised under DAY 14 and a footnote to say that participants who were discharged at Day 14 are summarised under DAY 14 will be included.

## 13.2.1.2. EXACT-Defined Recovery for CAT Trigger

Due to software limitations of the electronic PRO device, the study day following EXACT-defined recovery from the index exacerbation is not derived according to the EXACT User Manual. Instead, it has been derived using a 3-day Rolling Average that is calculated as the mean EXACT score [Day  $_{\text{X-2}}$ , Day  $_{\text{X-1}}$ , Day  $_{\text{X}}$ ] .

200879

# 13.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

### 13.3.1. Study Periods

#### 13.3.1.1. 12-Week Treatment Period

The 12-Week Treatment Period is assigned from Study Day 1 to Study Day 84.

## 13.3.1.2. 12-Week Follow-Up Period

The 12-Week Follow-up Period is assigned from Study Day 85 to Study Day 168.

Refer to Section 13.2.1 for details on how Study Days and Analysis Timepoints will be derived for participants who discontinue treatment prior to Day 84.

## 13.3.2. Study Phases

Exacerbation events during the 12-Week Treatment Period will be classified according to their occurrence from randomisation until treatment discontinuation/study withdrawal days, as detailed below.

| Study Phase | Occurring from randomisation until |
|---|---|
| On-Treatment during the 12-Week Treatment Period | Treatment Stop Day |
| On- or Off-Treatment during the 12-Week Treatment | Day 84 or Study Withdrawal Day if Treatment Stop |
| Period | Day is < Day 84 |

#### 13.3.2.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before Randomisation Date |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 13.3.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop |
| Emergent | date plus 10 days. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

200879

# 13.4. Appendix 4: Data Display Standards & Handling Conventions

#### 13.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | : \arprod\gsk2269557\mid200879 |
| Analysis Datasets | |
| <ul> <li>For all interim analyses, except for the End of Treatment Interim Analysis, datasets will be created<br/>according to Legacy GSK A&amp;R dataset standards.</li> </ul> | |
| <ul> <li>For the End of Treatment Interim Analysis and the final reporting effort, datasets will be created<br/>according to current CDISC standards</li> </ul> | |

### **Generation of RTF Files**

RTF files will be generated for the final reporting effort.

## 13.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless
  otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
  - Figures will be produced using PROC SGPLOT in SAS

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

200879

| Unscheduled Visits | Unscheduled Visits |
|---|---|
| <ul> <li>Unscheduled visits will be included in summary tables of the worst-case results by potential clinical<br/>importance criteria only.</li> </ul> | |
| All unscheduled vi | sits will be included in listings. |
| <b>Descriptive Summary</b> | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

# 13.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive Summary Statistics, Graphical | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 13.8.2 Population Pharmacokinetic (PopPK) Dataset Specification. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in the CPMS RAP. |

200879

## 13.5. Appendix 5: Derived and Transformed Data

#### 13.5.1. General

## Multiple Measurements at One Analysis Time Point

- If there are two values within a time window (as per Section 13.2.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety
  parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of
  related summary tables. This will also be applicable to relevant Potential Clinical Importance summary
  tables.

### **Study Day**

- Calculated as the number of days from Randomisation Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### Time from date of randomisation and time from date of last dose of study treatment

- For endpoints that use the time from the date of randomisation to a reference date, time will be calculated as
  - (Ref Date Randomisation Date) + 1
- For endpoints that use the time from the date of last dose of study treatment to a reference date, time will be calculated as
  - (Ref Date (Last Dose Date + 1)) +1

#### 13.5.2. Study Population

### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

The cumulative dose will be based on the formula:

Cumulative Dose = Sum of (Number of Days x Total Daily Dose)

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 13.5.3. Safety

### **Adverse Events**

## **AE'S of Special Interest**

 Post-inhalation cough is an AE of special interest. The lower level term (LLT) to be included is "coughing after drug inhalation"

200879

## 13.6. Appendix 6: Reporting Standards for Missing Data

## 13.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) is defined as completing all phases of the study including the last scheduled study visit |
| | A participant is considered to have completed the Treatment Period, if he/she has completed the last on-treatment study visit (Visit 6) |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 2: Assessment Windows otherwise they will not be summarised (and will be listed only). |

# 13.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 13.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events. |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> <li>Consequently, time to onset and duration of such events will be missing.</li> </ul> |

200879

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Age | <ul> <li>The eCRF collects year of birth only. Day and Month will be imputed by Data Management using a PP for the day and PPD for the month</li> <li>Age will then be derived referenced to the Screening Date</li> <li>A footnote to say that age has been imputed will be included in any outputs containing age.</li> </ul> |

200879

# 13.7. Appendix 7: Values of Potential Clinical Importance

# 13.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | G/DL | Male 18-64 years | 7.1 | 19.9 |
| Lloomodobio | | Male 65+ years | 7.1 | 19.9 |
| Haemoglobin | | Female 18-64 years | 7.1 | 19.9 |
| | | Female 65+ years | 7.1 | 19.9 |
| Lymphocytes | GI/L | | 0.85 | 4.1 |
| Total Absolute Neutrophil Count | GI/L | | 1.5 | 8 |
| Platelet Count | GI/L | | 31 | 1499 |
| White Blood Cell sount | GI/L | 18-64 years | 1.1 | 10.8 |
| White Blood Cell count | | 65+ years | 1.1 | 10.8 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 32 | 50 |
| Calcium | mmol/L | | 1.5 | 3.24 |
| | | Male 40-49 years | 69 | 160 |
| | | Male 50-59 years | 67.2 | 160 |
| | | Male 60-69 years | 67.2 | 160 |
| Creatinine | | Male 70+ years | 59.2 | 160 |
| Creatinine | | Female 40-49 years | 52.2 | 160 |
| | | Female 50-59 years | 53 | 160 |
| | | Female 60-69 years | 53 | 160 |
| | | Female 70+ years | 55.7 | 160 |
| | mmol/L | 13-49 years | 2.2 | 27.8 |
| Glucose | IIIIIOI/L | 50+ years | 2.2 | 27.8 |
| Potassium | mmol/L | | 2.8 | 6.5 |
| Sodium | mmol/L | | 120 | 160 |
| | | 13-64 years | 2.5 | 15 |
| Urea/BUN | mmol/L | 65+ years | 2.5 | 15 |

200879

| Liver Function | | | |
|--------------------|--------|----------|----------------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 2x ULN |
| | µmol/L | | 2xULN T.Bilirubin + ≥ 3x ULN ALT |
| T. Bilirubin + ALT | | High | |
| | U/L | | |
| Direct Bilirubin | µmol/L | | 0 – 6 |

## 13.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 530 |
| Absolute PR Interval | msec | < 110 | > 240 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 13.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 90 | > 140 |
| Diastolic Blood Pressure | mmHg | < 60 | > 90 |
| Heart Rate | bpm | < 40 | > 110 |

200879

## 13.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

## 13.8.1. Population Pharmacokinetic (PopPK) Methodology

All analysis will be performed in the validated Modelling and Analysis Platform (MAP). MAP consists of a Linux desktop containing various modelling applications, including NONMEM, PsN, Pirana, R and RStudio. All software versions used will be documented.

The population PK analysis will be performed in the following sequence of steps:

- 1. Exploratory data analysis/data check out.
- 2. Base structural model development.
- 3. Covariate analysis.
- 4. Model refinement.
- 5. Model evaluation.
- 6. Model application using simulation

The above analysis and reporting steps follow EMEA (http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC500003067.pdf) and FDA population PK guidances (https://www.fda.gov/downloads/drugs/guidances/UCM072137.pdf)

Key components of these regulatory guidelines on population PK are also included in the Global CPMS guidance for pop pk RAP (https://connect.gsk.com/sites/cpms/TandD/Guidances).

#### 13.8.2. Population Pharmacokinetic (PopPK) Dataset Specification

Statistics & Programming, in discussion with CPMS, will provide a NONMEM dataset.

Column headings in NONMEM-ready datasets and specifications should be consistent to minimise the programming process, and facilitate a smooth transfer of projects between users as needed. IDSL standards will be followed where possible.

A list of most common standardised variable names for NONMEM datasets can be found in Table below.

200879

## List of Variable Names for NONMEM-Ready Datasets for PopPK Analysis

| Variable | Label (Variable description) |
|---|---|
| С | NONMEM line exclusion identifier |
| ID | NONMEM subject identifier |
| STUD | Study ID |
| SUBJID | Subject identifier for study |
| SITEID | Unique identifier for a study site |
| AMT | NONMEM Amount of drug administered then EVID =1- dose event record |
| UAMT | Unit of AMT (mg) |
| ADDL | NONMEM Additional dose |
| CONC | Drug Concentration |
| UCONC | Unit of CONC (ng/mL) |
| LNCONC | Natural log of CONC column |
| ANALYTE | Drug label e.g 557 |
| LLQ | Lower Limit of quantification |
| LNLLQ | Natural log of LLQ column |
| DAY | Study day number of record or of dosing |
| TIME | Plasma sample time after last dose |
| UTIME | Unit of TIME (h) |
| DOSE | Dose amount |
| EVID | NONMEM Event ID If row has dose then EVID=1 else EVID=0 |
| | If EVID=1 then this is a dose event record |
| | If EVID = 0 then this is an observation record |
| II | NONMEM Inter-dose interval II=24 – dose every day |
| SS | Steady state item SS= 1 refers to steady state |
| MDV | NONMEM Missing data value then MDV=1 else MDV=0 |
| AGE | Subject Age (yrs) |
| SEX | Subject gender 0 = Male 1 =Female |
| SEXTEXT | Subject gender text Male or Female |
| BMI | Baseline Body Mass Index |
| WT | Baseline Subject weight |
| CONMED1 | Identifier for inhibitor CYP3A4 1 =Yes, 0 = No |
| CONMED1TXT | Inhibitor Name |
| CONMED2 | Identifier for inducer CYP3A4 1 =Yes, 0 = No |
| CONMED2TXT | Inducer Name |
| <u> </u> | 0010 "141" "1011 10010 1 "1 |

If observation record e.g CONC has "NA" or "NS" then assign CONC cell as "."

If observation record e.g CONC has "NQ" or "BQL" then assign CONC cell as "." and MDV = 1 -this means value can be estimated by model

Missing covariate data should be imputed as "-99.

200879

## 13.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

## 13.9.1. Pharmacokinetic/Pharmacodynamic Methodology

PK-PD analysis of Nemiralisib will be guided by the results of the formal statistical analyses on the key clinical endpoints. The aims of the PK-PD analyses will contribute towards the dose selection in future studies using an integrated longitudinal analysis framework.

The objective is to explore an integrated modelling framework to characterise the longitudinal FEV1 response versus dose (average systemic exposure) during on- & off-treatment phases

$$FEV1_i(t_{ij}) = FEV1_{i,base} \cdot (1 + f(t_{ij}, dose_i, x_i) + \varepsilon_{ij} \text{ with } \varepsilon_{ij} \sim N(0, \sigma^2)$$

A longitudinal nonlinear mixed-effects model will be used to describe the FEV1 response over time measured for each patient (i) at each visit (tij) with  $\varepsilon$  denoting the normal distributed residual variability with mean 0 and variance  $\sigma$ 2. The function f() describes the relative change from observed FEV1 at baseline (FEV1,<sub>base</sub>) and any influence of patient characteristics on FEV1 response will be assessed.

Joint relationship between time to first exacerbation and FEV1 change as function of dose/exposure and patient covariates will be assessed.

Details of these analyses will be described in a separate CPMS RAP and results will be reported separately to the CSR.

200879

# 13.10. Appendix 10: Abbreviations & Trade Marks

## 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |
200879

### 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| COPD Assessment Test (CAT) |
| ELLIPTA |
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| E-RS: COPD |
| EXACT-PRO |
| NONMEM |
| Propeller Sensor |
| SAS |
| SGRQ |

200879

## 13.11. Appendix 11: List of Data Displays

### 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays for SAC:

| Section | Tables | Figures |
|------------------|--------------|----------------|
| Study Population | 1.1 to 1.28 | Not applicable |
| Efficacy | 2.1 to 2.121 | 2.1 to 2.12 |
| Safety | 3.1 to 3.31 | 3.1 to 3.3 |
| Pharmacokinetic | 4.1 to 4.2 | Not applicable |
| Section | Lis | tings |
| ICH Listings | 1 to 27 | |
| Other Listings | 28 | to 30 |

## 13.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

#### 13.11.3. Deliverables

| Delivery | Description |
|---|---|
| IA | Interim Analyses (except the End of treatment Phase Interim Analysis) |
| EOT | End of Treatment Phase Interim Analysis |
| SAC Statistical Analysis Complete | |

200879

## 13.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | · |
| 1.1. | MITT | ES8 | Summary of Subject Status and Reason for Study Withdrawal | | EOT, SAC |
| 1.2. | MITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | EOT, SAC |
| 1.3. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| 1.4. | APE | NS1 | Summary of Number of Participants by Country and Site ID | | SAC |
| Protoc | ol Deviation | | | | <u> </u> |
| 1.5. | MITT | DV1 | Summary of Important Protocol Deviations | | EOT, SAC |
| 1.6. | MITT | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | EOT, SAC |
| Popula | tion Analysed | | | | |
| 1.7. | MITT | SP1 | Summary of Study Populations | | SAC |
| 1.8. | MITT | SP2 | Summary of Exclusions from the Per Protocol/Safety Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | · |
| 1.9. | MITT | DM1 | Summary of Demographic Characteristics | | EOT, SAC |
| 1.10. | APE | DM11 | Summary of Age Ranges | | SAC |
| 1.11. | MITT | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.12. | MITT | MH4 | Summary of Past Medical Conditions | | EOT, SAC |
| 1.13. | MITT | MH4 | Summary of Current Medical Conditions | | EOT, SAC |

| Study F | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.14. | MITT | FH1 | Summary of Family History of Cardiovascular Risk Factors | | EOT, SAC |
| 1.15. | MITT | SU1 | Summary of Smoking History at Screening | | EOT, SAC |
| 1.16. | MITT | SU1 | Summary of Smoking Status over the 12-Week Treatment Period | | EOT, SAC |
| 1.17. | MITT | SU1 | Summary of Smoking Status over the 12-Week Follow-Up<br>Period | | EOT, SAC |
| 1.18. | MITT | Example 7 | Summary of COPD Duration at Screening | | EOT, SAC |
| 1.19. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening | Use categories 0;1;2;3;≥3. Summarise moderate/severe, moderate; severe Include 7-Day History of COPD Exacerbations | EOT, SAC |
| 1.20. | MITT | Example 1 | Summary of COPD Exacerbation History at Screening by Country | | EOT, SAC |
| Concor | nitant Medicati | ons | | | |
| 1.21. | MITT | Example 14 | Summary of Baseline COPD Maintenance Therapy | | EOT, SAC |
| 1.22. | MITT | Example 15 | Summary of On-Treatment COPD Maintenance (Step-up)<br>Therapy | | EOT, SAC |
| 1.23. | MITT | CM1 | Summary of Concomitant Medications during 12-Week<br>Treatment Period | | EOT, SAC |
| 1.24. | MITT | Example 16 | Summary of OCS Use | | EOT, SAC |
| 1.25. | MITT | CM1 | Summary of Concomitant Medications during 12-Week Follow-<br>Up Period | | EOT, SAC |

200879

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.26. | MITT | EX1 | Summary of Exposure to Study Treatment | | EOT, SAC |
| 1.27. | MITT | Example 2 | Summary of Treatment Compliance | | EOT, SAC |
| 1.28. | MITT | Example 2 | Summary of actuations of study treatment measured by the clip-<br>on Propeller Sensor | | EOT, SAC |

## 13.11.5. Efficacy Tables

## 13.11.5.1. Efficacy tables for Interim Analysis 1

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | <u> </u> | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | IA1 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | IA1 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator (Dose Response Model) | | IA1 |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator (Dose Response Model) | | IA1 |
| 2.7. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.8. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA1 |
| 2.9. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post- bronchodilator (Repeated Measures Model) | | IA1 |
| 2.10. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre- bronchodilator (Repeated Measures Model) | | IA1 |
| 2.11. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post- bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| 2.12. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre- bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV₁ | | |
| 2.13. | MITT | Example 3 | Summary of Change from Hospital Discharge in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA1 |
| 2.14. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post- bronchodilator (Repeated Measures Model) | | IA1 |
| 2.15. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | IA1 |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post- bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| 2.17. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre- bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA1 |
| Rate of | Exacerbations | | | | |
| 2.18. | MITT | Example 5 | Summary of On-treatment Exacerbations | | IA1 |
| 2.19. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Severity | | IA1 |
| EXAcer | bations of Chro | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.20. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | Exclude statistical analysis information (summary only) | IA1 |
| 2.21. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | Exclude statistical analysis information (summary only) | IA1 |
| Other S | pirometry Mea | sures | | | |
| 2.22. | MITT | Example 3 | Summary of Spirometry Measurements | | IA1 |
| 2.23. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA1 |

200879

# 13.11.5.2. Efficacy tables for Interim Analysis 2

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | IA2 |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | IA2 |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.9. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.10. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.12. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.13. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.14. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.15. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| 2.16. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV₁ | | |
| 2.17. | MITT | Example 3 | Summary of Change from Hospital Discharge in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | IA2 |
| 2.18. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.19. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator (Dose Response Model) | | IA2 |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.20. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator (Dose Response Model) | | IA2 |
| 2.21. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.22. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.23. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | IA2 |
| 2.24. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.25. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | IA2 |
| 2.26. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| 2.27. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | IA2 |
| Rate of | Exacerbations | | | | |
| 2.28. | MITT | Example 5 | Summary of On-treatment Exacerbations | | IA2 |
| 2.29. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Severity | | IA2 |

| y: Tables | | | | |
|---|---|---|---|---|
| Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| MITT | Example 6 | Statistical Analysis of On-treatment Exacerbations | | IA2 |
| MITT | Example 6 | Subgroup Analysis of On-treatment Exacerbations by Index Exacerbation Severity | | IA2 |
| Next Exacerba | ation | | | |
| MITT | Example 8 | Summary and Statistical Analysis of Time to next On-treatment Exacerbation During the 12-Week Treatment Period | | IA2 |
| MITT | Example 8 | Subgroup Analysis of Time to next On-treatment Exacerbation During the 12-Week Treatment Period by Index Exacerbation Severity | | IA2 |
| bations of Chr | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | IA2 |
| MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | IA2 |
| Medication Us | e | | | • |
| MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | IA2 |
| MITT | RM1 | Summary of Percentage of Rescue-Free Days | | IA2 |
| pirometry Mea | sures | | <u> </u> | • |
| MITT | Example 3 | Summary of Spirometry Measurements | | IA2 |
| MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | IA2 |
| | Population MITT MITT Next Exacerba MITT MITT bations of Chra MITT Pirometry Mea | Population IDSL / Example Shell | Note | Population Example Shell Title Programming Notes |

200879

## 13.11.5.3. Efficacy tables for End of Treatment Interim Analysis and SAC

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change from Baseline in Clinic Visit trough FEV₁ | | | | | |
| 2.1. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.2. | MITT | Example 3 | Summary of FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator<br>Include additional row for hospital<br>discharge visit for Severe group | EOT, SAC |
| 2.3. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.4. | MITT | Example 3 | Summary of Change from Baseline in FEV <sub>1</sub> (L) by Index Exacerbation Severity | Include pre- and post-bronchodilator. Include additional row for hospital discharge visit for Severe group | EOT, SAC |
| 2.5. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.6. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.7. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.8. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.9. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.10. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.11. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | MITT | Example 26 | Statistical Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.13. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.14. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 14 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.15. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.16. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 28 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.17. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.18. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 56 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.19. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.20. | MITT | Example 26 | Subgroup Analysis of Change from Baseline in FEV <sub>1</sub> (L) at Day 84 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.22. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.23. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| 2.24. | MITT | Example 11 | Sensitivity Analysis of Change from Baseline in FEV <sub>1</sub> (L) measured pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV <sub>1</sub> | | |
| 2.25. | MITT | Example 3 | Summary of Change from Hospital Discharge in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.26. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.27. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 14 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.28. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.29. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.30. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.31. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.32. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.33. | MITT | Example 26 | Statistical Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured pre-bronchodilator (Dose Response Model) | | EOT, SAC |
| 2.34. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 14 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.35. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 14 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.36. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.37. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 28 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.38. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.39. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 56 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.40. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured post-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.41. | MITT | Example 26 | Subgroup Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) at Day 84 measured pre-bronchodilator by Index Exacerbation Severity (Dose Response Model) | | EOT, SAC |
| 2.42. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.43. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.44. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| 2.45. | MITT | Example 11 | Sensitivity Analysis of Change from Hospital Discharge in FEV <sub>1</sub> (L) measured pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| Change | from Day 84 ii | n Clinic Visit trouç | gh FEV <sub>1</sub> | | |
| 2.46. | MITT | Example 3 | Summary of Change from Day 84 in FEV <sub>1</sub> (L) | Include pre- and post-bronchodilator | EOT, SAC |
| 2.47. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) measured post-bronchodilator (Repeated Measures Model) | | EOT, SAC |
| 2.48. | MITT | Example 11 | Statistical Analysis of Change from Day 84 in FEV <sub>1</sub> (L) measured pre-bronchodilator (Repeated Measures Model) | | EOT, SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.49. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) measured post-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| 2.50. | MITT | Example 11 | Subgroup Analysis of Change from Day 84 in FEV <sub>1</sub> (L) measured pre-bronchodilator by Index Exacerbation Severity (Repeated Measures Model) | | EOT, SAC |
| Rate of | Exacerbations | i | | | |
| 2.51. | MITT | Example 5 | Summary of On-treatment Exacerbations | | EOT, SAC |
| 2.52. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.53. | MITT | Example 6 | Statistical Analysis of On-treatment Exacerbations | | EOT, SAC |
| 2.54. | MITT | Example 6 | Subgroup Analysis of On-treatment Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.55. | MITT | Example 5 | Summary of On-treatment Exacerbations by Index Exacerbation Type | | EOT, SAC |
| 2.56. | MITT | Example 5 | Summary of On-treatment Exacerbations by Number of Exacerbations in Previous 12 Months | | EOT, SAC |
| 2.57. | MITT | Example 5 | Summary of On-or Off-treatment Exacerbations During the 12-<br>Week Treatment Period | | EOT, SAC |
| 2.58. | MITT | Example 5 | Summary of On-or Off-treatment Exacerbations During the 12-<br>Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |
| 2.59. | MITT | Example 6 | Statistical Analysis of On- or Off-treatment Exacerbations During the 12-Week Treatment Period | | EOT, SAC |
| 2.60. | MITT | Example 6 | Subgroup Analysis of On- or Off-treatment Exacerbations During the 12-Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.61. | MITT | Example 5 | Summary of Off-treatment Exacerbations | | EOT, SAC |
| 2.62. | MITT | Example 5 | Summary of Off-treatment Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.63. | MITT | Example 6 | Statistical Analysis of Off-treatment Exacerbations | | EOT, SAC |
| 2.64. | MITT | Example 6 | Subgroup Analysis of Off-treatment Exacerbations by Index Exacerbation Severity | | EOT, SAC |
| 2.65. | MITT | Example 5 | Summary of On- and Off-treatment Exacerbations During the 24-Week Study Period | | EOT, SAC |
| 2.66. | MITT | Example 5 | Summary of On- and Off-treatment Exacerbations During the 24-Week Study Period by Index Exacerbation Severity | | EOT, SAC |
| 2.67. | MITT | Example 6 | Statistical Analysis of On- and Off-treatment Exacerbations During the 24-Week Study Period | | EOT, SAC |
| 2.68. | MITT | Example 6 | Subgroup Analysis of On- and Off-treatment Exacerbations During the 24-Week Study Period by Index Exacerbation Severity | | EOT, SAC |
| Time to | Next Exacerba | ation | | | |
| 2.69. | MITT | Example 8 | Summary and Statistical Analysis of Time to next On-treatment Exacerbation During the 12-Week Treatment Period | | EOT, SAC |
| 2.70. | MITT | Example 8 | Subgroup Analysis of Time to next On-treatment Exacerbation During the 12-Week Treatment Period by Index Exacerbation Severity | | EOT, SAC |
| 2.71. | MITT | Example 8 | Summary and Statistical Analysis of Time to next On- or Off-<br>treatment Exacerbation During the 12-Week Treatment Period | | EOT, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.72. | MITT | Example 8 | Statistical Analysis of Time to next On- or Off-treatment<br>Exacerbation During the 12-Week Treatment Period by Index<br>Exacerbation Severity | | EOT, SAC |
| 2.73. | MITT | Example 8 | Summary and Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment | | EOT, SAC |
| 2.74. | MITT | Example 8 | Statistical Analysis of Time to Next Exacerbation Following Cessation of Study Treatment by Index Exacerbation Severity | | EOT, SAC |
| EXAce | bations of Chro | onic Pulmonary D | isease Tool - Patient Reported Outcome (EXACT) | | |
| 2.75. | MITT | Example 9 | Statistical Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Visit | | EOT, SAC |
| 2.76. | MITT | Example 9 | Subgroup Analysis of Proportion of Participants Achieving the EXACT-definition of Recovery by Index Exacerbation Severity | | EOT, SAC |
| 2.77. | MITT | Example 8 | Summary and Statistical Analysis of Time to EXACT-defined Recovery | | EOT, SAC |
| 2.78. | MITT | Example 8 | Subgroup Analysis of Time to EXACT-defined Recovery by Index Exacerbation Severity | | EOT, SAC |
| 2.79. | MITT | Example 10 | Summary of severity of subsequent HCRU-defined exacerbation during 12-Week Treatment Period | Also split by moderate and severe | EOT, SAC |
| 2.80. | MITT | Example 10 | Summary of severity of subsequent HCRU-defined exacerbation during 12-Week Follow-up Period | Also split by moderate and severe | EOT, SAC |
| COPD | Assessment Te | st (CAT) | | | |
| 2.81. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score | | EOT, SAC |
| 2.82. | MITT | Example 3 | Summary of Change from Baseline in CAT Total Score by Index Exacerbation Severity | | EOT, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.83. | MITT | Example 9 | Statistical Analysis of Proportion of Responders Using the CAT Total Score by Visit | | EOT, SAC |
| 2.84. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders Using the CAT Total Score by Visit by Index Exacerbation Severity | | EOT, SAC |
| 2.85. | MITT | Example 11 | Statistical Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.86. | MITT | Example 11 | Subgroup Analysis of Change from Baseline in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |
| 2.87. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score | | EOT, SAC |
| 2.88. | MITT | Example 3 | Summary of Change from End of Treatment in CAT Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.89. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.90. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in CAT Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |
| St. Geo | rge's Respirato | ory Questionnaire | (SGRQ) | | |
| 2.91. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score | | EOT, SAC |
| 2.92. | MITT | Example 3 | Summary of Change from Baseline in SGRQ Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.93. | MITT | Example 9 | Statistical Analysis of Proportion of Responders on the SGRQ<br>Total Score by Visit | | EOT, SAC |
| 2.94. | MITT | Example 9 | Subgroup Analysis of Proportion of Responders on the SGRQ Total Score by Index Exacerbation Severity | | EOT, SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.95. | MITT | Example 11 | Statistical Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.96. | MITT | Example 11 | Subgroup Analysis of Change from Baseline SGRQ Total Score (Repeated Measures Model) by Index Exacerbation Severity | | EOT, SAC |
| 2.97. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score | | EOT, SAC |
| 2.98. | MITT | Example 3 | Summary of Change from End of Treatment in SGRQ Total Score by Index Exacerbation Severity | | EOT, SAC |
| 2.99. | MITT | Example 11 | Statistical Analysis of Change from End of Treatment in SGRQ Total Score (Repeated Measures Model) | | EOT, SAC |
| 2.100. | MITT | Example 11 | Subgroup Analysis of Change from End of Treatment in SGRQ<br>Total Score (Repeated Measures Model) by Index Exacerbation<br>Severity | | EOT, SAC |
| E-RS: C | OPD | | | | |
| 2.101. | MITT | Example 3 | Summary of Change from Baseline in E-RS: COPD and subscales | | SAC |
| Rescue | Medication Us | se . | | | |
| 2.102. | MITT | RM1 | Summary of Mean Number of Occasions of Rescue Medication Use Per Day | | EOT, SAC |
| 2.103. | MITT | RM1 | Summary of Percentage of Rescue-Free Days | | EOT, SAC |
| 2.104. | MITT | RM1 | Summary of Mean Number of Actuations of Rescue Medication Use Per Day via the clip-on Propeller Sensor for MDI | | EOT, SAC |
| 2.105. | MITT | RM1 | Summary of Percentage of Rescue-Free Days via the clip-on Propeller Sensor for MDI | | EOT, SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Compli | ance | | | | |
| 2.106. | MITT | IP1 | Summary of Overall IP Compliance | | EOT, SAC |
| 2.107. | MITT | IP1 | Summary of Overall IP Compliance via the clip-on Propeller Sensor for ELLIPTA | | EOT, SAC |
| Healtho | are Resource I | Utilisation | | | |
| 2.108. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilisation | | EOT, SA |
| 2.109. | MITT | Example 19 | Summary of Exacerbation Related Unscheduled Healthcare Resource Utilization by Index Exacerbation Severity | | EOT, SA |
| 2.110. | MITT | Example 21 | Summary of Exacerbation Related Hospitalizations | | EOT, SAC |
| 2.111. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation | | EOT, SAC |
| 2.112. | MITT | Example 19 | Summary of COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | EOT, SAC |
| 2.113. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation | | EOT, SAC |
| 2.114. | MITT | Example 20 | Summary of Non-COPD Related Unscheduled Healthcare Resource Utilisation by Index Exacerbation Severity | | EOT, SAC |
| 2.115. | MITT | Example 22 | Summary of Re-hospitalization Within 30 days of Index Exacerbation | | EOT, SAC |
| 2.116. | MITT | Example 24 | Summary of Time from Resolution of Index Exacerbation to Next Exacerbation | | EOT, SAC |
| 2.117. | MITT | Example 23 | Summary of Subsequent Exacerbation Treatment | | EOT, SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Other S | pirometry Mea | sures | | | |
| 2.118. | MITT | Example 3 | Summary of Spirometry Measurements | | EOT, SAC |
| 2.119. | MITT | Example 3 | Summary of Change from Baseline in Spirometry Measurements | | EOT, SAC |
| Inflamm | natory/infective | Markers in Blood | I and Sputum | | |
| 2.120. | MITT | Example 3 | Summary of Inflammatory Markers in Blood | | SAC |
| 2.121. | MITT | Example 3 | Summary of Inflammatory Markers in Sputum | | SAC |

200879

## 13.11.6. Efficacy Figures

## 13.11.6.1. Efficacy Figures for Interim Analysis 1

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator | | IA1 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator | | IA1 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA1 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA1 |

200879

## 13.11.6.2. Efficacy Figures for Interim Analysis 2

| Efficacy | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator | | IA2 |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator | | IA2 |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 measured post-bronchodilator | | IA2 |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 measured post-bronchodilator | | IA2 |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 14 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 56 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> at Day 84 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV <sub>1</sub> | | |
| 2.13. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 28 measured post-bronchodilator | | IA2 |
| 2.14. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 56 measured post-bronchodilator | | IA2 |
| 2.15. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 84 measured post-bronchodilator | | IA2 |
| 2.16. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.17. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> at Day 28 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.18. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 56 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |

200879

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.19. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 56 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |
| 2.20. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 84 measured post-bronchodilator by Index Exacerbation Severity: Moderate | | IA2 |
| 2.21. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ at Day 84 measured post-bronchodilator by Index Exacerbation Severity: Severe | | IA2 |

### 13.11.6.3. Efficacy Figures for End of Treatment Interim Analysis and SAC

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Change | from Baseline | in Clinic Visit tro | ugh FEV₁ | | |
| 2.1. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured post-bronchodilator | | EOT, SAC |
| 2.2. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured pre-bronchodilator | | EOT, SAC |
| 2.3. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC |
| 2.4. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.5. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured pre-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC |
| 2.6. | MITT | Example 18 | Plot of Dose Response Model of Change from Baseline in FEV <sub>1</sub> measured pre-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC |
| Change | from Hospital | Discharge in Clin | ic Visit trough FEV₁ | | |
| 2.7. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV₁ measured post-bronchodilator | | EOT, SAC |
| 2.8. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> measured pre-bronchodilator | | EOT, SAC |
| 2.9. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> measured post-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC |
| 2.10. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> measured post-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC |
| 2.11. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> measured pre-bronchodilator by Index Exacerbation Severity: Moderate | | EOT, SAC |
| 2.12. | MITT | Example 18 | Plot of Dose Response Model of Change from Hospital Discharge in FEV <sub>1</sub> measured pre-bronchodilator by Index Exacerbation Severity: Severe | | EOT, SAC |

200879

## 13.11.7. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term | | SAC |
| 3.2. | Safety | AE1 | Summary of Post-Treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Treatment Emergent Adverse Events by Overall Frequency | | SAC |
| 3.4. | Safety | AE1 | Summary of Treatment Emergent Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.5. | Safety | AE15 | Summary of Common (>=5%) Non-serious Treatment Emergent<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | | SAC |
| 3.6. | Safety | AE1 | Summary of Treatment Emergent Adverse Events for<br>Participants with Absolute Neutrophil Count Below Lower Value of PCI | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 3.7. | Safety | AE16 | Summary of Serious Treatment Emergent Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Participants and Occurrences) | | SAC |
| 3.8. | Safety | AE16 | Summary of Fatal Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | Only with subcategory: Number of Fatal SAEs | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | Safety | AE1 | Summary of Serious Treatment Emergent Drug-related Adverse<br>Events by System Organ Class and Preferred Term | | SAC |
| 3.10. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | SAC |
| 3.11. | Safety | AE1 | Summary of Post-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.12. | Safety | AE1 | Summary of Treatment Emergent Adverse Events of Special Interest by Lower Level Term | | SAC |
| 3.13. | Safety | Example 17 | Summary of Post-Inhalation Cough by Visit | | SAC |
| 3.14. | Safety | Example 28 | Summary of Post-Inhalation Cough by Visit and Cough Type | | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 3.15. | Safety | LB1 | Summary of Chemistry Data | | SAC |
| 3.16. | Safety | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.17. | Safety | LB1 | Summary of Hematology Data | | SAC |
| 3.18. | Safety | LB1 | Summary of Change from Baseline in Hematology | Only for WBC, lymphocytes, neutrophils | SAC |
| 3.19. | Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.20. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC |
| 3.21. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 3.22. | Safety | EG1 | Summary of ECG Findings | | SAC |
| 3.23. | Safety | EG2 | Summary of ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | SAC |
| 3.24. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | For the following parameters: QTcF, QTcB, PR, Heart rate | SAC |
| 3.25. | Safety | Example 27 | Summary of QTcF Categories | | SAC |
| 3.26. | Safety | Example 27 | Summary of QTcB Categories | | SAC |
| 3.27. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.28. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.29. | Safety | Example 25 | Summary of ECG Abnormalities for Participants with Any Abnormal Clinically Significant ECG Interpretation | | SAC |
| Vital Si | gns | | | | |
| 3.30. | Safety | VS1 | Summary of Vital Signs | | SAC |
| 3.31. | Safety | VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | | SAC |

200879

# 13.11.8. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory | | | | |
| 3.1. | Safety | LB7 | LFT Shift from Baseline to Maximum | | SAC |
| 3.2. | Safety | Example 13 | Median (range) Absolute Neutrophil Count by Time and Treatment | | SAC |
| ECG | ECG | | | | |
| 3.3. | Safety | EG8 | Distribution of QTcF Change by Time and Treatment | | SAC |

## 13.11.9. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetic Concentration-Time Data | | | | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK2269557 Pharmacokinetic Concentration-Time Data | | SAC |
| 4.2. | PK | PK05 | Summary of Log-Transformed Plasma GSK2269557<br>Pharmacokinetic Concentration-Time Data | | SAC |

200879

# 13.11.10. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | MITT | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | MITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 4. | MITT | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | | SAC |
| 5. | MITT | TA1 | Listing of Planned and Actual Treatments | | SAC |
| Protoc | ol Deviations | 1 | | | |
| 6. | MITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 7. | MITT | IE3 | Listing of Participants with Inclusion/Exclusion Criteria<br>Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 8. | MITT | SP3 | Listing of Participants Excluded from Any Population | For participants excluded from MITT population (i.e. participants in the MITT but not in PP) | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | MITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 10. | MITT | DM9 | Listing of Race | | SAC |
| Prior and Concomitant Medications | | | | | |
| 11. | MITT | CP_CM3 | Listing of Concomitant Medications | | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | Exposure and Treatment Compliance | | | | |
| 12. | Safety | EX3 | Listing of Exposure Data | | SAC |
| Advers | e Events | | | | |
| 13. | Safety | AE8 | Listing of All Adverse Events | | SAC |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | • |
| 16. | Safety | AE8 | Listing of Fatal Serious Adverse Events | | SAC |
| 17. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 18. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| Hepatobiliary (Liver) | | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping<br>Events | | SAC |
| All Lab | oratory | | | | • |
| 22. | Safety | LB5 | Listing of All Chemistry Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 23. | Safety | LB14 | Listing of Chemistry Data with Character Results | | SAC |

200879

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Safety | LB5 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| 25. | Safety | LB14 | Listing of all Hematology Data with Character Results | | SAC |
| ECG | | | | | |
| 26. | Safety | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | | SAC |
| 27. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal Finding | | SAC |

# 13.11.11. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 28. | MITT | Example 29 | Listing of Subjects who Received Incorrect Medication | | SAC |
| 29. | PK | PK07 | Listing of Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 30. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC |

200879

# 13.12. Appendix 12: Example Mock Shells for Data Displays

#### 13.12.1. Example shell 1

Example Shell X

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Exacerbation History at Screening

| | Treatment A (N=100) | Treatment B (N=100) | Total (N=200) |
|---|---|---|---|
| Moderate COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Severe COPD exacerbations | | | |
| n | X | X | X |
| 0 | xx (x%) | xx (x%) | xx (x%) |
| 1 | xx (x%) | xx (x%) | xx (x%) |
| >=2 | xx (x%) | xx (x%) | xx (x%) |
| Total number of moderate/severe COPD exacerbations | | | |
| n | 911 | 899 | 1810 |
| 0 | 313 (34%) | 317 (35%) | 630 (35%) |
| 1 | 252 (28%) | 253 (28%) | 505 (28%) |
| >=2 | 346 (38%) | 329 (37%) | 675 (37%) |

Note: Number of COPD exacerbations reported in the 12 months prior to the Screening Visit.

PPD
200879

# 13.12.2. Example Shell 2

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific
Table X

Summary of Treatment Compliance

| | Treatment A (N=100) | Treatment B (N=100) | Total (N=200) |
|---|---|---|---|
| Overall compliance (%) | | | |
| n | XX | XX | XX |
| Mean | XX | XX | XX |
| SD | XX | XX | XX |
| Median | XX | XX | XX |
| Min. | XX | XX | XX |
| Max. | xx | XX | XX |
| Compliance interval | | | |
| < 80% | xx (x%) | xx (x%) | xx (x%) |
| 80% - < 100% | xx (x%) | xx (x%) | xx (x%) |
| 100% - < 120% | xx (x%) | xx (x%) | xx (x%) |
| >=120% | xx (x%) | xx (x%) | xx (x%) |

200879

## 13.12.3. Example shell 3

Example Shell X Protocol: ABC123456

cocol: ABC123456 Page 1 of n

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of Change from Baseline in FEV1 (L)  $\begin{tabular}{ll} Measured post-bronchodilator \end{tabular}$ 

| Visit | N | Treatment Arm | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| Day 1 | 200 | Placebo | 200 | 0.111 | 0.1111 | 0.100 | -0.11 | 1.11 |
| - | 200 | GSK2269557 12.5 mc | g 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | 200 | GSK2269557 50 mc | g 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | 200 | GSK2269557 100 mc | g 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | 200 | GSK2269557 250 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 500 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 750 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| Day 14 | 200 | Placebo | 200 | 0.111 | 0.1111 | 0.100 | -0.11 | 1.11 |
| | 200 | GSK2269557 12.5 mc | g 190 | 0.222 | 0.2222 | 0.200 | -0.22 | 1.22 |
| | 200 | GSK2269557 50 mc | g 195 | 0.333 | 0.3333 | 0.300 | -0.33 | 1.33 |
| | 200 | GSK2269557 250 mc | g 195 | 0.444 | 0.4444 | 0.400 | -0.44 | 1.44 |
| | 200 | GSK2269557 500 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |
| | 200 | GSK2269557 750 mc | g 190 | 0.555 | 0.5555 | 0.500 | -0.55 | 1.55 |

200879

## 13.12.4. Example Shell 4

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Statistical Analysis of Change from Baseline in FEV1 (ml)  $$\operatorname{Measured}$ \operatorname{post-bronchodilator}$ 

| Visit | N | Treatment Arm | : | | osterior<br>Median | 95% Credible<br>Interval |
|---|---|---|---|---|---|---|
| Day 14 | Х | Placebo | X | Κ. | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 12.5 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 50 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 100 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 250 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 500 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 750 m | mcg x | X | X.XX | (x.xx, x.xx) |
| Day 28 | Х | Placebo | X | K | x.xx | (x.xx, x.xx) |
| | Х | GSK2269557 12.5 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 50 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 100 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 250 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 500 m | mcg x | K | X.XX | (x.xx, x.xx) |
| | Х | GSK2269557 750 m | mcg x | K | X.XX | (x.xx, x.xx) |

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Statistical Analysis of Change from Baseline in FEV1 (ml)
Measured post-bronchodilator

| Visit | Treatment Comparison | Adjusted<br>Median<br>Difference | Std Dev | 95% Credible<br>Interval | Prob Treat. Diff >0 (%) |
|---|---|---|---|---|---|
| Day 14 | GSK2269557 12.5 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 50 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 100 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 250 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 500 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 750 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| Day 28 | GSK2269557 12.5 mg vs<br>Placebo | x.xx | X.XX | (x.xx, x.xx) | x.xx |
| | GSK2269557 50 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |
| | GSK2269557 100 mg vs<br>Placebo | x.xx | x.xx | (x.xx, x.xx) | x.xx |

200879

## 13.12.5. Example Shell 5

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific
Table X

Summary of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Number of moderate & severe exacerbations per subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |
| 4 | 0 | 2 (2%) |
| 5 | 0 | 1 (1%) |
| >5 | 0 | 1 (1%) |
| Subjects with >=1 moderate & severe exacerbation | 13 (13%) | 28 (28%) |
| Total Number of moderate & severe exacerbations | 21 | 49 |
| Number of moderate exacerbations per Subject | | |
| 0 | 50 (50%) | 98 (98%) |
| 1 | 6 (6%) | 15 (15%) |
| 2 | 6 (6%) | 9 (9%) |
| 3 | 1 (1%) | 1 (1%) |

200879

## 13.12.6. Example Shell 6

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Statistical Analysis of On-treatment Exacerbations

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Moderate and severe exacerbations | | |
| Annual exacerbation rate (95% CrI) | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx) |
| Active vs. Placebo | | |
| Ratio | | 0.85 (x.xx, x.xx) |
| Pr Diff <1 | | x.xx |
| Percent reduction in rate (95% CrI) | | 15% (x.xx, x.xx) |
| Moderate exacerbations | | |
| Annual exacerbation rate (95% CrI) | 0.35 (x.xx, x.xx) | 0.30 (x.xx, x.xx) |
| Active vs. Placebo | | |
| Ratio | | 0.85 (x.xx, x.xx) |
| Pr Diff <1 | | x.xx |
| Percent reduction in rate (95% CrI) | | 15% (x.xx, x.xx) |

200879

## 13.12.7. Example Shell 7

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Duration at Screening

| | Treatment A (N=100) | | Treatment B (N=100) | | Total (N=200) | |
|---|---|---|---|---|---|---|
| Duration of COPD: | | | | | | |
| n | 100 | | 99 | | 199 | |
| <1 year | XX | (x%) | XX | (x%) | XX | (x%) |
| >=1 to <5 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=5 to <10 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=10 to <15 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=15 to <20 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=20 to <25 years | XX | (x%) | XX | (x%) | XX | (x%) |
| >=25 years | XX | (x%) | XX | (x%) | XX | (x%) |

200879

## 13.12.8. Example Shell 8

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary and Analysis of Time to Next On-treatment Moderate or Severe Exacerbation (days) up to Day  $84\,$ 

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Number of Subjects with Event<br>Number of Subjects Censored | 10 (10%)<br>90 (90%) | 14 (14%)<br>86 (86%) |
| Probability of Having Event (%) 95% C.I. | X.X<br>(x.x, x.x) | XX<br>(x.x, x.x) |
| Treatment A vs. Placebo<br>Hazard Ratio<br>95% Credible Interval | X.XX<br>(x.xx, x.xx) | |

Note: Probability of having event, 95% C.I. are taken from the Kaplan-Meier analysis. Note: Hazard ratio and 95% Credible Interval are from a Bayesian Cox proportional hazards model

200879

## 13.12.9. Example Shell 9

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Statistical Analysis of Proportion of Participants Achieving EXACT-definition of Response

| | Treatment A (N=100) | |
|----------------------|--------------------------|--------------------------|
| Day 14 | | |
| n | x.xx | x.xx |
| Responder | x.xx (x%) | x.xx (x%) |
| Non-responder | x.xx (x%) | x.xx (x%) |
| Active vs. Placebo | | |
| Odds Ratio (95% CrI) | x.xx ( $x.xx$ , $x.xx$ ) | x.xx ( $x.xx$ , $x.xx$ ) |
| Pr Diff >1 | x.xx | X.XX |
| Day 28 | | |
| n | X.XX | x.xx |
| Responder | x.xx (x%) | x.xx (x%) |
| Non-responder | x.xx (x%) | x.xx (x%) |
| Active vs. Placebo | | |
| Odds Ratio (95% CrI) | x.xx ( $x.xx$ , $x.xx$ ) | x.xx ( $x.xx$ , $x.xx$ ) |
| Pr Diff >1 | x.xx | X.XX |

200879

## 13.12.10. Example Shell 10


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of severity of subsequent HCRU-defined exacerbation during 12-Week Treatment Period

| Treatment | N | n | Mean | SD | Median | Min. | Max. |
|-----------|----|----|-------|-------|--------|-------|-------|
| Placebo | 30 | 30 | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |
| Trt A | 30 | 30 | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx |
| Trt B | 30 | 30 | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |

200879

## 13.12.11. Example Shell 11

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Mixed Model Repeated Measures Analysis of CAT Total Score

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Day 28 | | |
| n | X.XX | x.xx |
| Adjusted mean score change (SE) | x.xx (x) | x.xx (x) |
| Active - Placebo | | |
| Difference (SE) | x.xx (x.xx) | x.xx (x.xx) |
| 95% (CrI) | X.XX | X.XX |
| Pr Diff >0 | X.XX | X.XX |
| Day 56 | | |
| n | X.XX | x.xx |
| Adjusted mean score change (SE) | x.xx (x) | x.xx (x) |
| Active - Placebo | | |
| Difference (SE) | x.xx (x.xx) | x.xx (x.xx) |
| 95% (CrI) | X.XX | X.XX |
| Pr Diff >0 | X.XX | x.xx |

200879

## 13.12.12. Example Shell 12

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | | ment A<br>0) | Treatment B (N=100) | |
|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | | (97%)<br>( 3%) | | (19%)<br>(81%) |
| Number of Home Visits (day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>90<br>4<br>0<br>0<br>0 | (90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2<br>4 | (92%)<br>(4%)<br>(<1%) |
| Number of Home Visits (night) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>100 (3<br>0<br>0<br>0<br>0 | 100%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) |

<sup>[1]</sup> Total number of contacts across all subjects.

PPC

<sup>[2]</sup> Total number of days across all subjects.

200879

## CONFIDENTIAL

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Trea<br>(N=1 | atment A<br>.00) | Trea<br>(N=1 | atment B<br>LOO) |
|---|---|---|---|---|---|
| Number of Office/Practice Visits | n | 911 | | 899 | |
| | 0 | 846 | (93%) | 808 | (90%) |
| | 1 | 42 | (5%) | 58 | (6%) |
| | 2 | | (1%) | 23 | (3%) |
| | 3 | | (<1%) | | (<1%) |
| | >3 | | (<1%) | | (<1%) |
| | Total [1] | 103 | | 140 | |
| Number of Urgent Care/Outpatient Visits | n | 911 | | 899 | |
| Name of orgone date, daspasions vision | 0 | | (97%) | | (98%) |
| | 1 | | (2%) | | (1%) |
| | 2 | | (<1%) | | (<1%) |
| | 3 | | (<1%) | | (<1%) |
| | >3 | | (<1%) | | (<1%) |
| | Total [1] | 54 | | 37 | |
| Number of Proposition People Visite | | 911 | | 899 | |
| Number of Emergency Room Visits | n | | (>000) | | (>000) |
| | 0<br>1 | 906<br>5 | (>99%)<br>(<1%) | | (>99%)<br>(<1%) |
| | 2 | 0 | (<10) | | (<1%)<br>(<1%) |
| | 3 | 0 | | 0 | ( < ± 0 ) |
| | >3 | 0 | | 0 | |
| | Total [1] | 5 | | 7 | |
| | 10001 [1] | 9 | | , | |

<sup>[1]</sup> Total number of contacts across all subjects.

PPD

104

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table 2.159

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Days in Intensive Care | n | 911 | 899 |
| <del>-</del> | 0 | 910 (>99%) | 894 (>99%) |
| | 1 | 0 | 0 |
| | 2 | 0 | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 1 (<1%) | 4 (<1%) |
| | Total [2] | 12 | 40 |
| Number of Days in General Ward | n | 911 | 899 |
| | 0 | 896 (98%) | 878 (98%) |
| | 1 | 0 | 2 (<1%) |
| | 2 | 1 (<1%) | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 14 (2%) | 18 (2%) |
| | Total [2] | 119 | 258 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

## 13.12.13. Example shell 13

Protocol: XYZ100001 

Population: Intent-to-Treat/Safety/Other study specific



200879


# 13.12.14. Example Shell 14

Protocol: XYZ100001
Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Baseline COPD Maintenance Therapy

| Therapy category | Treatment A (N=81) | Treatment B (N=79) |
|---|---|---|
| Any medication at baseline | 70 (86%) | 50 (63%) |
| Monotherapy<br>LAMA only | X (x%)<br>x (x%) | X (x%)<br>x (x%) |
| Dual therapy<br>ICS/LABA<br>Dual bronchodilator | x (x%)<br>x (x%)<br>xx (xx%) | x (x%)<br>x (x%)<br>xx (xx%) |
| Triple therapy<br>LAMA/ICS/LABA | X (x%)<br>x (x%) | X (x%) |

200879

# 13.12.15. Example Shell 15


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of On-Treatment COPD Maintenance (Step-up) Therapy

| | Treatment A | Treatment B |
|---------------------|-------------|-------------|
| Therapy category | (N=81) | (N=79) |
| Any Step-up Therapy | 70 (86%) | 50 (63%) |

200879

## 13.12.16. Example shell 16


Population: Intent-to-Treat/Safety/Other study specific

Table X
Summary of OCS use

| | Treatment A<br>(N=81) | Treatment B (N=79) |
|---------------------------------|-----------------------|--------------------|
| OCS use for index exacerbation | 81 (100%) | 79 (100%) |
| Total number of Days of OCS use | | |
| Mean | Xx | XX |
| SD | Xx | xx |
| Median | Xx | XX |
| Min. | Xx | xx |
| Max. | Xx | XX |
| On-treatment OCS use | xx (xx%) | xx (xx%) |
| Total number of Days of OCS use | | |
| Mean | Xx | XX |
| SD | Xx | XX |
| Median | Xx | XX |
| Min. | Xx | XX |
| Max. | Xx | xx |

200879

## 13.12.17. Example Shell 17


Population: Safety

Table X
Summary of Post-Inhalation Cough by Visit

Visit: VISIT 2 (RANDOMISATION)

| · · · | | acebo | 50 | K2269557<br>mcg<br>i=14) | 10 | K2269557<br>0 mcg<br>=15) | 25 | K2269557<br>0 mcg<br>=16) | 50 | SK2269557<br>)0 mcg<br>J=14) | 750 | (2269557<br>) mcg<br>=42) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Did subject experience PI cough? [1] | | | | | | | | | | | | |
| n | 20 | | 10 | | 12 | | 15 | | 1 | .2 | 35 | 5 |
| Yes | 7 | (35%) | 4 | (40%) | 6 | (50%) | 3 | (20%) | | 6 (50%) | 12 | 2 (34%) |
| No | 13 | (65%) | 6 | (60%) | 6 | (50%) | 12 | (80%) | | 6 (50%) | 23 | 8 (66%) |
| Type of cough | | | | | | | | | | | | |
| Single cough | 4 | (57%) | 2 | (50%) | 1 | (17%) | 1 | (33%) | 1 | (17%) | 2 | (17%) |
| Intermittent cough | 2 | (29%) | 2 | (50%) | 5 | (83%) | 1 | (33%) | 4 | (67%) | 5 | (42%) |
| Continuous cough | 1 | (14%) | 0 | | 0 | | 1 | (33%) | 1 | (17%) | 5 | (42%) |
| Severity of cough | | | | | | | | | | | | |
| Mild | 5 | (71%) | 3 | (75%) | 3 | (50%) | 2 | (67%) | 1 | (17%) | 6 | (50%) |
| Moderate | 2 | (29%) | 1 | (25%) | 2 | (33%) | 1 | (33%) | 5 | (83%) | 4 | (33%) |
| Severe | 0 | | 0 | | 1 | (17%) | 0 | | 0 | | 2 | (17%) |
| Time to onset of PI cough (minutes) | | | | | | | | | | | | |
| 0-1 | 6 | (86%) | 3 | (75%) | 6 | (100%) | 3 | (100%) | 6 | (100%) | 12 | (100%) |
| >1-2 | 1 | (14%) | 1 | (25%) | 0 | | 0 | | 0 | | 0 | |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| Duration of PI cough (minutes) | | | | | | | | | | | | |
| <=1 | 6 | (86%) | 3 | (75%) | 5 | (83%) | 3 | (100%) | 5 | (83%) | 11 | (92%) |
| >1-2 | 1 | (14%) | 1 | (25%) | 1 | (17%) | 0 | | 1 | (17%) | 1 | (8%) |
| >2-3 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >3-4 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| >4-5 | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |

# 2019N398117\_00

200879

## CONFIDENTIAL

| >5-10 | Х | | Х | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| >10-30 | Х | | X | | | | | | | | | |
| >30 | Х | | Х | | | | | | | | | |
| Number of subjects reporting cough as AE/SAE Mild Moderate Severe | 2<br>x<br>x | (29%)<br>(x%)<br>(x%)<br>(x%) | 1<br>x<br>x | (25%) | 4 | (67%) | 0 | 2 | 2 | (33%) | 3 | (25%) |

<sup>[1]</sup> Percentages are calculated using the number of subjects evaluated at visit as the denominator.

All other percentages are calculated using the number of subjects with a PI cough at visit as the denominator.

200879


## 13.12.18. Example shell 18

Protocol: ABC123456
Population: Intent-to-Treat/Safety/Other study specific

Figure X

Plot of Dose Response Model of Change from Baseline in FEV1



[Footnote to describe the fitted model]

200879

## 13.12.19. Example Shell 19

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | | ent A<br>) | | tment B |
|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | | 97%)<br>3%) | | (19%)<br>(81%) |
| Number of Home Visits (day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | | 90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2<br>4 | (92%)<br>(4%)<br>(<1%) |
| Number of Home Visits (night) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | 100<br>100 (10<br>0<br>0<br>0<br>0 | 00%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Office/Practice Visits | n | 911 | 899 |
| | 0 | 846 (93%) | 808 (90%) |
| | 1 | 42 (5%) | |
| | 2 | 13 (1%) | 23 (3%) |
| | 3 | 7 (<1%) | 8 (<1%) |
| | >3 | 3 (<1%) | 2 (<1%) |
| | Total [1] | 103 | 140 |
| Number of Urgent Care/Outpatient Visits | n | 911 | 899 |
| Number of orgent care, outpatient visits | 0 | 886 (97%) | |
| | 1 | 15 (2%) | |
| | 2 | , , | 2 (<1%) |
| | 3 | 3 (<1%) | 3 (<1%) |
| | >3 | 4 (<1%) | |
| | Total [1] | , , | 37 |
| North and G. Francisco Description | - | 011 | 0.00 |
| Number of Emergency Room Visits | n | 911 | 899 |
| | 0 | 906 (>99%) | |
| | 1<br>2 | 5 (<1%) | 5 (<1%)<br>1 (<1%) |
| | ∠<br>3 | 0 | 1 (<1%)<br>0 |
| | >3 | 0 | 0 |
| | 73<br>Total [1] | 5 | 7 |
| | IUCAI [I] | J | / |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific Table  ${\tt X}$ 

Summary of COPD Related Unscheduled Healthcare Resource Utilization

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Number of Days in Intensive Care | n | 911 | 899 |
| | 0 | 910 (>99%) | 894 (>99%) |
| | 1 | 0 | 0 |
| | 2 | 0 | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 1 (<1%) | 4 (<1%) |
| | Total [2] | 12 | 40 |
| Number of Days in General Ward | n | 911 | 899 |
| | 0 | 896 (98%) | 878 (98%) |
| | 1 | 0 | 2 (<1%) |
| | 2 | 1 (<1%) | 1 (<1%) |
| | 3 | 0 | 0 |
| | >3 | 14 (2%) | 18 (2%) |
| | Total [2] | 119 | 258 |

<sup>[1]</sup> Total number of contacts across all subjects.

<sup>[2]</sup> Total number of days across all subjects.

200879

## 13.12.20. Example Shell 20


Population: Intent-to-Treat/Safety/Other study specific

Summary of Non-COPD Related Unscheduled Healthcare Resource Utilization

| | | | tment A | | atment B | \$ |
|---|---|---|---|---|---|---|
| Unscheduled Healthcare Utilisation | Yes<br>No | | (97%)<br>(3%) | | (19%)<br>(81%) | |
| Number of Days in Accident and emergency | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>90<br>4<br>0<br>0<br>0 | (90%)<br>(4%) | 100<br>92<br>4<br>0<br>0<br>2 | (92%)<br>(4%)<br>(<1%) | |
| Number of Days in General Ward | n<br>0<br>1<br>2<br>3<br>>3<br>Total | 100<br>100<br>0<br>0<br>0<br>0 | (100%) | 100<br>100<br>0<br>0<br>0<br>0 | (100%) | |

200879

# 13.12.21. Example Shell 21

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of Exacerbation Related Hospitalizations

| | Treatment A (N=100) | |
|-----------------------------------|---------------------|------|
| Index exacerbation | | |
| Participants with hospitalization | x.xx | x.xx |
| Number of hospitalizations | x.xx | x.xx |
| Mean duration (days) | X.XX | x.xx |
| SD | X.XX | x.xx |
| Median duration (days) | X.XX | x.xx |
| Minimum duration (days) | X.XX | X.XX |
| Maximum duration (days) | X.XX | X.XX |
| Subsequent exacerbations | | |
| Participants with hospitalization | X.XX | x.xx |
| Number of hospitalizations | X.XX | x.xx |
| Mean duration (days) | X.XX | x.xx |
| SD | X.XX | x.xx |
| Median duration (days) | X.XX | x.xx |
| Minimum duration (days) | X.XX | x.xx |
| Maximum duration (days) | X.XX | X.XX |

200879

## 13.12.22. Example Shell 22

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Re-hospitalization Within 30 days of Index Exacerbation

| | | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|---|
| Re-hospitalization Within 30 days | Yes | 97 (97%) | 19 (19%) |
| | No | 3 (3%) | 81 (81%) |

200879

## 13.12.23. Example Shell 23


Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Subsequent Exacerbation Treatment

| | Treatment A (N=81) | Treatment B (N=79) |
|-------------------------|--------------------|--------------------|
| Subsequent exacerbation | 70 (86%) | 50 (63%) |
| ocs | X (x%) | X (x%) |
| Antibiotics | x (x%) | x (x%) |
| OCS and antibiotics | X (x%) | X (x%) |

200879

## 13.12.24. Example Shell 24

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Table X

Summary of Time from Resolution of Index Exacerbation to Next Exacerbation

| | Treatment A (N=100) | Treatment B (N=100) |
|-------------------------|---------------------|---------------------|
| Subsequent exacerbation | x.xx | x.xx |
| Mean duration (days) | x.xx | X.XX |
| SD | x.xx | x.xx |
| Median duration (days) | x.xx | x.xx |
| Minimum duration (days) | x.xx | x.xx |
| Maximum duration (days) | x.xx | x.xx |

200879

## 13.12.25. Example Shell 25


Population: Intent-to-Treat/Safety/Other study specific

Summary of ECG Abnormalities for Participants with Any Abnormal Clinically Significant ECG Interpretation

| | Treatment A (N=100) | Treatment B (N=100) |
|---|---|---|
| Visit 2 (Day 1) | | |
| Abnormal - Clinically significant | 10 (10%) | 15 (15%) |
| Any finding | 5 (50%) | 5 (33%) |
| ST depression | 5 (50%) | 5 (33%) |
| Short PR Interval | 0 | 5 (33%) |
| T wave inversion | 0 | 5 (33%) |

Includes Scheduled, unscheduled and Early Withdrawal visits. Participants may have more than one abnormality at each visit.

200879

## 13.12.26. Example Shell 26


Population: Intent-to-Treat/Safety/Other study specific

Table X

Statistical Analysis of Change from Baseline in FEV1 (mL) (Dose Response Model)  $\qquad \qquad \text{Measured post-bronchodilator}$ 

| | Placebo<br>(N=xx) | DNX 5mg<br>(N=xx) | DNX 10mg<br>(N=xx) | DNX 25mg<br>(N=xx) | DNX 35mg (N=xx) | DNX 50mg<br>(N=xx) |
|---|---|---|---|---|---|---|
| n [1] Posterior Mean Change (SD) Posterior Median Change 95% Credible Interval | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) | xx<br>x.xx<br>(x.xxx)<br>x.xx<br>(x.xx,x.xx) |
| Column vs. Placebo Posterior Difference 80% Credible Interval | (****/*****) | x.xx<br>(x.xx, | x.xx<br>(x.xx, | x.xx<br>(x.xx, | x.xx<br>(x.xx, | x.xx<br>(x.xx, |
| Prob(Difference>0) Predictive probability (%) [2] [only if required] | | x.xx)<br>xx%<br>xx% | x.xx)<br>xx%<br>xx% | x.xx)<br>xx%<br>xx% | x.xx)<br>xx%<br>xx% | x.xx)<br>xx%<br>xx% |

<sup>[1]</sup> Number of subjects with data contributing to the analysis.

<sup>[2]</sup> Predictive posterior probability of success at end of study, where success is Pr(Difference>0)>90%. Note: Model fitted was a....[insert as appropriate].

200879

## 13.12.27. Example Shell 27

Protocol: ABC123456 

Population: Intent-to-Treat/Safety/Other study specific

Summary of QTc(F) (msec) Categories

| | Treat<br>(N=10 | ment A | Trea<br>(N=1 | tment B<br>00) |
|------------------|----------------|--------|--------------|----------------|
| Screening | | | | |
| n | XX | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |
| Day 1 (Baseline) | | | | |
| n | xx | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |
| Day 14 | | | | |
| n | XX | | XX | |
| <=450 | XX | (xx%) | XX | (xx%) |
| >450 to <=480 | XX | (xx%) | XX | (xx%) |
| >480 to <=500 | XX | (xx%) | XX | (xx%) |
| >500 | XX | (xx%) | XX | (xx%) |

200879

## 13.12.28. Example Shell 28


Population: Safety

| Visit 2 | (Day 1) |
|-----------|---------------------|
| mrrs o of | acuah. Cinala acuah |

>30

| Type of cough: Single cough | Treatment A (N=100) |
|-------------------------------------|---------------------|
| Did subject experience event [1]? | 12 (24%) |
| Cough severity | |
| Mild | 6 (50%) |
| Moderate | 5 (42%) |
| Severe | 1 (8%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 2 (17%) |
| >1-2 | 3 (25%) |
| >2-3 | 4 (33%) |
| >3-4 | 3 (25%) |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 7 (58%) |
| >1 - 2 | 2 (17%) |
| >2 - 3 | 3 (25%) |
| >3 - 4 | 0 |
| >4 - 5 | 0 |
| >5 - 10 | 0 |
| >10 - 30 | 0 |

<sup>[1]</sup> Percentages are calculated using the number of subjects evaluated at visit as the denominator.

All other percentages are calculated using the number of subjects with particular cough type at visit as the denominator.

# 2019N398117\_00


200879

Protocol: ABC123456
Population: Safety

Table X

Severe

Summary of Post-Inhalation Cough by Visit and Cough Type

Visit 2 (Day 1)
Type of cough: Single cough

Number of subjects reporting cough as AE/SAE

Mild

Moderate

Treatment A

(N=100)

4 (33%)

2 (17%)

2 (17%)

200879

Protocol: ABC123456
Population: Safety

#### 

| Type of cough: Intermittent cough | Treatment A (N=100) |
|-------------------------------------|---------------------|
| Did subject experience event [1]? | 11 (22%) |
| Cough severity | |
| Mild | 2 (18%) |
| Moderate | 6 (55%) |
| Severe | 3 (27%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 1 (9%) |
| >1-2 | 4 (36%) |
| >2-3 | 6 (55%) |
| >3-4 | 0 |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 0 |
| >1 - 2 | 3 (27%) |
| >2 - 3 | 6 (55%) |
| >3 - 4 | 1 (9%) |
| >4 - 5 | 0 |
| >5 - 10 | 0 |
| >10 - 30 | 1 (9%) |
| >30 | 0 |

200879


Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

Visit 2 (Day 1)

| Type of cough: Intermittent cough | Treatment A (N=100) |
|----------------------------------------------|---------------------|
| Number of subjects reporting cough as AE/SAE | 5 (45%) |
| Mild | 1 (9%) |
| Moderate | 2 (18%) |
| Severe | 2 (18%) |

200879

Protocol: ABC123456
Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

| Type of cough: Continuous cough | Treatment A<br>(N=100) |
|-------------------------------------|------------------------|
| Did subject experience event [1]? | 4 (8%) |
| Cough severity | |
| Mild | 1 (25%) |
| Moderate | 2 (50%) |
| Severe | 1 (25%) |
| Time to onset of PI cough (minutes) | |
| 0-1 | 3 (75%) |
| >1-2 | 1 (25%) |
| >2-3 | 0 |
| >3-4 | 0 |
| >4-5 | 0 |
| >5 | 0 |
| Duration of PI cough (minutes) | |
| <=1 | 0 |
| >1 - 2 | 0 |
| >2 - 3 | 0 |
| >3 - 4 | 1 (25%) |
| >4 - 5 | 1 (25%) |
| >5 - 10 | 0 |
| >10 - 30 | 1 (25%) |
| >30 | 1 (25%) |

200879


Population: Safety

Table X

Summary of Post-Inhalation Cough by Visit and Cough Type

Visit 2 (Day 1)

| Type of cough: Continuous cough | Treatment A (N=100) |
|----------------------------------------------|---------------------|
| Number of subjects reporting cough as AE/SAE | 2 (50%)<br>1 (25%) |
| Moderate<br>Severe | 1 (25%)<br>0 |

REPEAT FOR EACH VISIT

200879

## 13.12.29. Example Shell 29

Protocol: MID200879 

Population: Intent-to-Treat

| Randomized<br>Treatment | Centre/<br>Subj | Start<br>Date of<br>Dosing | End<br>Date of<br>Dosing | Duration<br>(Days) | Dispense Visit | Dispense<br>Date | Actual<br>Treatment<br>Dispensed |
|---|---|---|---|---|---|---|---|
| GSK2269557 500 mcg | PPD | xxxxxxxx | xxxxxxxx | xx | Visit 3 (Week 0) | XXFEB2013 | GSK2269557 500 mcg |
| | | XXXXXXXXX<br>XXXXXXXXX | XXXXXXXXX<br>XXXXXXXXX | XX<br>XX | Visit 5 (Week 4)<br>Visit 6 (Week 8) | | GSK2269557 100 mcg<br>GSK2269557 500 mcg |